| Division | ÷ | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for Study 206817: A Single Centre, Double Blind (Sponsor Open), Placebo Controlled, 3-Period Crossover, Ascending Dose Study in Japanese Healthy Elderly Male Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Danirixin in the Fed State (Part1) and an open label, 2-way crossover to evaluate food effect on the pharmacokinetics of Danirixin (Part2).

Compound Number : GSK1325756

Effective Date : 11-JUL-2017

#### **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the clinical pharmacology study report for protocol 206817.
- This RAP is intended to describe the safety, pharmacokinetics analyses required for the study.
- This document will be provided to the study team members to convey the content of the statistical analysis complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | |
|---|---|
| Biostatistics Group 1 Manager, Biomedical Data Sciences | 5-Jul-2017 |
| Department, Japan. | |
| PPD | |
| Clinical Pharmacology & Science Promotion Office, Medicines Development, Japan. | 5-Jul-2017 |

#### Approved:

| PPD | |
|----------------------------------------------------------|-------------|
| Department Manager, Biomedical Data Sciences Department, | 11-Jul-2017 |
| Japan. | |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | PRTING & ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMW<br>2.1.<br>2.2.<br>2.3.<br>2.4. | MARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s) Study Design Statistical Hypotheses | 6<br>6<br>7 |
| 3. | PLANN<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | 9 |
| 4. | ANALY | YSIS POPULATIONS | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 10 |
| 6. | STUD'<br>6.1. | Y POPULATION ANALYSESOverview of Planned Analyses | |
| 7. | SAFET<br>7.1.<br>7.2.<br>7.3. | TY ANALYSES Overview of Planned Adverse Events Analyses Overview of Planned Clinical Laboratory Analyses Overview of Planned Other Safety Analyses | 12<br>12 |
| 8. | PHAR<br>8.1.<br>8.2.<br>8.3. | Overview of Planned Pharmacokinetic Analyses Drug Concentration Measures Pharmacokinetic Parameters 8.3.1. Deriving Pharmacokinetic Parameters 8.3.2. Summary of Pharmacokinetic Parameters 8.3.3. Statistical Analysis of Pharmacokinetic Parameters | 14<br>15<br>15<br>17 |
| 9. | REFE | RENCES | 19 |
| 10. | APPEN<br>10.1.<br>10.2.<br>10.3.<br>10.4. | Appendix 1: Protocol Deviation Management Appendix 2: Time & Events Appendix 3: Treatment States and Phases 10.3.1. Treatment Phases 10.3.2. Treatment States Appendix 4: Data Display Standards & Handling Conventions 10.4.1. Study Treatment & Sub-group Display Descriptors 10.4.2. Sequence group Display Descriptors 10.4.3. Baseline Definition & Derivations 10.4.4. Reporting Process & Standards Appendix 5: Derived and Transformed Data | 21<br>25<br>25<br>26<br>26<br>26<br>27 |

#### **CONFIDENTIAL**

| | | 10.5.1. | General | 30 |
|---|---|---|---|---|
| | | 10.5.2. | Study Population | |
| | | 10.5.3. | Safety | |
| | | 10.5.4. | Pharmacokinetics | 32 |
| | 10.6. | | x 6: Premature Withdrawals & Handling of Missing Data | |
| | | 10.6.1. | Premature Withdrawals | |
| | | 10.6.2. | Handling of Missing Data | |
| | | 10.6.3. | Handling of Partial Dates | |
| | | 10.6.4. | Handling of Missing Data for Statistical Analysis | |
| | 10.7. | Appendix | x 7: Values of Potential Clinical Importance | |
| | | 10.7.1. | Laboratory Values (Healthy Volunteers) | |
| | | 10.7.2. | ECG (Healthy Volunteers) | |
| | | 10.7.3. | Vital Signs (Healthy Volunteers) | |
| | 10.8. | Appendix | x 8 - Abbreviations & Trade Marks | |
| | | 10.8.1. | Abbreviations | 36 |
| | | 10.8.2. | Trademarks | 37 |
| | 10.9. | Appendix | x 9: List of Data Displays | 38 |
| | | 10.9.1. | Data Display Numbering | |
| | | 10.9.2. | Mock Example Referencing | |
| | | 10.9.3. | Deliverable [Priority] | |
| | | 10.9.4. | Study Population Tables | |
| | | 10.9.5. | Safety Tables | |
| | | 10.9.6. | Pharmacokinetic Tables | |
| | | 10.9.7. | Pharmacokinetic Figures | 45 |
| | | 10.9.8. | ICH Listings | 47 |
| | 10.10. | Appendix | x 10: Example Mock Shells for Data Displays | 53 |
| | | 10.10.1. | Study population | 53 |
| | | 10.10.2. | Safety population | 76 |
| | | | PK population | |
| 11 | DE\/IS | | rodiv | 100 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206817. |
| Protocol | Reporting and Analysis Plan is based on original protocol (Dated:11-Apr-2017) for study GSK1325756 / 206817 [GlaxoSmithKline Document Number:2016N309585_0] |
| Objectives | Part 1 |
| | <ul> <li>To assess the safety, tolerability and PK following single doses of GSK1325756H 10,<br/>50 and 100 mg in the fed state in healthy Japanese subjects of over 65 years of age<br/>inclusive.</li> </ul> |
| | Part 2 |
| | <ul> <li>To investigate the safety, tolerability and food effect on PK of GSK1325756 following a<br/>single dose of 50 mg in the fed and fasted state, in healthy Japanese subjects of over<br/>65 years of age inclusive.</li> </ul> |
| Endpoints | Part 1 and 2. |
| | Adverse events (AEs) |
| | Change from baseline of clinical laboratory values, vital signs, and electrocardiogram (ECG) parameters |
| | Blood concentration of GSK1325756 |
| | <ul> <li>Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, tlag, tlast of the blood<br/>concentration of GSK1325756, as data permit</li> </ul> |
| Study | This study consists of two parts. |
| Design | <ul> <li>Part 1 is a double blind, placebo-controlled, 3-period crossover, ascending dose, single<br/>oral administration in the fed condition</li> </ul> |
| | Part 2 is an open label, 2-way crossover, single oral dose in the fed and fasted state. |
| Analysis | Screened: Consisting of all subjects screened in the study |
| Population | Screening Failure: Subjects who screened in the study but are never subsequently randomized. |
| | Safety: All randomized subjects who take at least one dose of study treatment. |
| | Pharmacokinetic: This population is defined as all subjects administered at least one dose of study treatment and who have PK sample taken and analysed. |
| Hypothesis | The objectives of this study are to evaluate safety and tolerability of GSK1325756 and to estimate GSK1325756 Pharmacokinetic parameters. No formal statistical hypotheses will be tested in Part 1 and Part 2. Descriptive statistics will be used to assess safety and tolerability objectives. An estimation approach will be used to address the pharmacokinetic study objectives, where point estimates and corresponding 90% confidence intervals will be constructed. |
| Safety<br>Analyses | Safety data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. |
| Pharmacoki<br>netic<br>Analyses | Individual GSK1325756 blood concentration-time profiles (by part, treatment and subject) and median/mean (±SD) profiles by part and treatment will be plotted and listed. Treatment indicates dose group in Part 1 and the fed and fasted condition in Part 2. |
| | Blood concentration time data for GSK1325756 will be analyzed by non-compartmental methods using WinNonlin and derived PK parameters graphically present, summarised |

#### **CONFIDENTIAL**

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| | and listed. No formal statistical analyses will be conducted. |
| | <ul> <li>Statistical analyses will be carried out to explore the dose proportionality of<br/>GSK1325756 as assessed by AUC(0-t) and Cmax using the Power Model (Part 1).</li> </ul> |
| <ul> <li>Statistical analyses will be carried out to explore the food effect of GSK132<br/>assessed by AUC(0-t) and Cmax using a mixed effects mode (Part 2).</li> </ul> | |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [Dated: 11/APR/2017].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Part 1 | Part 1 and Part 2 |
| <ul> <li>To assess the safety, tolerability and PK<br/>following single doses of GSK1325756H 10,<br/>50 and 100 mg in the fed state in healthy<br/>Japanese subjects of over 65 years of age<br/>inclusive.</li> </ul> | <ul> <li>Adverse events (AEs)</li> <li>Change from baseline of clinical laboratory values, vital signs, and electrocardiogram (ECG) parameters</li> <li>Blood concentration of GSK1325756</li> </ul> |
| <ul> <li>Part 2</li> <li>To investigate the safety, tolerability and food effect on PK of GSK1325756 following a single dose of 50 mg in the fed and fasted state, in healthy Japanese subjects of over 65 years of age inclusive.</li> </ul> | <ul> <li>Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2,<br/>tlag, tlast of the blood concentration of<br/>GSK1325756, as data permit</li> </ul> |

# 2.3. Study Design

# **Overview of Study Design and Key Features**

Subjects will be divided into Part 1 and 2, and receive the following study treatment doses shown in Table below.

#### Part 1:

| Group | n | Period 1 | Washout | Period 2 | Washout | Period 3 |
|---|---|---|---|---|---|---|
| Α | 6 | 10 mg | | 50 mg | | Placebo |
| В | 6 | 10 mg | at least 7<br>days | Placebo | at least 7<br>days | 100 mg |
| С | 6 | Placebo | | 50 mg | - | 100 mg |

#### Part 2:

| Group | n | Period 1 | Washout | Period 2 |
|-------|---|---------------|------------|---------------|
| D | 8 | 50 mg, fed | at least 7 | 50 mg, fasted |
| Е | 8 | 50 mg, fasted | days | 50 mg, fed |

| Design<br>Features | Part 1: This is a double blind, placebo-controlled, 3-period crossover, ascending dose, single oral administration in the fed condition. |
|---|---|
| | Part 2: This is an open label, 2-way crossover, single oral dose in the fed and fasted state study. |
| Dosing | Part 1: Subjects will have a screening visit within 30 days prior to the first dose of study. A minimum washout period of 7 days will be required between each treatment period. Subjects will receive three treatment periods in the study. Subjects will be housed in the Clinical Research Unit from Day -1 (the day before dosing) through Day 3 for Period 1 and 2, and from Day -1 (the day before dosing) through Day 4 for Period 3. Subjects will return to the clinic 7 days (at least) after the previous administration day for Period 1 and 2, and subjects will visit the unit on Day 8 (+/- 1 day) of the last dosing for Period 3 for follow-up. |
| | Part 2:<br>Subjects will have a screening visit within 30 days prior to the first dose of study treatment, two treatment periods separated by at least 7 days, and follow-up. Subjects will be housed in the Clinical Research Unit from Day -1 (the day before dosing) through Day 3 (for Period 1 and 2), and re-visit 7 (±1) days after the last dose of Period 2 for follow-up. |
| Treatment<br>Assignment | • Sufficient participants will be randomised such that approximately 18 in Part 1 and 16 in Part 2 evaluable participants complete the study of |

# **Overview of Study Design and Key Features** each part. If participants prematurely discontinue the study, additional participants may be enrolled as replacement participants and assigned to the same treatment sequence, if applicable, at the discretion of the sponsor in consultation with the investigator. On Day 1 of each Part, participants will be assigned a unique number (randomization number) in ascending numerical order. The randomization number encodes the participant's assignment to one of the 3 sequences in Part 1 and one of the 2 sequences in Part 2. according to the randomization schedule generated prior to the study by the Biomedical Data Sciences Department at GSK. Participants will be randomized in a 1:1:1 ratio to receive sequence (A:B:C) for Part 1, or will be randomized in a 1:1 ratio to receive sequence (D:E) for Part 2. Each participant will be dispensed blinded study treatment, labeled with his unique randomization number, throughout the study. Investigators, participants and sponsor will remain blinded to each participant's assigned study treatment throughout the course of the study. For the concentration evaluation after Period 2 of Part 1, the pre-specified sponsor's person who is responsible for the confirmation of the concentration will review blood drug concentration data under unblended. No formal statistical analysis is planned. Interim **Analysis** A blind review of preliminary safety data (AE, clinical laboratory values, vital signs, ECG) and blood concentration will be conducted between Period 2 and Period 3 in Part 1 and prior to Part 2. After completion of Part 1, formal analysis for Part 1 is to be conducted.

# 2.4. Statistical Hypotheses

The objectives of this study are to evaluate safety, tolerability and PK profile of single dose of GSK1325756H and to investigate food effect of PK profile of single dose of GSK1325756H in healthy Japanese elderly subjects. No formal statistical hypotheses will be tested in Part 1 and Part 2. Descriptive statistics will be used to assess safety and tolerability objectives. An estimation approach will be used to address the PK study objectives, where point estimates and corresponding 95% confidence intervals will be constructed, unless otherwise stated.

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal statistical analysis is planned. However, following Period 1 and Period 2 of Part 1, a blind review of preliminary safety data (AE, clinical laboratory values, vital signs, ECGs) will be conducted between Period 2 and Period 3 in Part 1 and prior to Part 2. Furthermore, the sponsor's person who is responsible for the confirmation of the concentration will review blood drug concentration data under unblended.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects in each part have completed the study as defined in the protocol.
- 2. All required database cleaning activities in each part have been completed and final database release and database freeze has been declared by Data Management for each part.
- 3. All criteria for unblinding the randomisation codes have been met for Part 1.
- 4. Randomisation codes have been distributed according to RandAll NG procedures. After completion of Part 1, formal analysis for Part 1 is to be conducted.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Screened | Consisting of all subjects screened in the study. | Study Population |
| | Note: This definition indicates the same meaning as 'All subjects who have subject number' in a programming point of view. | |
| Screening Failure | Subjects who screened in the study but are<br>never subsequently randomized. All<br>participants who sign the ICF have the<br>screening test in the study. | Study Population |
| | Note: This definition indicates the same meaning as 'Subjects who have subject number but are never subsequently randomized' in a programming point of view. | |
| Safety | All randomized subjects who take at least and does of study treatment. Participants will | Study Population |
| | one dose of study treatment. Participants will be analyzed according to the treatment they actually received. | Safety |
| Pharmacokinetic | This population is defined as all subjects | • PK |

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| | administered at least one dose of study treatment and who have PK sample taken and analysed. Participants will be analyzed according to the treatment they actually received. | |

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - o This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided. This will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|--------------------------------------------------------------|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Treatment States and Phases |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety Population, unless otherwise specified. These analyses will be performed in each part.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Disposition Disposition and Reason for Study Withdrawal ng Status and Reasons for Screen Failure s for Whom the Treatment Blind was Broken | Table | Figure | Listing |
|---|---|---|---|
| Disposition and Reason for Study Withdrawal ng Status and Reasons for Screen Failure s for Whom the Treatment Blind was Broken | Υ | 1 | |
| ng Status and Reasons for Screen Failure<br>s for Whom the Treatment Blind was Broken | Y | | |
| for Whom the Treatment Blind was Broken | | | Υ |
| | Y | | Υ |
| 14 / 17 / | | | Υ |
| and Actual Treatments | | | Υ |
| l Deviations | | | |
| nt Protocol Deviations | Y | | Υ |
| n/Exclusion Criteria Deviations | | | Υ |
| ions Analysed | | | |
| opulations | Y | | |
| Excluded from Any Population | | | Υ |
| raphic and Baseline Characteristics | • | | |
| aphic Characteristics | Y | | Υ |
| aphic Characteristics for Screening Failure | | | Υ |
| nges | Y | | |
| d Racial Combinations | Y | | Υ |
| d Racial Combinations for Screening Failure | | | Υ |
| Conditions and Concomitant Medications | • | | |
| Conditions | | | Υ |
| itant Medications | | | Υ |
| re and Treatment Compliance | • | | |
| e to Study Treatment | | | Υ |
| | • | • | |
| rt and end days/times on fed treatment | | | Υ |

#### NOTES:

• Y = Yes display generated.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety Population, unless otherwise specified. These analyses will be performed in each part.

Adverse events occurred in washout period will be included in adverse events analyses for previous period. Also adverse events occurred in follow up period will be included in safety analyses for the last period.

#### 7.1. Overview of Planned Adverse Events Analyses

Table 3 provides an overview of the planned adverse events analyses with full details of data displays being presented in Appendix 9: List of Data Displays.

Table 3 Overview of Planned Adverse Event Analyses

| Display Type | | Absolute | |
|---|---|---|---|
| | Sumr | Individual | |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Y | | Υ |
| All AEs by Maximum Intensity | Y | | |
| Drug-Related AEs by SOC and PT | Y | | |
| Drug-Related AEs by Maximum Intensity | Y | | |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Serious AEs | | | Υ |
| AEs Leading to Withdrawal from Study | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.2. Overview of Planned Clinical Laboratory Analyses

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 4 Overview of Planned Clinical Laboratory Analyses

| Display Type | play Type Absolute | | | Change from BL | | |
|---|---|---|---|---|---|---|
| | | mary | Individual | Summary | | Individual |
| | Т | F | L | T | F | L |
| Chemistry | | | | | | |
| Chemistry Data | Υ | | Y | Υ | | Y |

| Display Type | | Absolute | | | Change from BL | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry Results Relative to Normal Range | | | | Υ | | |
| All Chemistry Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | Y |
| Hematology | | | | | | |
| Hematology Data | Υ | | Υ | Υ | | Υ |
| Hematology Results Relative to Normal Range | | | | Υ | | |
| All Hematology Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | Y |
| Urinalysis | _ | | | | | |
| Dipstick Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) | Υ | | Υ* | | | |
| Gravity and pH | Υ | | Y | | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | | | Υ | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.3. Overview of Planned Other Safety Analyses

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 5 Overview of Planned Other Safety Analyses

| Display Type | | Absolute | | | Change from BL | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | l Summary | | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Υ | | | |
| ECG Values | Υ | | Y | Υ | | Y |
| All ECG Values for Subjects with any Value of PCI | | | Y | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | Υ |
| All Vital Signs for Subjects with any Value of PCI | | | Y | | | |

<sup>\*:</sup> If blood or protein is abnormal, microscopic examination will be included.

| Display Type | | Abso | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | | mary | Individual | Summary | | Individual |
| | Т | F | L | T | F | L |
| Ophthalmic examinations | | | | | | |
| Ophthalmic examinations | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8. PHARMACOKINETIC ANALYSES

## 8.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic population, unless otherwise specified. These analyses will be performed in each part.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| Display Type | ι | Intrans | sformed | | | ned | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Stats<br>analysis | Summary | | Individua | |
| | F | Т | F | L | | F T | | F | L |
| Descriptive statistics | | | | | | | | | |
| Blood Drug Concentrations | Y [1] [2] | Υ | <b>Y</b> [1] | Υ | | | | | |
| Derived PK Parameters | Υ | Υ | | Υ | | | Υ | | |
| Statistical Analysis of PK Parameters | | | | | | | | | |
| Power model (Part 1) | | · | | | Y | | | | |
| Food effect (Part 2) | | | | | Y | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (+ SD) and Median plots will be generated.

# 8.2. Drug Concentration Measures

Blood concentrations of GSK1325756 will be listed and summarised by part, treatment and nominal time. Standard summary statistics will be calculated (i.e. mean, standard deviation, median, minimum and maximum).

Individual blood concentration-time profiles and median/mean profiles by treatment will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.4 Reporting Process & Standards).

#### 8.3. Pharmacokinetic Parameters

#### 8.3.1. Deriving Pharmacokinetic Parameters

- Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology & Science Promotion Office, GlaxoSmithKline K.K.
- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.4 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis using WinNonlin (version 6.3 or higher)
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.
- Pharmacokinetic parameters described in Table 7 will be determined from blood GSK1325756 concentration-time data, as data permits.

Table 7 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-24)<br>(h*ng/mL) | Area under the concentration-time curve will be calculated to fixed nominal time 24 hours after administration (AUC(0-24)), using the combination of linear and logarithmic trapezoidal methods (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| | If a sampling time deviation occurred at nominal time 24 hours after administration (and 24 < t), AUC(0-24) will be calculated using the concentration at time 24 hours after administration post-dose estimated by the method of interpolation. |
| | If nominal time 24 hours after administration > t (or if the concentration at time 24 hours after administration was below then limit of quantification), then the concentration (y) at time 24 hours after administration is estimated using lambda_z and last observed Ct according to the formula: |
| | y=Ct(obser) x e-lambda_z(24-t) |
| | Then the following equation will be used to calculate (AUC(0-24)) where t is the time of last quantifiable blood concentration. |

| Parameter | Parameter Description |
|---|---|
| | AUC(0-24) = AUC(0-t) + AUC(t-24) |
| | If lambda_z is not estimable, a partial AUC is not calculated (when 24 > t). |
| AUC(0-t)<br>(h*ng/mL) | Area under the concentration-time curve from zero time (pre-dose) to the time of the last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| AUC(0-inf)<br>(h*ng/mL) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: |
| | AUC(0-inf) = AUC(0-t) + Ct / lambda_z |
| Cmax (ng/mL) | Maximum observed concentration will be obtained directly from the concentration-time data. |
| Tmax (h) | Time to first occurrence of Cmax will be obtained directly from the concentration-time data. |
| t1/2 (h) | Terminal phase half-life will be calculated as follows: |
| | t1/2 = ln2 / lambda_z |
| tlag (h) | Lag time before observation of drug concentrations in sampled matrix. |
| tlast (h) | The time of the last measurable (positive) concentration. |
| %AUCex (%) | The area under the curve (AUC) from the last predicted non-zero concentration value to infinity as a percentage of the area under the curve extrapolated to infinity. |
| lambda_z (/h) | The first order rate constant associated with the terminal (log-linear) portion of the curve. |
| lambda_z_lower (h) | The lower limit on time for values to be included in the calculation of Lambda z. |
| lambda_z_upper (h) | The upper limit on time for values to be included in the calculation of Lambda z. |
| #pts | The number of time points used in computing Lambda z. |
| R2 | The goodness of fit statistic for the terminal elimination phase. |

# NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.
- Ct is the last observed quantifiable concentration.

#### 8.3.2. Summary of Pharmacokinetic Parameters

- For each of these parameters, except for tmax, tlag and tlast, the following summary statistics will be calculated for each treatment:
  - o Non-transformed: arithmetic mean, median, maximum, minimum, 95% confidence interval for the arithmetic mean and standard deviation
  - Loge-transformed: geometric mean, 95% confidence interval for the geometric mean, standard deviation of logarithmically transformed data and between geometric coefficient of variation (CVb (%))
- Median, maximum, minimum, arithmetic mean, 95% confidence interval and standard deviation will be calculated for tmax, tlag and tlast.

#### 8.3.3. Statistical Analysis of Pharmacokinetic Parameters

#### 8.3.3.1. Dose proportionality

For Part 1, the PK-dose relationship will be investigated graphically in order to assess dose proportionality of GSK1325756. Plots of AUC (0-t) and Cmax versus dose will be plotted.

Also statistical analyses will be carried out to explore the dose proportionality of GSK1325756 as assessed by AUC(0-t) and Cmax, using the Power Model:

```
\log_e (Y_{ii}) = \mu + S_i + \beta * \log_e (D_i) + \varepsilon_{ii}
```

Y<sub>ij</sub>: PK parameter (AUC(0-t), Cmax) on the *j*th dose for *i*th subject

μ: Overall mean (Intercept)

 $S_i$ : Random effect for subject i following normal distribution  $N(0, \sigma_b^2)$ 

β: Slope for log<sub>e</sub> transformed dose

 $D_i$ : Dose (j=1:10mg, 2:50mg, 3:100mg)

 $\varepsilon_{ii}$ : Random error following normal distribution N(0,  $\sigma_{w}^{2}$ )

Following loge-transformation, AUC (0-t) and Cmax will be separately analyzed, if data permitted. A mixed effect model will be fitted with the loge transformed dose and period as fixed effects. Subject will be fitted as a random effect. The Kenward & Roger (KR) degrees of freedom approach will be used. Point estimates and their associated 90% confidence intervals will be constructed.

#### 8.3.3.2. Food effect

For Part 2, statistical analyses will be carried out to assess treatment (food effect) of GSK1325756 for AUC(0-t) and Cmax using Mixed effect model:

$$\log_e(Y_{ij}) = \mu + S_i + t_j + p_k + \varepsilon_{ij}$$

 $Y_{ij}$ : PK parameter (AUC(0-t), Cmax) on the *j*th treatment for *i*th subject

μ: Overall mean (Intercept)

 $S_i$ : Random effect for subject i following normal distribution  $N(0, \sigma_b^2)$ 

t<sub>i</sub>: Treatment effect (j=fasted, fed)

p<sub>k</sub>: Period effect (k=period 1, period 2)

 $\varepsilon_{ij}$ : Random error following normal distribution N(0,  $\sigma_w^2$ )

Following loge-transformation, AUC (0-t) and Cmax will be separately analysed using a mixed effects model fitting terms for treatment and period as fixed effects, and subject as a random effect in order to assess food effect of GSK1325756 (Fed vs. Fasted). The Kenward & Roger (KR) degrees of freedom approach will be used.

Point estimates for the adjusted means on the loge scale, the mean difference between treatments and associated 90% confidence interval will be constructed using the residual variance. The point estimate and confidence interval will then be exponentially backtransformed to obtain adjusted (least square) geometric means for each treatment, and point estimates and associated 90% confidence interval for the ratio of fasted/fed.

Estimates of within-subject variability (CVw (%)) for AUC (0-t) and Cmax will also be provided. CVw (%) will be calculated based on the loge-normal distribution where:

CVw (%)= SQRT(exp(MSE)-1) \* 100. (MSE is the residual mean squared error from the model)

## 9. REFERENCES

GlaxoSmithKline Document Numbers 2016N309585\_01: Study Protocol of 206817. A Single Centre, Double Blind (Sponsor Open), Placebo Controlled, 3-Period Crossover, Ascending Dose Study in Japanese Healthy Elderly Male Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Danirixin in the Fed State (Part1) and an open label, 2-way crossover to evaluate food effect on the pharmacokinetics of Danirixin (Part2).

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General |
| | Study Population |
| | Safety |
| | Pharmacokinetics |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | General |
| | Study Population & Safety |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Other RAP App | endices |
| Section 10.8 | Appendix 8: Abbreviations & Trade Marks |
| Section 10.9 | Appendix 9: List of Data Displays |
| Section 10.10 | Appendix 10: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management

Details will be referred latest Protocol Deviation Management Plan and data handling will be decided prior to final data base release.

# 10.2. Appendix 2: Time & Events

# Part 1, Period 1-2

| Day | | | | | | | | | Day 1 | | | | | | | Day 2 | Day 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose | Screening | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5 h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Subject demography<br>/Medical history | X | | | | | | | | | | | | | | | | |
| Height, Weight, BMI | X | | | | | | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | | | | | | | |
| Serological test | X | | | | | | | | | | | | | | | | |
| Physical examination | X | Х | Х | | | | | | | | Х | | | | | X | Х |
| Vital signs (PR, BP, temp) | х | Х | Х | | | | | | | | Х | | | | | Х | X |
| 12-lead ECG | X | Х | Х | | | | | | | | Х | | | | | X | Х |
| Ophthalmic examination | X3 | | | | | | | | | | | | | | | | |
| SAEs <sup>2</sup> | <====== | | | | | | | | | | | | | | | | ====> |
| AEs <sup>2</sup> | | | | <==: | | | | | | | | | | | | | ====> |
| Con Med review | <====== | | | | | | | | | | | | | | | | ====> |
| Hematology, clinical<br>chemistry and urinalysis | X | Х | | | | | | | | | | | | | | | X |
| Administration | | | | Χ | | | | | | | | | | | | | |
| PK sampling | | | Х | | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Х | X |
| Admission | | Χ | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | Х |

Screening visit will occur only prior to the first dosing. Treatment Period 2 will occur after at least 7-days wash-out period. High fat meal will be started and completed before within 30 minutes of GSK1325756H/Placebo dosing.

All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified (see Section 9.1 Adverse Events).

<sup>3.</sup> Ophthalmic examinations are conducted on the day between Screening and Day-1. However, it is not carried out for those who are ineligible due to other screening criteria.

# Part 1, Period 3

| Day | | | | | | | | Day 1 | | | | | | | Day 2 | Da | y 3 | Day 4 | Follow |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5<br>h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h | 60 h | 72 h | up <sup>2,3</sup> |
| Physical examination | Х | Х | | | | | | | | Х | | | | | Х | Х | | Х | х |
| Vital signs (PR,<br>BP, temp) | Х | Х | | | | | | | | Х | | | | | Х | Х | | х | Х |
| 12-lead ECG | Х | Х | | | | | | | | Х | | | | | Х | Х | | Х | Х |
| Ophthaimic<br>examination | | | | | | | | | | | | | | | | | | | X |
| SAEs | <=== | | | | | | | | | | | | | | | | | | :===> |
| AEs | <=== | | | | | | | | | | | | | | | | | | ====> |
| Con Med review | <=== | ====== | ===== | | ===== | | ===== | | | ===== | ===== | | | | | ====== | | | ===> |
| Hematology,<br>clinical chemistry<br>and urinalysis | x | | | | | | | | | | | | | | | | | x | x |
| Administration | | | Х | | | | | | | | | | | | | | | | |
| PK sampling | | Χ | | X | X | X | Х | X | X | Χ | X | X | X | X | Χ | X | X | Х | |
| Admission | X | | | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | | X | |

Treatment Period 3 will occur after at least 7-days wash-out period. High fat meal will be started and completed before within 30 minutes of GSK1325756/Placebo dosing.
 Follow up visit will occur after 7 days (+/- 1day) of the last dosing.
 In the case where the subject has discontinued the study prematurely, the assessments for follow up will be carried out.

### Part 2, Period 1-2

| Day | | | | | | | | | Day 1 | | | | | | | Day 2 | Day 3 | Follow |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose Screen | Screening | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5<br>h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h | up <sup>3,5</sup> |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Subject demography<br>/Medical history | Х | | | | | | | | | | | | | | | | | |
| Height, Weight, BMI | X | | | | | | | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | | | | | | | | |
| Serological test | X | | | | | | | | | | | | | | | | | |
| Physical examination | Х | Х | Х | | | | | | | | Х | | | | | Х | X | Х |
| Vital signs (PR, BP, temp) | Х | х | Х | | | | | | | | Х | | | | | Х | Х | Х |
| 12-lead ECG | X | Х | Х | | | | | | | | Х | | | | | Х | Х | Х |
| Ophthalmic<br>examination | X6 | • | | | | | | | | | | | | | | | | Х |
| SAEs4 | <===== | | | | | | | | | | | | | | | | | ====> |
| AEs4 | | | | <== | | | | | | | | | | | | | | -===> |
| Con Med review | <===== | | | | | | | | | | | | | | | | | :===> |
| Hematology, clinical<br>chemistry and<br>urinalysis | х | х | | | | | | | | | | | | | | | х | х |
| Administration | | | | Χ | | | | | | | | | | | | | | <del> </del> |
| PK sampling | | | Х | | Х | Х | Х | Х | Х | Χ | Х | Х | Χ | X | Χ | Х | Х | $\vdash$ |
| Admission | | Х | | | | | | | | | | | | | | | | 1 |
| Discharge | | | | | | | | | | | | | | | | | Х | 1 |

- 1. Screening visit will occur only prior to the first dosing. Treatment Period 2 will occur after at least 7-days wash-out period.
- 2. For the fed condition, meal will be started and completed before within 30 minutes of GSK1325756H dosing.
- 3. Follow up visit will occur after 7-days (+/- 1day) of the last dosing.
- 4. All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified (see Section 9.1.Adverse Events).
- 5. In the case where the subject has discontinued the study prematurely, the assessments for follow up will be carried out.
- 6. Ophthalmic examinations are conducted on the day between Screening and Day-1. However, it is not carried out for those who are ineligible due to other screening criteria.

# 10.3. Appendix 3: Treatment States and Phases

#### 10.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the assessment date.

| Treatment Phase | Definition |
|---|---|
| Part 1: Period 1 | Assessment Date < Previous Day of Dosing Start Date in Period 2 (Part 1) |
| Part 1: Period 2 | Previous Day of Dosing Start Date in Period 2 ≤ Assessment Date < Previous Day of Dosing Start Date in Period 3 (Part 1) |
| Part 1: Period 3 | Previous Day of Dosing Start Date in Period 3 ≤ Assessment Date (Part 1) |
| Part 2: Period 1 | Assessment Date < Previous Day of Dosing Start Date in Period 2 (Part 2) |
| Part 2: Period 2 | Previous Day of Dosing Start Date in Period 2 ≤ Assessment Date (Part 2) |

#### 10.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.3.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date and Time < Dosing Start Date and Time |
| Part 1: Period 1 | Dosing Start Date and Time in Period 1 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 2 (Part 1) |
| Part 1: Period 2 | Dosing Start Date and Time in Period 2 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 3 (Part 1) |
| Part 1: Period 3 | Dosing Start Date and Time in Period 3 ≤ AE Start Date and Time (Part 1) |
| Part 2: Period 1 | Dosing Start Date and Time in Period 1 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 2 (Part 2) |
| Part 2: Period 2 | Dosing Start Date and Time in Period 2 ≤ AE Start Date and Time (Part 2) |
| 0 17 0 | If Dosing Start Date and Time > AE Onset Date and Time = AE Onset Date and Time – Dosing Start Date and Time |
| Onset Time Since<br>First Dose (Minute) | If dosing Start Date and Time ≤ AE Onset Date and Time = AE Onset Date and Time - Dosing Start Date and Time +1 |
| | Missing otherwise |
| Onset Time Since<br>Last Dose (Minute) | AE Start Date and Time – Most Recent Treatment Start Date and Time + 1 |
| Duration (Minute) | AE Resolution Date and Time – AE Onset Date and Time + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF |

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

#### 10.4.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | Part1 (So | cedule1) | |
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| Р | Placebo, Fed | Placebo, Fed | 1 |
| X1 | GSK1325756H 10 mg, Fed | GSK1325756H 10 mg, Fed | 2 |
| X2 | GSK1325756H 50 mg, Fed | GSK1325756H 50 mg, Fed | 3 |
| Х3 | GSK1325756H 100 mg, Fed | GSK1325756H 100 mg, Fed | 4 |
| | Part2 (Scedule2) | | |
| X2 | GSK1325756H 50 mg, Fed | GSK1325756H 50 mg, Fed | 1 |
| X4 | GSK1325756H 50 mg, Fasted | GSK1325756H 50 mg, Fasted | 2 |

#### NOTES:

#### 10.4.2. Sequence group Display Descriptors

| | Sequence Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description [1] | Order |
| Α | X1/X2/P | A | 1 |
| В | X1/P/X3 | В | 2 |
| С | P/X2/X3 | С | 3 |
| D | X2/X4 | D | 4 |
| E | X4/X2 | Е | 5 |

#### NOTES:

Footnote will be added in displays as follows.
 A: 10mg (Fed) / 50mg (Fed) / Placebo (Fed), B: 10mg (Fed) / Placebo (Fed) / 100mg (Fed), C: Placebo (Fed) / 50mg (Fed) / 100mg (Fed), D: 50mg (Fed) / 50mg (Fasted) , E: 50mg (Fasted) / 50mg (Fed)

<sup>1.</sup> Order in which treatments are to be presented in Listings. Note that the order in which treatments are to be presented in Tables, active treatment (X1, X2, X3 in Part 1, X2, X4 in Part 2) is shown in the first and placebo (P in Part 1) in the second.

#### 10.4.3. Baseline Definition & Derivations

#### 10.4.3.1. Baseline Definitions

| Parameter | Study Asse | essments (<br>as Baselin | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| raidilletei | Screening Day -1 | | | |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | Х | Х | Day 1<br>(Pre Dose) |
| Haematology | Х | Χ | | Day -1 |
| Clinical Chemistry | Χ | Χ | | Day -1 |

#### NOTES:

• The baseline will be defined for each period in Part 1 and Part 2.

#### 10.4.3.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.3.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.4.4. Reporting Process & Standards

| Reporting Pro | ocess |
|---|---|
| Software | Software |
| The curre | ntly supported versions of SAS software will be used. |
| Reporting Ar | ea |
| HARP<br>Server | : uk1salx00175 |
| HARP Area | Part1:/arenv/arprod/gsk1325756/mid206817/primary_01 |
| | Part2:/arenv/arprod/gsk1325756/mid206817/final_01 |
| QC | Part1:/arenv/arprod/gsk1325756/mid206817/primary_01/qc |
| Spreadsheet | Part2:/arenv/arprod/gsk1325756/mid206817/final_01/qc |
| Analysis Data | Analysis Datasets |
| Analysis c | Analysis datasets will be created according to GSK IDSL A&R dataset standards |
| Generation of RTF Files | |
| • N/A | • N/A |

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (4.24) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | 5 |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data N, n, frequency, % | |
| Reporting of Pharmac | Reporting of Pharmacokinetic Concentration Data |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

| Reporting Standards | |
|---|---|
| Reporting of Pharmaco | Reporting of Pharmacokinetic Parameters |
| Descriptive Summary<br>Statistics.<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb/w (%)) will be reported. |
| | CVb (%) = SQRT (exp(SD <sup>2</sup> ) - 1) * 100 |
| | (SD = SD of loge-transformed data) |
| | CVw (%) =SQRT (exp(MSE) - 1) * 100 |
| | (MSE = mean square error from mixed effect model of loge-transformed data). |
| Parameters Not Being Log Transformed | tmax, tlag, tlast |
| Parameters Not Being<br>Summarised | The following PK parameters will not be summarised but listed: %AUCex, lambda_z, lambda_z_lower, lambda_z_upper, #pts, R2. |
| <b>Graphical Displays</b> | Graphical Displays |
| Refer to IDSL Statis | Refer to IDSL Statistical Principals 7.01 to 7.13. |

### 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from start of dosing date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < of start of dosing Date → Study Day = Ref Date of start of dosing Date</li>
- Ref Data ≥ of start of dosing Date → Study Day = Ref Date (of start of dosing Date) + 1

## 10.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Reference will be Randomization date for Part 1 and Part 2
- Reference date for calculation of age at screening will be from visit 1 (Screening visit) date, however this will be from screen failure date for a screen failure subject.
- Analysis age group will be categorized (Years):
  - <=18, 19-64, 65-74, >=75
- Age will be categorized for EudraCT:
  - <=17 years, 18-64 years, 65-84 years, >=85 years

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### 10.5.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
- Example 1: 2 Significant Digits = '< x ' becomes x 0.01
- Example 2: 1 Significant Digit = '> x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x 1

| Laboratory Assessments | |
|---|---|
| Haematology | Platelet Count, RBC Count, Haemoglobin, Hematocrit, RBC Indices (MCV, MCH, %Reticulocytes), WBC count with Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils) |
| Clinical Chemistry | BUN, Creatinine, Glucose (fasting), Uric acid, HDL-cholesterol, Amylase, Potassium, Sodium, Calcium, TG, LDH, Chloride, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatise, Total Cholesterol, GGT, Phosphorus, Total and direct bilirubin, Total Protein, Albumin, LDL-cholesterol, CK (CPK) |
| Routine Urinalysis | <ul> <li>Specific gravity, pH (assessed by dipstick)</li> <li>glucose, protein, blood, ketones, bilirubin, urobilinogen by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> |

#### ECG (12-lead ECG)

ECG findings, ECG values (Heart rate, PR interval, QRS duration, QT interval and QTcF intervals)

#### **Vital Signs**

Pulse rate, Blood pressure (Systolic, Diastolic), Temperature

#### **Ophthalmic examinations**

Ophthalmic examinations

#### 10.5.4. Pharmacokinetics

#### **PK Parameters**

- If one or more non-quantifiable (NQ) values occur in a profile before the first measurable
  concentration, they will be assigned a value of zero concentration. For linear plots, zero
  concentration value(s) before the first measurable concentration will be included in the plot. For
  log-linear plots, zero concentration value(s) before the first measurable concentration will be
  assigned a missing value.
- If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be set to missing in the derivation of pharmacokinetic parameters, statistical analysis, and the individual subject plots.
- If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be set to missing.
- NQs which occur after the last measurable concentration will be omitted (set to missing) in the
  derivation of pharmacokinetic parameters and from the individual subject plots.
- Individual's PK parameters reported as 'NC' (Not Calculable) or 'ND' (Not Determined) will be
  included in listings but omitted (set to missing) from figures, summaries and statistical
  analyses.

# 10.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion was defined as a participant has completed all periods of the study including the last visit or the last scheduled procedure (Follow-up) for each period as described in the protocol. |
| | Withdrawn subjects maybe replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |

## 10.6.3. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.6.4. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|------------|--------------------------------------------------|
| Imputation | No imputation will be performed for missing data |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. Laboratory Values (Healthy Volunteers)

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | ~/! | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

# 10.7.2. ECG (Healthy Volunteers)

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-----------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 [1] | |

#### NOTES:

# 10.7.3. Vital Signs (Healthy Volunteers)

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>1.</sup> Represent standard ECG values of PCI for HV studies

# 10.8. Appendix 8 - Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| AUC(0-24) | Area under the concentration-time curve from pre-dose to 24 hours |
| AUC(0-inf) | Area under the concentration-time curve from time zero (pre-dose) |
| AUC(0-IIII) | extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to |
| AUC(0-1) | |
| | 1 |
| PMI | |
| LLN | |
| LLQ | |
| | Medical Dictionary for Regulatory Activities |
| MG | Milligrams |
| msec | Milliseconds |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| ULN | Upper Limit of Normal |
| SOP | Standard Operation Procedure |
| t1/2 | Terminal half-life |
| Tmax | |
| | Ÿ |
| BMI BP CI Cmax CSR CVb CVw ECG eCRF GSK HR hrs IDSL IMMS LLN LLQ MedDRA MG msec PDMP PK QC QTcF RAP SAC SAE SAS SD ULN SOP t1/2 | last time of quantifiable concentration within a subject across all treatments Body mass index Blood pressure Confidence Interval Maximum observed concentration Clinical Study Report Coefficient of variation (Between) Coefficient of Variation (Within) Electrocardiogram Electronic Case Report Form GlaxoSmithKline Heart rate Hours Integrated Data Standards Library International Modules Management System Lower Limit of Normal Lower Limit of Quantification Medical Dictionary for Regulatory Activities Milligrams Milliseconds Protocol Deviation Management Plan Pharmacokinetic Quality Control Frederica's QT Interval Corrected for Heart Rate Reporting and Analysis Plan Statistical Analysis Complete Serious Adverse Event(s) Statistical Analysis Software Standard Deviation Procedure |
### 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

None

# Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

### 10.9. Appendix 9: List of Data Displays

### 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section Tables Figures | | |
|------------------------|------------------------|-----|
| Study Population | 1.1 to 1.14 | N/A |
| Safety | 2.1 to 2.34 N/A | |
| Pharmacokinetic | 3.1 to 3.8 3.1 to 3.10 | |
| Section | Listings | |
| ICH Listings | 1 to 70 | |
| Other Listings | N/A | |

### 10.9.2. Mock Example Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Indicate display is Non-Standard in the 'IDSL/TST ID / Example Shell' or 'Programming Notes' column.

### 10.9.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|---------------------------------------------|
| PR [1] | Primary Report (Part 1 only) |
| SAC [2] | Statistical Analysis Complete (Part 2 only) |

#### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

## 10.9.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | CP_ES1 | Summary of Subject Disposition (Part 1) | Completed or withdrawn and the reason for withdrawal. | PR [1] |
| 1.2. | Safety | ES4 | Summary of Subject Disposition at each period (Part 1) | Completed or withdrawn at each period. | PR [1] |
| 1.3. | Safety | CP_ES1 | Summary of Subject Disposition (Part 2) | Completed or withdrawn and the reason for withdrawal. | SAC [2] |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | The number (%) of Randomized or screening failure subjects as the screening status, and the reason for screening failure. | SAC [2] |
| Protoc | ol Deviation | | | | |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations (Part 1) | Data is from DV1 dataset. | PR [1] |
| 1.6. | Safety | DV1 | Summary of Important Protocol Deviations (Part 2) | Data is from DV1 dataset. | SAC [2] |
| Popula | tion Analysed | | | | |
| 1.7. | Safety | SP1 | Summary of Study Populations (Part 1) | Only PK population (Yes or No) is summarized. | PR [1] |
| 1.8. | Safety | SP1 | Summary of Study Populations (Part 2) | Only PK population (Yes or No) is summarized. | SAC [2] |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.9. | Safety | DM3 | Summary of Demographic Characteristics (Part 1) | | PR [1] |
| 1.10. | Safety | DM3 | Summary of Demographic Characteristics (Part 2) | | SAC [2] |
| 1.11. | Screened | DM11 | Summary of Age Ranges (Part 1) | <=17 years, 18-64 years, 65-84 years, >=85 years | PR [1] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.12. | Screened | DM11 | Summary of Age Ranges (Part 2) | <=17 years, 18-64 years, 65-84 years, >=85 years | SAC [2] |
| 1.13. | Safety | DM5 | Summary of Race and Racial Combinations (Part 1) | | PR [1] |
| 1.14. | Safety | DM5 | Summary of Race and Racial Combinations (Part 2) | | SAC [2] |

## 10.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 1) | | PR [1] |
| 2.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity (Part 1) | | PR [1] |
| 2.3. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term (Part 1) | | PR [1] |
| 2.4. | Safety | AE5A | Summary All Drug-Related Adverse Events by Maximum Intensity (Part 1) | | PR [1] |
| 2.5. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 2) | | SAC [2] |
| 2.6. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity (Part 2) | | SAC [2] |
| 2.7. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term (Part 2) | | SAC [2] |
| 2.8. | Safety | AE5A | Summary All Drug-Related Adverse Events by Maximum Intensity (Part 2) | | SAC [2] |
| Labora | tory: Chemistry | / | | | |
| 2.9. | Safety | LB1 | Summary of Chemistry (Part 1) | | PR [1] |
| 2.10. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 1) | | PR [1] |
| 2.11. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 1) | | PR [1] |
| 2.12. | Safety | LB1 | Summary of Chemistry (Part 2) | | SAC [2] |
| 2.13. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 2) | | SAC [2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 2) | | SAC [2] |
| Labora | tory: Hematolo | gy | | | |
| 2.15. | Safety | LB1 | Summary of Hematology (Part 1) | | PR [1] |
| 2.16. | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 1) | | PR [1] |
| 2.17. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 1) | | PR [1] |
| 2.18. | Safety | LB1 | Summary of Hematology (Part 2) | | SAC [2] |
| 2.19. | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 2) | | SAC [2] |
| 2.20. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 2) | | SAC [2] |
| Labora | tory: Urinalysis | 5 | | | |
| 2.21. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 1) | | PR [1] |
| 2.22. | Safety | LB1 | Summary of Urinalysis Data (Specific Gravity and pH) (Part 1) | | PR [1] |
| 2.23. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 2) | | SAC [2] |
| 2.24. | Safety | LB1 | Summary of Urinalysis Data (Specific Gravity and pH) (Part 2) | | SAC [2] |
| ECG | | | | | |
| 2.25. | Safety | EG1 | Summary of ECG Findings (Part 1) | | PR [1] |
| 2.26. | Safety | EG2 | Summary of ECG Value (Part 1) | | PR [1] |
| 2.27. | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 1) | | PR [1] |
| 2.28. | Safety | EG1 | Summary of ECG Findings (Part 2) | | SAC [2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.29. | Safety | EG2 | Summary of ECG Value (Part 2) | | SAC [2] |
| 2.30. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit (Part 2) | | SAC [2] |
| Vital Si | gns | | | | • |
| 2.31. | Safety | VS1 | Summary of Vital Signs (Part 1) | | PR [1] |
| 2.32. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 1) | | PR [1] |
| 2.33. | Safety | VS1 | Summary of Vital Signs (Part 2) | | SAC [2] |
| 2.34. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 2) | | SAC [2] |

### 10.9.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part 1 | | | | | |
| 3.1. | PK | PK01: pkct1 | Summary of GSK1325756 Blood Concentration (Part 1) | | PR [1] |
| 3.2. | PK | PK03: pkpt1 | Summary of GSK1325756 Pharmacokinetic Parameters (non-transformed) (Part 1) | | PR [1] |
| 3.3. | PK | PK05: pkpt3 | Summary of GSK1325756 Pharmacokinetic Parameters (loge-transformed) (Part 1) | | PR [1] |
| 3.4. | PK | Study Specific (PK_T1) | Analysis of Power Model Analysis for GSK1325756 Dose Proportionality of Pharmacokinetic Parameters (AUC(0-t), Cmax) (Part 1) | Parameter, Effect, n, Point estimate of Slope, SE, 90% CI | PR [1] |
| Part 2 | | | | | |
| 3.5. | PK | PK01: pkct1 | Summary of GSK1325756 Blood Concentration (Part 2) | | SAC [2] |
| 3.6. | PK | PK03: pkpt1 | Summary of GSK1325756 Pharmacokinetic Parameters (non-transformed) (Part 2) | | SAC [2] |
| 3.7. | PK | PK05: pkpt3 | Summary of GSK1325756 Pharmacokinetic Parameters (loge-transformed) (Part 2) | | SAC [2] |
| 3.8. | PK | Study Specific (PK_T2) | Analysis of food effect for Pharmacokinetic Parameters (AUC(0-t), Cmax) (Part 2) | n, Geometric mean of Fasted and Fed, ratio (Fasted/Fed), 90% Cl and CVw(%) | SAC [2] |

## 10.9.7. Pharmacokinetic Figures

| Pharm | acokinetic: Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part 1 | <u> </u> | | | , | |
| 3.1. | PK | PK16b: pkcf1x | Individual GSK1325756 Blood Concentration-Time Plots by Subject (Part 1) | By Subject (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | PR [1] |
| 3.2. | PK | PK24: pkcf6 | Individual GSK1325756 Blood Concentration-Time Plots by treatment (Part 1) | By Treatment (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | PR [1] |
| 3.3. | PK | Study Specific<br>(PK_F1) | Mean (+SD) GSK1325756 Blood Concentration-Time Plots (Part 1) | Unit of x-axis is Hours | PR [1] |
| 3.4. | PK | PK18: pkcf3 | Median GSK1325756 Blood Concentration-Time Plots (Part 1) | Unit of x-axis is Hours | PR [1] |
| 3.5. | PK | PK28 | Plot of GSK1325756 Treatment and PK Parameters (AUC (0-t), Cmax) (Part 1) | | PR [1] |
| Part 2 | | | | | |
| 3.6. | PK | PK16b: pkcf1x | Individual GSK1325756 Blood Concentration-Time Plots by Subject (Part 2) | By Subject (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | SAC [2] |
| 3.7. | PK | PK24: pkcf6 | Individual GSK1325756 P Blood Concentration-Time Plots by Treatment (Part 2) | By Treatment (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | SAC [2] |
| 3.8. | PK | Study Specifics (PK_F1) | Mean (+SD) GSK1325756 Blood Concentration-Time Plots (Part 2) | Unit of x-axis is Hours | SAC [2] |
| 3.9. | PK | PK18: pkcf3 | Median GSK1325756 Blood Concentration-Time Plots (Part 2) | Unit of x-axis is Hours | SAC [2] |

| Pha | Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|---|
| No | <b>o</b> . | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10 | ). | PK | PK28 | Plot of GSK1325756 Treatment and PK Parameters (AUC(0-t), Cmax) (Part 2) | | SAC [2] |

## 10.9.8. ICH Listings

Note: 'Inv.' in the standard displays will be replaced to 'Centre'.

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screening<br>Failure | ES7 | Listing of Reasons for Screen Failure | | PR [1] |
| 2. | Safety | CP-ES10x | Listing of Reasons for Study Withdrawal (Part 1) | | PR [1] |
| 3. | Safety | CP-ES10x | Listing of Reasons for Study Withdrawal (Part 2) | | SAC [2] |
| 4. | Safety | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken (Part 1) | | PR [1] |
| 5. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 1) | | PR [1] |
| 6. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 2) | | SAC [2] |
| Protoc | ol Deviations | | | | |
| 7. | Safety | DV2 | Listing of Important Protocol Deviations (Part 1) | Column for Treatment Sequence/Period of Protocol deviation will be displayed after Centre./Subj. Period day will be displayed in the same column of Date of Deviation/Study day. | PR [1] |
| 8. | Safety | DV2 | Listing of Important Protocol Deviations (Part 2) | | SAC [2] |
| 9. | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [2] |
| Popula | tions Analysed | | | | |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10. | Safety | Study Specifics (POP_L1) | Listing of Subjects Excluded from PK Population (Part 1) | | PR [1] |
| 11. | Safety | Study Specifics (POP_L1) | Listing of Subjects Excluded from PK Population (Part 2) | SAC [2] | |
| Demog | raphic and Bas | eline Characteris | tics | | • |
| 12. | Safety | DM4 | Listing of Demographic Characteristics (Part 1) | "Age at Screening" is added. | PR [1] |
| 13. | Safety | DM4 | Listing of Demographic Characteristics (Part 2) | "Age at Screening" is added. | SAC [2] |
| 14. | Screening<br>Failure | DM4 | Listing of Demographic Characteristics for Screening Failure Subjects | | SAC [2] |
| 15. | Safety | DM10 | Listing of Race (Part 1) | Listing of Race (Part 1) | |
| 16. | Safety | DM10 | Listing of Race (Part 2) | Listing of Race (Part 2) | |
| 17. | Screening<br>Failure | DM10 | Listing of Race for Screening Failure Subjects | Treatment is not needed to display. | SAC [2] |
| Medica | Conditions ar | d Concomitant M | edications | | |
| 18. | Screened | MH3 | Listing of Medical Conditions | | PR [1] |
| 19. | Safety | CM5 | Listing of Concomitant Medications (Part 1) | | PR [1] |
| 20. | Safety | CM5 | Listing of Concomitant Medications (Part 2) | | SAC [2] |
| Exposu | ire and Treatmo | ent Compliance | | | |
| 21. | Safety | EX4 | Listing of Exposure Data (Part 1) | | PR [1] |
| 22. | Safety | EX4 | Listing of Exposure Data (Part 2) | | SAC [2] |
| Meal | | | | | |
| 23. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days (Part 1) | | PR [1] |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days (Part 2) | | SAC [2] |
| Advers | e Events | | | | • |
| 25. | Safety | AE9CP | Listing of All Adverse Events (Part 1) | | SAC [1] |
| 26. | Safety | AE9CP | Listing of All Adverse Events (Part 2) | | SAC [2] |
| 27. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 1) | | PR [1] |
| 28. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 2) | | SAC [2] |
| 29. | Screened | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | SAC [2] | |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 30. | Safety | AE9CP | Listing of Serious Adverse Events (Part 1) | | PR [1] |
| 31. | Safety | AE9CP | Listing of Serious Adverse Events (Part 2) | | SAC [2] |
| 32. | Screening<br>Failure | AE9CP | Listing of Serious Adverse Events for Screening Failure Subject | Treatment is not needed to display. | SAC [2] |
| 33. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 1) | | PR [1] |
| 34. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 2) | | SAC [2] |
| Labora | tory (Chemistry | y Data) | | | |
| 35. | Safety | CP_LB6 | Listing of All Chemistry Data (Part 1) | Change from baseline is included. | PR [1] |
| 36. | Safety | CP_LB6 | Listing of All Chemistry Data (Part 2) | Change from baseline is included. | SAC [2] |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 37. | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 38. | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | SAC [2] | |
| Labora | tory (Hematolo | gy Data) | | | |
| 39. | Safety | CP_LB6 | Listing of All Hematology Data (Part 1) | Change from baseline is included. | PR [1] |
| 40. | Safety | CP_LB6 | Listing of All Hematology Data (Part 2) | Change from baseline is included. | SAC [2] |
| 41. | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 42. | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Labora | tory (Urinalysis | Data) | | | |
| 43. | Safety | UR2b | Listing of All Urinalysis Dipstick Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 1) | Time will be displayed after 'Date'. | PR [1] |
| 44. | Safety | CP_LB6 | Listing of Urinalysis Data (Gravity and pH) (Part 1) | | PR [1] |
| 45. | Safety | UR2b | Listing of All Urinalysis Dipstick Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 2) | Time will be displayed after 'Date'. | SAC [2] |
| 46. | Safety | CP_LB6 | Listing of Urinalysis Data (Gravity and pH) (Part 2) | | SAC [2] |
| Hepato | biliary (Liver) | | | | |
| 47. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 1) | Column for Treatment/Period will be displayed after the column for Age/Sex/Race Detail. | PR [1] |
| 48. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 2) | | SAC [2] |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 49. | Safety | МН3 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part 1) | | PR [1] |
| 50. | Safety | МН3 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part 2) | | SAC [2] |
| 51. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 1) | | |
| 52. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 2) | SAC [2] | |
| ECG | | | | • | |
| 53. | Safety | CP_EG4 | Listing of All ECG Values (Part 1) | | PR [1] |
| 54. | Safety | CP_EG4 | Listing of All ECG Values (Part 2) | | SAC [2] |
| 55. | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 1) | | PR [1] |
| 56. | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 2) | | SAC [2] |
| 57. | Safety | CP_EG6 | Listing of ECG Findings (Part 1) | | PR [1] |
| 58. | Safety | CP_EG6 | Listing of ECG Findings (Part 2) | | SAC [2] |
| 59. | Safety | CP_EG4 | Listing of All ECG Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 60. | Safety | CP_EG4 | Listing of All ECG Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Vital Si | gns | | | • | • |
| 61. | Safety | CP_VS5 | Listing of All Vital Signs (Part 1) | Change from baseline is included. | PR [1] |
| 62. | Safety | CP_VS5 | Listing of All Vital Signs (Part 2) | Change from baseline is included. | SAC [2] |
| 63. | Safety | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 64. | Safety | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Others | | | | | |
| 65. | Safety | Study Specifics (SAFE_L1) | Listing of Ophthalmic examinations (Part 1) | | PR [1] |
| 66. | Safety | Study Specifics (SAFE_L1) | Listing of Ophthalmic examinations (Part 2) | | SAC [2] |
| PK | | | | | |
| 67. | PK | PK08: pkcl1x | Listing of GSK1325756 Blood Concentration (Part 1) | | PR [1] |
| 68. | PK | PK08: pkcl1x | Listing of GSK1325756 Blood Concentration (Part 2) | | SAC [2] |
| 69. | PK | Study Specifics (PK_L1) | Listing of GSK1325756 Pharmacokinetic Parameters (Part 1) | | PR [1] |
| 70. | PK | Study Specifics (PK_L1) | Listing of GSK1325756 Pharmacokinetic Parameters (Part 2) | | SAC [2] |

### 10.10. Appendix 10: Example Mock Shells for Data Displays

### 10.10.1. Study population

Example CP\_ES1 (XO studies)

Protocol: GSK123456
Population: xxxxx


## Table x.x

| | Tota<br>(N=1 | al<br>100) |
|-----------------------------------------|--------------|------------|
| Completion Status | | |
| Completed | 50 | (50%) |
| Withdrawn | 50 | (50%) |
| Primary*/subreason^ for withdrawal | | |
| Adverse event | 10 | (10%) |
| Elevated ALT levels | 2 | (2%) |
| Severe vomiting | 5 | (5%) |
| Lack of efficacy | 0 | |
| Protocol deviation | 0 | |
| Subject reached stopping criteria | 10 | (10%) |
| CD4 levels below continuation threshold | 10 | (10%) |
| Study closed/terminated | 0 | |
| Lost to follow-up | 0 | |
| Investigator discretion | 0 | |
| Withdrew consent | 30 | (30%) |
| Burden of procedures | 10 | (10%) |
| Pursue alternative treatment | 20 | (20%) |
| Other | 0 | |

206817

Example: ES4


Population: xxxxx

## Table x.x

| Phase | | Not Randomized (N=10) | Placebo<br>(N=100) | Curitol<br>10mg<br>(N=100) |
|---|---|---|---|---|
| Screening | Entered<br>Completed | 10(100%)<br>0 | 100 (100%)<br>100 (100%) | 100 (100%)<br>100 (100%) |
| | Withdrawn | 10 (100%) | 0 | 0 |
| Double blind | Entered | | 100 (100%) | 100 (100%) |
| | Completed | | 50 (50%) | 50 (50%) |
| | Withdrawn | | 50 (50%) | 50 (50%) |
| Follow-up | Entered | | 50 (50%) | 50 (50%) |
| | Completed | | 50 (50%) | 50 (50%) |
| | Withdrawn | | 0 | 0 |

206817

Example: ES6 (SF for CONSORT)

Population: xxxxx

#### 

| | Screened<br>Subjects<br>(N=100) |
|---|---|
| Screening Status | |
| ENROLLED | 50 (50%) |
| FAILED | 50 (50%) |
| Reason(s) for Failure | |
| DID NOT MEED INCLUSION/EXCLUSION CRITERIA | 25 (25%) |
| STUDY CLOSED/TERMINATED | 5 (5%) |
| PHYSICIAN DECISION | 10 (10%) |
| PROTOCOL DEVIATION | 10 (10%) |

206817

Example: CP\_ES10x Protocol: GSK123456


Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre<br>ID/<br>Subj. | Treatment<br>Sequence/<br>Period of<br>Withdrawal | Last<br>Treatment<br>Before<br>Withdrawal | Date of Withdrawal/ Study Day of Withdrawal/ Period Day of Withdrawal | Primary Reason<br>for Withdrawal | Subreason for<br>Withdrawal | Date of Last<br>Contact/<br>Study Day of<br>Last Contact |
|---|---|---|---|---|---|---|
| xxxxxx/ | PAB/ | A | DDMMMYYYY/ | Adverse Event | Elevated ALT levels | DDMMMYYYY/ |
| XXX | Period 1 | | xx/ | | | X |
| | | | X | | | |
| xxxxxx/ | BPC/ | В | DDMMMYYYY/ | | | DDMMMYYYY/ |
| XXX | Period 2 | | x/ | | | X |
| | | | X | | | |

206817

Example: ES7 (for SF) Protocol: GSK123456


Population: xxxxx

#### 

| Centre ID/ | Date of<br>Screen<br>Failure | Reason Term(s) for Screen Failure |
|---|---|---|
| Subj. | | <u> </u> |
| XXXXXX/ | DDMMMYYYY | DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| XXX | | |
| xxxxxx/<br>xxx | DDMMMYYYY | PHYSICIAN DECISION<br>DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| xxxxxx/<br>xxx | DDMMMYYYY | DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| | DDMMMYYYY | PHYSICIAN DECISION |

206817

Example: BL2 (for XO studies)


Population: xxxxx Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID | Subj. | Sequence/<br>Treatment<br>when Blind<br>broken | Date<br>Blind<br>Broken | Time<br>Blind<br>Broken | Study<br>Day | Period<br>Day | Reason |
|---|---|---|---|---|---|---|---|
| xxxxx | xxxx | PBC/<br>Treatment A | DDMMMYYYY | hh:ss | xx | X | Other: PT REQUESTED TO KNOW<br>FOR MEDICAL REASONS |
| xxxxx | XXXX | APC/<br>Treatment C | DDMMMYYYY | hh:ss | XX | XX | Medical Emergency |

206817

Example: TA2 (for XO studies)

Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

Country: Canada
Centre ID: PPD
Investigator: PPD

| Subject<br>ID | Randomization<br>Number | Randomization Date | Period | Randomization<br>Treatment | Actual Treatment | Deviation |
|---|---|---|---|---|---|---|
| PPD | | 01JAN08 | 1 | Curital 10mg | Curital 10mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Placebo | No treatment | Y |
| | | | 4 | Curital 20mg | No treatment | Y |
| | | 03JAN08 | 1 | Curital 20mg | Curital 20mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Curital 10mg | Curital 10mg | |
| | | | 4 | Placebo | Placebo | |
| | | 01.777.00 | 1 | <b>7</b> 1 | D1 1 | |
| | | 01FEB08 | 1 | Placebo | Placebo | |
| | | | 2 | Curital 10mg | Curital 10mg | |
| | | | 3 | Placebo | Placebo | |
| | | | 4 | Curital 20mg | Curital 10mg | Y |
| | | 15FEB08 | 1 | Curital 10mg | Curital 10mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Placebo | Placebo | |
| | | | 4 | Curital 10mg | Curital 20mg | Y |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: IE4 (for XO studies)


Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID | Subj. | Treatment sequence | Туре | Criterion |
|---|---|---|---|---|
| xxxxxx | XXX | APC | INCLUSION | Is the subject 18 years of age or older? |
| xxxxx | XXX | PAB | EXCLUSION | Has the subject had an asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to Visit 1? |

206817

Example: DV1


Population: xxxxx

#### 

| Category/Coded Term | | tal<br>=200) |
|---|---|---|
| Any important protocol deviations | 60 | (30%) |
| Informed consent WRONG INFORMED CONSENT/ASSENT VERSION SIGNED | | (5%)<br>(5%) |
| Eligibility criteria not met | 14 | (7%) |
| Not withdrawn after developing withdrawal criteria<br>Not discontinued from study treatment<br>Not withdrawn from study | 10 | (9%)<br>(5%)<br>(4%) |
| EXCLUDED MEDICATION, VACCINE OR DEVICE MEDICATION, EXCLUDED BY THE PROTOCOL, WAS ADMINISTERED | | (2%)<br>(2%) |
| Assessment or time point completion OUT OF WINDOW EFFICACY ASSESSMENT | | (1%)<br>(1%) |
| WRONG STUDY TREATMENT/ADMINISTRATION/DOSE<br>STUDY TREATMENT NOT ADMINISTERED PER PROTOCOL<br>EXPIRED STUDY TREATMET ADMINISTERED | 2 | (2%)<br>(1%)<br>(1%) |
| Failure to report SAFETY EVENTS PER Protocol<br>SAE NOT REPORTED WITHIN THE EXPECTED TIME FRAME<br>LIVER FUNCTION ABNORMALITIES PER PROTOCOL | 4 | (5%)<br>(2%)<br>(2%) |

Example: DV2


Population: xxxxx

#### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| | | | | Deviation R | Requires Excl | usion from |
|---|---|---|---|---|---|---|
| Site Id./ | Date of<br>Deviation/ | Category/<br>Coded Term | Term | Intent to Treat Population | Safety<br>Population | Per<br>Protocol<br>Population |
| PPD | 28 | ILURE TO REPORT SAFETY EVENTS PER PROTOCOL / SAE NOT REPORTED WITHIN THE EXPECTED TIME FRAME | SAE OF FEVER WITH SEVERE CHILLS REQUIRING IV HYDRATION WAS NOT REPORTED TO GSK WITHIN 24 HOURS. | | | |
| | 31 | ELIGIBILITY CRITERIA<br>NOT MET / ELIGIBILITY<br>CRITERIA NOT MET | SUBJECT SCREEN<br>FAILED BUT WAS<br>RANDOMIZED IN<br>ERROR. | | Y | Y |
| | PPD 1 | WRONG STUDY TREATMENT/ ADMINISTRATION/DOSE / STUDY TREATMENT NOT ADMINISTERED PER PROTOCOL | SUBJECT MISSED<br>WEEK 8<br>TREATMENT | | | |
| | 2<br>2 | WRONG STUDY TREATMENT/ ADMINISTRATION/DOSE / STUDY TREATMENT NOT ADMINISTERED PER PROTOCOL | INTERRUPTION OF IP FOR GREATER THAN 20 PERCENT OF TIME | | | Y |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: SP1


Population: xxxxx

#### 

| Population | No Treatment (N=50) | Placebo<br>(N=xxx) | Treatment 1 (N=200) | Treatment 2 (N=250) | Total<br>(N=500) |
|---|---|---|---|---|---|
| Screened | 50 (100%) | xx (xxx%) | 200 (100%) | 250 (100%) | 500 (100%) |
| Enrolled | 10 (20%) | xx (xxx%) | 200 (100%) | 250 (100%) | 460 (92%) |
| Randomized | 5 (10%) | xx (xx%) | 200 (100%) | 250 (100%) | 455 (91%) |
| Safety | | xx (xx%) | 195 (98%) | 245 (98%) | 440 (88%) |
| PK | | xx (xx%) | 200 (100%) | 250 (100%) | 455 (91%) |

206817


Example: POP\_L1
Protocol: GSK123456

Population: xxxxx (Randomised subjects)

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID/<br>Subj. | Treatment sequence | PK<br>population |
|---------------------|--------------------|------------------|
| xxxxxx/<br>xxx | ABC | Y |
| xxxxxx/<br>xxx | CBA | Y |
| xxxxxx/<br>xxx | BAC | Y |

USER ID: directory/program.sas DDMMMYYYY hh:mm


Example: DM3 (for XO studies)

Protocol: GSK123456
Population: xxxxx

## Table x.x

| | Total (N=100) |
|------------------------|----------------------|
| Sex | 100 |
| n<br>R | 100 |
| F<br>M | 50 (50%)<br>50 (50%) |
| Age (YEARS)[1] | |
| n | 100 |
| Mean | 50.0 |
| SD | 10.00 |
| Median | 50.0 |
| Min. | 18 |
| Max. | 65 |
| Age Group(YEARS)[1] | |
| <=18 | 5 (5%) |
| 19-64 | 50 (50%) |
| >=65 | 45 (45%) |
| Ethnicity | |
| n | 100 |
| HISPANIC OR LATINO | 10 (10%) |
| NOT HISPANIC OR LATINO | 90 (90%) |

Example: DM3 (continued) Protocol: GSK123456

Population: xxxxx


#### 

| | | Total |
|---------------------------------------|----|---------|
| | | (N=100) |
| Race Detail | | |
| AMERICAN INDIAN OR ALASKA NATIVE | 1 | ` ' |
| ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 3 | (3%) |
| ASIAN - EAST ASIAN HERITAGE | 4 | (4%) |
| ASIAN - JAPANESE HERITAGE | 3 | (3%) |
| ASIAN - SOUTH EAST ASIAN HERITAGE | 1 | (1%) |
| BLACK OR AFRICAN AMERICAN | 2 | (2%) |
| NATIVE HAWAIIAN OR OTHER PACIFIC | 59 | (59%) |
| ISLANDER | | |
| WHITE - ARABIC/NORTH AFRICAN HERITAGE | 26 | (26%) |
| WHITE - WHITE/CAUSASIAN/EUROPEAN | 1 | (1%) |
| HERITAGE | | |
| MIXED ASIAN RACE | 1 | (1%) |
| MIXED WHITE RACE | 1 | (1%) |
| ${\it MULTIPLE}$ | 1 | (1%) |
| Height (cm) | | |
| n | 1 | 00 |
| Mean | 1 | 50.0 |
| SD | | 10.00 |
| Median | | 50.0 |
| Min. | | 18 |
| Max. | | 65 |
| max. | | 0.5 |

Example: DM3 (continued)

Protocol: GSK123456
Population: xxxxx


#### 

| | Total |
|-------------|---------|
| | (N=100) |
| Weight (kg) | |
| n | 100 |
| Mean | 50.0 |
| SD | 10.00 |
| Median | 50.0 |
| Min. | 18 |
| Max. | 65 |

Options (units)

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: DM4 (for XO studies)


Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID/<br>Subj. | Treatment<br>Sequence | Partial<br>Date of<br>Birth | Age<br>(YEARS)<br>[1] | Sex | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Option (unit) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/<br>xxx | ABC | MMYYYY | xx | F | HISPANIC OR LATINO | xxx | xx | |
| xxxxxx/<br>xxx | BCA | MMYYYY | xx | М | NOT HISPANIC OR LATINO | XXX | xx | |
| xxxxxx/<br>xxx | CAB | ҮҮҮҮ | XX | М | NOT HISPANIC OR LATINO | XXX | XX | |

Example: DM5


Population: xxxxx

## Table x.x Xxxxxxxxxxxxxxxxxxxxxxxx

| | | | ment A<br>=XXX) | | tment B<br>=XXX) | | otal<br>=XXX) |
|---|---|---|---|---|---|---|---|
| Race | n | 100 | | 100 | | 200 | |
| | African American/African Heritage | 30 | (30%) | 30 | (30%) | 60 | (30%) |
| | American Indian or Alaskan Native | 0 | | 0 | | 0 | |
| | Asian | 15 | (15%) | 15 | (15%) | 30 | (15%) |
| | Central/South Asian Heritage | 3 | (3%) | 3 | (3%) | 6 | (3%) |
| | Japanese/East Asian Heritage/South | 11 | (11%) | 11 | (11%) | 22 | (11%) |
| | East Asian Heritage | | | | | | |
| | Mixed Asian Heritage | 1 | (1%) | 1 | (1%) | 2 | (1%) |
| | Native Hawaiian or other Pacific | 10 | (10%) | 10 | (10%) | 20 | (10%) |
| | Islander | | | | | | |
| | White | 35 | (35%) | 35 | (35%) | 70 | (35%) |
| | Native Hawaiian or other Pacific | 2 | (2%) | 2 | (2%) | 4 | (4%) |
| | Islander & American Indian or Alaskan | | | | | | |
| | Native | | | | | | |
| | White & African American/African | 3 | (3%) | 3 | (3%) | 6 | (3%) |
| | Heritage | | | | | | |
| | White & Asian | 5 | (5%) | 5 | (5%) | 10 | (5%) |

206817

Example: DM11


Population: xxxxx

## Table x.x

| | No Treatment (N=1) | Total (N=201) |
|---|---|---|
| Age Ranges [1] In utero Preterm newborn infants (gestational age <37 weeks) | 0<br>0 | 4 (2%)<br>2 (1%) |
| Newborns (0-27 days) | 0 | 6 (3%) |
| Infants and toddlers (28 days-23 months) | 0 | 8 (4%) |
| Children (2-11 years) | 0 | 6 (3%) |
| Adolescents (12-17 years) | 0 | 2 (1%) |
| Adult (18-64 years) | 0 | 118 (59%) |
| >=65-84 years | 0 | 52 (26%) |
| >=85 years | 1 (100%) | 3 (1%) |

206817


Example: DM10 (for XO studies)

Protocol: GSK123456
Population: xxxxx

### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre<br>ID | Subj. | Treatment sequence | Race | Race Detail |
|---|---|---|---|---|
| xxxxxx | XXX | ABC | BLACK OR AFRICAN AMERICAN | BLACK OR AFRICAN AMERICAN |
| | XXX | BCA | Mixed race | ASIAN - EAST ASIAN HERITAGE<br>ASIAN - JAPANESE HERITAGE |
| | XXX | CAB | WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE | WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE |
| | XXX | ABC | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE |
| xxxxxx | XXX | ABC | Mixed race | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAG<br>ASIAN - JAPANESE HERITAGE |
| | XXX | BCA | NATIVE HAWAIIAN OR OTHER PACIFIC<br>ISLANDER | NATIVE HAWAIIAN OR OTHER PACIFIC<br>ISLANDER |
| | XXX | CAB | BLACK OR AFRICAN AMERICAN | BLACK OR AFRICAN AMERICAN |
| | XXX | ABC | WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE | WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE |
| xxxxx | xxx | BCA<br>CAB | AMERICAN INDIAN OR ALASKA NATIVE<br>Mixed race | AMERICAN INDIAN OR ALASKA NATIVE<br>BLACK OR AFRICAN AMERICAN<br>WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE |

206817

Example: MH3


Population: xxxxx

| _In | V. | Subject | Treatment<br>Sequence | Classification | Condition | Status |
|---|---|---|---|---|---|---|
| PPD | | | AB | Hepatobiliary<br>Psychiatric | HEPATITIS A<br>PARANOIA COMBINED WITH MANIA. | Current<br>Past |
| | | | AB | Eye | ASTIGMATISM | Current |
| | | | ВА | Metabolism and nutrition | RICKETS | Current |
206817

Example: CM5

Population: xxxxx

Listing x.x

| Inv./<br>Subj./<br>Seq | Treat-<br>ment/<br>Period | ATC Level 1/<br>Ingredient/<br>Verbatim Text/<br>Indication | Dose/<br>Units/<br>Freq/<br>Route | Start<br>Date/Time<br>Study Day/<br>Period Day | Stop<br>Date/Time<br>Study Day/<br>Period Day | Started<br>Pre-<br>Trial? | Ongoing<br>Medi-<br>cation? |
|---|---|---|---|---|---|---|---|
| PPD<br>ABC | Tmt A/<br>Per 1 | <pre>Endocrine &amp; metabolic/ Fluticasone propionate/ FLIXOTIDE/</pre> | 2/<br>MG/<br>2XD/ | PPD<br>12:30/<br>15/ | | | Y |
| ADC | | Asthma | IH | 7 | | | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: EX4


Population: xxxxx

## Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre<br>ID | Subj. | Treatment | Start Date/ Start Time of Dose | Stop Date/<br>Stop Time<br>of Dose | Duration (days) | Dose | | Formulat ion/ | Freque<br>ncy | Cumulat ive Dose |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx | Treatment A | DDMMMYYYY/ hh:ss DDMMMYYYY/ | DDMMMYYYY/<br>hh:ss | xx<br>xx | xx | mg<br>mg | Tablet/<br>Oral<br>Tablet/ | 1xday<br>1xday | |
| | | Treatment C | hh:ss<br>DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Oral<br>Tablet/<br>Oral | 1xday | |
| | PPD | Placebo Treatment B | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | xx | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Treatment C | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Treatment A | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | xx | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Placebo<br>Treatment B | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_ML1x Protocol: GSK123456 Population: xxxxx


## Listing x.x Xxxxxxxxxxxxxxxxxxxx

| <pre>Cohort_<br/>(Optional)</pre> | Investigator OR Centre ID (Optional) | Subj. | Treatment | Meal type (Optional) | Period<br>(Optional)<br>/Visit | <u>Visit</u><br>Date | Dose<br>Time | Meal_Start_Time | Meal End Time (Optional) | Meal ended within 20 minutes of Meal Start Time (Optional) | Time from Start of Meal to Dosing (min) (Optional) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | PPD | | 50mg<br>GSK123456<br>25mg<br>GSK123456<br>10mg<br>GSK123456 | High-fat<br>breakfast<br>High-fat<br>breakfast<br>High-fat<br>breakfast | Period<br>2/Day 4<br>Period<br>2/Day 4<br>Period<br>2/Day 4 | PPD | | 7:30<br>7:28<br>7:27 | 7:41<br>7:42<br>7:35 | Y<br>Y<br>Y | 43<br>44<br>43 |
| 2 | | | 50mg<br>GSK123456<br>50mg<br>GSK123456<br>25mg<br>GSK123456<br>10mg<br>GSK123456 | High-fat<br>breakfast<br>High-fat<br>breakfast<br>High-fat<br>breakfast<br>High-fat<br>breakfast | Period<br>2/Day 4<br>Period<br>2/Day 4<br>Period<br>2/Day 4<br>Period<br>2/Day 4 | | 8:09<br>8:11<br>8:09<br>8:10 | 7:30 | 7:50<br>7:41<br>7:42<br>7:36 | N<br>Y<br>Y | 41<br>41<br>44<br>43 |

USER ID: directory/program.sas DDMMMYYYY hh:mm

## 10.10.2. Safety population

Example: AE1


Population: xxxxx

#### 

| System Organ Class | Placebo | Drug A | Drug B |
|----------------------------|----------|----------|----------|
| Preferred Term | (N=78) | (N=78) | (N=78) |
| ANY EVENT | 58 (74%) | 64 (82%) | 64 (85%) |
| Gastrointestinal disorders | | | |
| Any event | xx (xx%) | xx (xx%) | xx (xx%) |
| Dyspepsia | xx (xx%) | xx (xx%) | xx (xx%) |
| Nausea | xx (xx%) | xx (xx%) | xx (xx%) |
| Vomiting Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Constipation | xx (xx%) | xx (xx%) | xx (xx%) |
| Diarrhoea Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Toothache | xx (xx%) | xx (xx%) | xx (xx%) |
| Abdominal Pain Upper | xx (xx%) | xx (xx%) | xx (xx%) |
| Dry Mouth | xx (xx%) | xx (xx%) | xx (xx%) |
| Flatulence | xx (xx%) | xx (xx%) | xx (xx%) |
| Gastrointestinal Upset | xx (xx%) | xx (xx%) | xx (xx%) |
| Haemorrhoids | xx (xx%) | xx (xx%) | xx (xx%) |
| Loose Stools | xx (xx%) | xx (xx%) | xx (xx%) |
| Abdominal Pain Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Faecal Incontinence | xx (xx%) | xx (xx%) | xx (xx%) |
| Gastritis Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Lip Disorder Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Lip Dry | xx (xx%) | xx (xx%) | xx (xx%) |
| Stomach Discomfort | xx (xx%) | xx (xx%) | xx (xx%) |
| Nervous system disorders | | | |
| Any event | xx (xx%) | xx (xx%) | xx (xx%) |
| Headache | xx (xx%) | xx (xx%) | xx (xx%) |
| Dizziness | xx (xx%) | xx (xx%) | xx (xx%) |
| Extrapyramidal Disorder | xx (xx%) | xx (xx%) | xx (xx%) |

206817

Example: AE5A


Population: xxxxx

Table x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

Treatment: Treatment A (N=200)

| Quarters Quarter Q1 | | | | | | | | 40 DED 3 EE | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | | MILD | M | ODERATE | | SEVERE | 1 | MODERATE<br>/SEVERE | UN | IKNOWN | | Total |
| ANY EVENT | 30 | (15%) | 40 | (20%) | 40 | (20%) | 80 | (40%) | 1 | (<1%) | 151 | (76%) |
| Cardiovascular | | | | | | | | | | | | |
| Any Event | 20 | (10%) | 40 | (20%) | 40 | (20%) | 80 | (40%) | 0 | | 140 | (70%) |
| Hypertension | 0 | | 20 | (10%) | 20 | (10%) | 20 | (10%) | 0 | | 40 | (20%) |
| Syncope | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| Hypotension | 20 | (10%) | 0 | | 0 | | 40 | (20%) | 0 | | 60 | (30%) |
| Nervous system | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |
| disorders | | | | | | | | | | | | |
| Any Event | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |
| Dizziness | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |

206817

Example: LB1


Population: xxxxx

#### 

| | | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | N | Time | n | Mean | SD | Median | Min. | Max. |
| Trt A | 202 | Week 8 | 150 | 2.1 | 7.95 | 1 | -25 | 32 |
| | | Week 12 | 133 | 0.4 | 10.05 | 1 | -64 | 33 |
| | | Week 24 | 55 | -1.6 | 18.22 | 0 | -339 | 44 |
| Trt B | 220 | | | | | | _ | 32 |
| | | Week 12 | 133 | 0.4 | 10.05 | 1 | -64 | 33 |
| | | Week 24 | 55 | -1.6 | 18.22 | 0 | -339 | 44 |
| Trt A | 202 | Week 8 | 150 | -1.2 | 16.32 | 0 | -320 | 38 |
| | | Week 12 | 133 | 0.7 | 10.55 | 1 | -64 | 32 |
| | | Week 24 | 55 | -3.3 | 29.50 | 0 | -235 | 36 |
| Trt B | 220 | Week 8<br>Week 12<br>Week 24 | 150<br>133<br>55 | -1.2<br>0.7<br>-3.3 | 16.32<br>10.55<br>29.50 | 0<br>1<br>0 | -320<br>-64<br>-235 | 38<br>32<br>36 |
| | Trt A Trt B Trt A | Trt A 202 Trt B 220 Trt A 202 | Treatment N Time Trt A 202 Week 8 Week 12 Week 24 Trt B 220 Week 8 Week 12 Week 24 Trt A 202 Week 8 Week 12 Week 24 Trt B 220 Week 8 Week 12 Week 24 Trt B 220 Week 8 Week 12 Week 12 | Treatment N Time n Trt A 202 Week 8 12 133 Week 24 55 Trt B 220 Week 8 150 Week 12 133 Week 24 55 Trt A 202 Week 8 150 Week 24 55 Trt B 202 Week 8 150 Week 24 55 Trt B 220 Week 8 150 Week 24 55 | Treatment N Time n Mean Trt A 202 Week 8 | Treatment N Time n Mean SD Trt A 202 Week 8 Week 12 133 0.4 10.05 Week 24 55 -1.6 18.22 Trt B 220 Week 8 150 2.1 7.95 Week 12 133 0.4 10.05 Week 12 133 0.4 10.05 Week 24 55 -1.6 18.22 Trt A 202 Week 8 150 -1.2 16.32 Week 24 55 -3.3 29.50 Trt B 220 Week 8 150 -1.2 16.32 Week 24 55 -3.3 29.50 Trt B 220 Week 8 150 -1.2 16.32 Week 12 133 0.7 10.55 | Treatment N Time n Mean SD Median Trt A 202 Week 8 Week 8 Week 12 Week 24 150 2.1 7.95 1 Week 24 10.05 1 Week 24 10.0 | Treatment N Time n Mean SD Median Min. Trt A 202 Week 8 |

Example: LB4


Population: xxxxx

## Table x.x

Test= Alanine Aminotransferase (IU/L), Treatment=Treatment A

| | | | | | | | Time Pe | riod V | alue | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Planned<br>Time | N | n | Baseline<br>Value | High | 1 | Norn | nal | Low | | Tota | al |
| Week 1 | 100 | 100 | High<br>Normal<br>Low<br>Total | 0<br>10<br>0<br>10 | (10%) | 1<br>84<br>0<br>85 | (1%)<br>(84%)<br>(85%) | 3<br>2<br>0<br>5 | (3%)<br>(2%)<br>(5%) | 4<br>96<br>0<br>100 | (4%)<br>(96%)<br>(100%) |
| Week 4 | 100 | 100 | High<br>Normal<br>Low<br>Total | 0<br>10<br>0<br>10 | (10%)<br>(10%) | 1<br>84<br>0<br>85 | (1%)<br>(84%)<br>(85%) | 3<br>2<br>0<br>5 | (3%)<br>(2%)<br>(5%) | 4<br>96<br>0<br>100 | (4%)<br>(96%)<br>(100%) |
| Worst Case<br>Post-Baseline | 100 | 100 | High | 0 | | 1 | (1%) | 3 | (3%) | 4 | (4%) |
| | | | Normal<br>Low<br>Total | 10<br>0<br>10 | (10%)<br>(10%) | 84<br>0<br>85 | (84%)<br>(85%) | 2<br>0<br>5 | (2%)<br>(5%) | 96<br>0<br>100 | (96%)<br>(100%) |

Example: UR3b


Population: xxxxx

#### 

| | Period/Planned | | _ | atment A<br>N=100) | _ | atment B<br>N=100) |
|---|---|---|---|---|---|---|
| Test | Relative Time | Result | | | | |
| Urine General<br>Dipstick | SCREENING/<br>SCREENING | Positive | 30 | (30%) | 60 | (60%) |
| | | Negative | 40 | (40%) | 30 | (30%) |
| | | No Result | 30 | (30%) | 10 | (10%) |
| | PERIOD 1/DAY 1 | Positive | 40 | (40%) | 50 | (50%) |
| | | Negative | 30 | (30%) | 40 | (40%) |
| | | No Result | 30 | (30%) | 10 | (10%) |
| Urine Occult Blood (Dipstick) | SCREENING/<br>SCREENING | None | 40 | (40%) | 40 | (40%) |
| | | Trace | 25 | (25%) | 25 | (25%) |
| | | 1+ | 10 | (10%) | 15 | (15%) |
| | | 2+ | 0 | | 0 | |
| | | 3+ | 0 | | 0 | |
| | | No Result | 10 | (10%) | 20 | (20%) |
| | PERIOD 1/DAY 1 | None | 40 | (40%) | 40 | (40%) |
| | | Trace | 30 | (30%) | 30 | (30%) |
| | | 1+<br>2+ | 5<br>2 | (5응)<br>(2응) | 5<br>4 | (5응)<br>(4응) |
| | | 3+ | 0 | | 0 | |

206817

Example: EG1


Population: xxxxx

## Table x.x

| | | Treatment A Treatment (N=157) (N=160 | | atment B<br>(N=160) |
|---|---|---|---|---|
| Time Period 1 | | | | |
| n | 156 | | 160 | |
| Normal | 81 | (52%) | 90 | (56%) |
| Abnormal, not clinically significant | 75 | (48%) | 69 | (43%) |
| Abnormal, clinically significant | 0 | , , | 1 | (<1%) |
| Time Period 2 | | | | |
| n | 117 | | 123 | |
| Normal | 50 | (43%) | 67 | (54%) |
| Abnormal, not clinically significant | 64 | (55%) | 55 | (45%) |
| Abnormal, clinically significant | 2 | (2%) | 1 | (<1%) |
| n | 117 | | 122 | |
| Clinically significant change from baseline | 2 | (2%) | 1 | (<1%) |
| Not a clinically significant change | 115 | (98%) | | (>99%) |
| Not applicable | 0 | | 0 | |

206817

Example: EG1 (continued)


Population: xxxxx

#### 

| | | atment A<br>(N=157) | | atment B<br>(N=160) |
|---|---|---|---|---|
| Any time post-baseline | | | | |
| n | 117 | | 123 | |
| Normal | 50 | (43%) | 67 | (54%) |
| Abnormal, not clinically significant | 65 | (56%) | 55 | (45%) |
| Abnormal, clinically significant | 2 | (2%) | 1 | (<1%) |
| No result (not available) | 0 | | 0 | |
| n | 117 | | 122 | |
| Clinically significant change from baseline | 2 | (2%) | 1 | (<1%) |
| Not a clinically significant change | 115 | (98%) | 121 | (>99%) |
| Not applicable | 0 | | 0 | |

206817

Example: EG2


Population: xxxxx

## Table x.x

### Planned Relative

Time

| | Treatment | N | | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Heart Rate | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (bpm) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| PR Interval | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (msec) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |

206817

Example: VS1


Population: xxxxx

#### 

Planned Relative Time

| | Treatment | N | | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Systolic BP | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (mmHg) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| Diastolic BP | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (mmHq) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| . 5. | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |

Example: AE7


Population: xxxxx

## Listing x.x

#### 

| System Organ Class Preferred Term | Treatment | No.<br>with<br>Event | Unique Subject Id. |
|---|---|---|---|
| Gastrointestinal disorders<br>Dyspepsia | Placebo | 9 | PPD |
| | Treatment A | 11 | |
| | Treatment B | 4 | |
| Nausea | Placebo | 6 | |
| | Treatment A | 8 | |
| | Treatment B | 4 | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: AE9CP


Population: xxxxx

### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Site Id./ Unique Subject Id./ /Arm | Treatme nt/ | Age(YEARS)/<br>Sex/<br>Race<br>Detail/<br>Weight<br>(kg) | System Organ Class/<br>Preferred Term/<br>VERBATIM TEXT | Outcome/<br>Onset Datetime/<br>Datetime of<br>Resolution/<br>Duration | Time since Study 1st Dose/ Period 1st Dose/ Last Dose | Maximum Intensity/ Maximum Grade/ Serious/ Withdrawal | Frequency/ Action Taken/ Relation to Study Treatment |
|---|---|---|---|---|---|---|---|
| AB-BA-<br>BA | Tmt A/<br>Per 1 | 57/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE/<br>62.0 | Gastrointestinal<br>Disorders/<br>Internal spasm/<br>ENTERO - SPASM | RECOVERED/RESOLVE<br>D/<br>PPD | 31d 26h 4m/<br>31d 26h 4m/<br>-29d 7h 0m | MILD/<br>1<br>N/<br>N | INTERMITTENT/<br>DOSE REDUCED/<br>Y |
| | Tmt B/<br>Per 2 | 65/<br>M/<br>MIXED WHITE<br>RACE/<br>75.0 | Musculoskeletal and<br>connective tissue<br>disorders/<br>Arthralgia/<br>PAIN IN RIGHT<br>SHOULDER | RECOVERED/RESOLVE<br>D/<br>PPD | 83d 1h 12m/<br>83d 1h 12m/<br>-17d 2h 5m | MODERATE/<br>2/<br>N/<br>N | SINGLE EVENT/<br>DOSE NOT<br>CHANGED/<br>N |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: AE2

Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| System Organ Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system disorders | Lymphadenopathy | ENLARGED LYMPH NODE |
| Cardiac disorders | Palpitations | CLOGGED EARS WITH EAR WAX |
| | Ear pain | EARACHES IN BOTH EARS |
| | | RIGHT EAR PAIN |
| | Tinnitus | RINGING IN RIGHT EAR |
| Eye disorders | Asthenopia | TIRED EYES |
| | Conjunctivitis | BILATERAL ACUTE CONJUNCTIVITIS |
| | | CONJUNCTIVITIS |
| | Dry eye nos | DRY EYES |
| | Eye redness | REDDENED EYES |
| | Vision blurred | BLURRED VISION |
| | | BLURRY VISION |
| | | WORSENING OF BLURRED VISION |
| Gastrointestinal disorders | Abdominal pain nos | ABDOMEN PAIN |
| | Abdominal pain upper | MID-EPIGASTRIC AREA PAIN |
| | | STOMACH ACHE |
| | • | |

206817

Example: CP\_LB6
Protocol: GSK123456


### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./<br>Subj./ | Age(y)/<br>Sex/ | Treat-<br>ment/ | Lab test | Planned<br>Relative | | Study<br>Day/<br>Period | Co | nverted Data | Fl | ag[1 | ] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Seq | Race | Period | (units) | Time | Date/Time | Day | Value | Normal Range | NR | CI | BL |
| PPD | 63/ | Trt A/ | Alk Phos | Screening | PPD<br>12:05 | -1/-1 | 64.00 | 32.0- 92.0 | | | |
| | Male/ | Per 1 | (0, 2) | Week 12 | PPD<br>13:45 | 85/85 | 84.00 | 32.0- 92.0 | | | |
| | White | | | | 10.10 | | | | | | |
| | | | ALT (U/L) | Screening | PPD<br>13:32 | -1/-1 | 29.00 | 10.0- 40.0 | | | |
| | | | | Week 12 | PPD<br>09:55 | 85/85 | 70.00 | 10.0- 40.0 | Н | Н | Н |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: UR2b


Population: xxxxx

#### 

| Inv. | Subject | Treatment | Period | Visit | Sample Date | Study<br>Day | Period<br>Day | Urinalysis<br>Test | Result |
|---|---|---|---|---|---|---|---|---|---|
| PPD | | Trt A | 1 | 1 | PPD | 1 | 1 | Blood | ++ or 2+ |
| | | Trt B | 2 | 8 | | 137 | 1 | Blood | + or 1+ |
| | | Trt B | 1 | 1 | | 1 | 1 | Blood | + or 1+ |
| | | Trt A | 2 | 8 | | 137 | 1 | Protein | +++ or 3+<br>+ or 1+ |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: LIVER5 Protocol: GSK123456


### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

Treatment: Treatment A

| S | Site Id./<br>Jnique Subject | Age(YEARS)/<br>Sex/ | Maximum Status of<br>the Liver Event | Date First<br>Detected/<br>Study Day | Time<br>Since<br>First<br>Dose<br>(days) | Time<br>Since<br>Last<br>Dose<br>(days) | Restart/Re-<br>challenge After<br>Stopping Criteria<br>Was Met | Resolved?/<br>Date<br>resolved |
|---|---|---|---|---|---|---|---|---|
| PF | PD | 63/<br>M/<br>WHITE -<br>WHITE/CAUSAS<br>IAN/EUROPEAN<br>HERITAGE | LIVER MONITORING<br>CRITERIA | <b>PPD</b> 101 | 101 | 1 | N | Y/<br>2010-02-19 |
| | | 61/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | LIVER EVENT<br>STOPPING CRITERIA | <b>PPD</b> 68 | 68 | 1 | Y | Y/<br>2010-04-10 |
| | | I | LIVER EVENT<br>STOPPING CRITERIA | <b>PPD</b> 134 | 134 | 7 | N | N |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: SU2


Population: xxxxx

#### 

| Treat-<br>ment | Inv./<br>Subj. | Visit | Study<br>Day | Assess-<br>ment<br>Date | Smoking<br>History | Cur-rently<br>Smoke | Last<br>Smoked | Smoked<br>Since<br>Last<br>Visit | Days<br>Smoked<br>Since<br>Last<br>Visit | Years<br>Smoked | Ciga-<br>rettes<br>/day | Smoki<br>ng<br>Pack<br>Years |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trt A | PPD | Visit 1 | 1 | PPD | Never | No | | No | Zero | | | |
| | | Visit 1 | 1 | | Current | Yes | | Yes | A few | 5 | 20 | 5 |
| Trt B | | Visit 1 | 1 | | Former | No | 31DEC1<br>990 | No | Zero | 18 | 30 | 27 |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_EG4
Protocol: GSK123456


#### Listing x.x xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| | | | | | Actual | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Inv./ | Age | Treat- Planned | | Study | Relative | Heart | PR | QRS | RR | QΤ | | |
| Subj. | (y)/ | ment/ Relative | ECG | Day | Time | Rate | Int. | Dur. | Int. | Int. | QTcB | QTcF |
| /Seq. | Sex/ | Period Time | Date/Time | /Period | (optional) | (bpm) | (msec | (mse | (msec) | (msec) | (msec) | (msec) |
| | Race | | | Day | | | ) | C) | | | | |
| PPD | 65/ | Trt A/ Time 1 | PPD | 1/1 | -30m | 60 L | 150 | 350 | 750 | 450 | 520 | 495 |
| | White/ | Per 1 | 14:00 | | | | | | | | | |
| /AB | Female | | | | | | | | | | | |
| | | Time 2 | PPD | 7/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 15:00 | , | | | | | | | | |
| | | Trt B/ Time 1 | PPD | 14/1 | -30m | 80 | 150 | 390 | 750 | 450 | 520 | 495 |
| | | Per 2 | 19:00 | ± 1/ ± | 3 0 III | 0.0 | 100 | Н | 700 | 100 | 020 | 130 |
| | | | PPD | 01/7 | 2 ( | 0.0 | 1 = 0 | | 750 | 450 | EOO | 4 O E |
| | | Time 2 | | 21/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 20:00 | | | | | | | | | |
| PPD | | , | DDD | | | | | | | | | |
| 110 | 58 | Trt A/ Time 1 | PPD | 1/1 | -30m | 80 | 90 L | 350 | 800 H | 450 | 520 | 495 |
| , | Male/ | Per 2 | 14:00 | | | | | | | | | |
| /BA | White/ | | | | | | | | | | | |
| | | T | PPD | - / - · | 0.6 | 0.0 | 1 = 0 | 250 | 550 | 4.5.0 | F 0 0 | 405 |
| | | Time 2 | | 7/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 15:00 | | | | | | | | | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_EG6
Protocol: GSK123456
Population: xxxxx


### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./<br>Subj./<br>Seq. | Age (y)/<br>Sex/<br>Race | Treat-<br>ment/<br>Period | Planned<br>Relative<br>Time/ECG<br>Date/Time | Study<br>Day/<br>Period<br>Day | ECG Finding | Clinically<br>Significant<br>Change from<br>Baseline? | Clinically<br>Significant Abnormality |
|---|---|---|---|---|---|---|---|
| PPD<br>A/B | 65/<br>Female/<br>White | Trt A/<br>Per 1 | Visit 1/ PPD /14:00 | 1/1 | Normal | | |
| | | | Visit 2/<br>PPD<br>/12:00 | 4/4 | Abnormal-not clinically significant | No | |
| | | Trt B/<br>Per 2 | Visit 3/PPD/19:00 | 8/1 | Abnormal-<br>clinically<br>significant | | Sinus tachycardia |
| | | | Visit 4/PPD/13:00 | 12/4 | No result (not available) | | |
| PPD<br>B/A | 58<br>Male/<br>White | Trt B/<br>Per 1 | Visit 1/<br>PPD<br>/14:00 | 16/1 | Abnormal-<br>clinically<br>significant | | Ectopic ventricular beats |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_VS5 Protocol: GSK123456


Listing x.x

#### 

| | | | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|---|---|
| Inv./ | Age(y)/ | Treat- | Planned | | | Blood | Blood | Vital Sign |
| Subj./ | / Sex/ | ment/ | Relative | Actual | Study Day/ | Pressure | Pressure | 3 |
| Seq. | Race | Period | Time | Date/Time | Period Day | (mmHg) | (mmHg) | (units) |
| PPD | 23/ | Tmt B/ | Time 1 | PPD | 1/1 | 190 н | 60 | xx H |
| | Male/ | Per 1 | Time 2 | PPD | 5/5 | 95 | 50 L | xx H |
| B/C/A | White | | Time 3 | PPD | 10/10 | 95 | 60 | XX |
| | | Tmt C/ | Time 1 | PPD | 15/1 | 185 Н | 90 н | xx H |
| | | Per 2 | Time 2 | PPD | 20/5 | 95 | 50 | xx H |
| | | | Time 3 | PPD | 25/10 | 95 | 60 | XX |
| | | Tmt A/ | Time 1 | PPD | 30/1 | 200 Н | 45 L | хх Н |
| | | Per 3 | Time 2 | PPD | 35/5 | 95 | 60 | xx H |
| | | | Time 3 | PPD | 40/10 | 95 | 85 Н | xx |

Example: SAFE\_L1
Protocol: GSK123456


Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./ | Age(y)/ | Treat-ment/ | Planned | Actual | Study Day/ | Location/ | Test type | Side | Test |
|---|---|---|---|---|---|---|---|---|---|
| Subj./ | Sex/ | Period | Relative | Date/Time | Period Day | Category | | | Result |
| Seq. | Race | | Time | | | | | | |
| PPD | 23/ | Tmt B/ | Time 1 | PPD | 1/ | Eye/ | Indirect<br>fundoscopic<br>exam | Left | Normal |
| | Male/ | Period x | | | 1 | Ophthalmological examination | | Right | XXXXX |
| B/C/A | White | | | | | | Slit lamp | Left | XXXXXX |
| | | | | | | | | Right | XXXXXX |
| | | | Time 2 | | 5/ | | xxxxxxxxx | xxxxx | XXXXXXX |
| | | | | | 5 | | | XXXXX | XXXXXXX |
| | | | | | | | XXXXXXXXX | XXXXX | XXXXXXX |
| | | | | | | | | XXXXX | XXXXXXX |
| | | Tmt C/ | Time 1 | | 15/ | | xxxxxxxx | xxxxx | XXXXXXX |
| | | Period 2 | | | 1 | | | xxxxx | xxxxxxx |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

## 10.10.3. PK population

Example: PK01


Population: xxxxx

Table x.x

{Add Planned

| Treatmen<br>t | N | time var.} | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | {95% CI (Lower, Upper)} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 50mg | 24 | | Pre-dose | 24 | 20 | xxxx.x | (xxxx.x,xxxx.x) | | xxxx.x | XXXX | xxxx |
| | | | 30 min | 24 | 1 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 1 hr | 23 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 2 hr | 24 | 0 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 100mg | 24 | | Pre-dose | 24 | 3 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | xxxx |
| | | | 30 min | 21 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 1 hr | 21 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 2 hr | 21 | 0 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 200mg | 24 | | Pre-dose | 24 | 0 | xxxx.x | (xxxx.x, xxxx.x) | xx.xx | XXXX.X | xxxx | xxxx |
| _ | | | 30 min | 23 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 1 hr | 24 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 2 hr | 24 | 0 | xxxx.x | (xxxx.x, xxxx.x) | XX.XX | xxxx.x | XXXX | XXXX |

206817

Example: PK03


Population: xxxxx

#### 

| Parameter | Treatment | N | {Additio<br>nal<br>time<br>variable<br>s} | n | Mean | {95% CI<br>(Lower,Upper)<br>} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| AUC(0-t) (units) | 50mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | xx.xx | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 24 | XXXX.XX | (xxxx.xx,xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | xxxx.x |
| | 100mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | xx.xx | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 23 | XXXX.XX | (xxxx.xx,xxxx<br>.xx) | XX.XX<br>X | XXXX.XX | xxxx.x | xxxx.x |
| Cmax (units) | 50mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | xx.xx<br>x | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 23 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | xxxx.x |
| | 100mg | 24 | 1 | 24 | XXXX.XX | (xxxx.xx,xxxx<br>.xx) | xx.xx<br>x | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 21 | XXXX.XX | (xxxx.xx, xxxx<br>.xx) | | XXXX.XX | xxxx.x | xxxx.x |

Example: PK05


Population: xxxxx

## Table x.x Xxxxxxxxxxxxxxxxxxxx

# 

| | | | (IIAAI CIOIIA | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | 1 | | Geom. | 95% CI | | |
| Parameter | Treatment | N | time | n | Mean | (Lower, Upper) | SD | {%CVb} |
| | | | variables} | | | | (logs) | |
| AUC(0-t) (units) | 50mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | xx.xx |
| | | | 14 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.XX |
| | 100mg | 24 | 1 | 24 | XXXX.XX | (xxxx.xx, xxxx.xx) | xx.xxx | XX.XX |
| | | | 14 | 23 | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xxx | xx.xx |
| | 200mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx, xxxx.xx) | xx.xxx | XX.XX |
| | - | | 14 | 21 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.XX |
| Cmax<br>(units) | 50mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.XX |
| | | | 14 | 24 | xxxx.xx | (xxxx.xx, xxxx.xx) | xx.xxx | xx.xx |
| | 100mg | 24 | 1 | 24 | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.XX |
| | | | 14 | 23 | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.XX |
| | 200mg | 24 | 1 | 24 | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.XX |
| | | | 14 | 21 | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.XX |

206817

Example: PK\_T1

Population: xxxxx

Table x.x

| Parameter | Effect | n | Slope Point | SE | 90% CI |
|-------------------|------------------|----|-------------|-----|----------|
| | | | Estimate | | |
| Parameter1 (unit) | Log(dose levels) | XX | XXX | xxx | (xx, xx) |
| Parameter2 (unit) | Log(dose levels) | XX | XXX | XXX | (xx, xx) |
| | • | | • | • | • |
| | • | | | | |

206817

Example: PK\_T2
Protocol: GSK123456


Population: xxxxx

## Table x.x

| Parameter | Treatment | N | n | Geometric LS Mean | Ratio (Fasted/Fed) | 90% CI | CVw(%)[1] |
|---|---|---|---|---|---|---|---|
| Parameter1 (unit) | Trt1 | XX | XX | xxx | Xxx | (xx, xx) | XX |
| | Trt2 | XX | XX | xxx | | | |
| Parameter2 (unit) | Trt1 | XX | XX | xxx | xxx | (xx, xx) | XX |
| • | | | | | • | | • |
| • | • | • | • | • | • | • | • |
| • | • | • | • | • | • | • | • |
| ParameterX (unit) | XX | XX | XX | xxx | xxx | (xx, xx) | XX |

Example: PK16b


Population: xxxxx

#### 



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK24


Population: xxxxx

### 

#### Treatment = tablet original fed



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK18




USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK\_F1

Population: xxxxx

Figure x.x



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK28


Population: xxxxx

#### 



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK08 (pkcl1x) Protocol: GSK123456


Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| _ | {Inv./}<br>Subj. | {Age(y)/<br>Sex/<br>Race} | Period<br>/Tmt. | Date | Study<br>Day /<br>Period<br>Day | Planned<br>Relative<br>Time | Actual<br>time | Time dev. (units) | Actual<br>Relative<br>Time | Concentration (units) |
|---|---|---|---|---|---|---|---|---|---|---|
| | PPD | 36/<br>M/<br>Mixed Race | 1/<br>50mg | PPD | 1/1 | pre-dose | 11:55 | 0 | 0h 0m 0s | 123 |
| | | 1121100 11000 | | | | 5m | 12:05 | 0 | 0h 5m 0s | 1434 |
| | | | | | | 1h | 13:00 | 0 | 1h 0m 0s | NQ (<0.23) |
| | | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |
| | | | 2/<br>100mg | | 17/1 | pre-dose | 11:57 | 0 | 0h 0m 0s | 435 |
| | | | | | | 5m | 12:10 | 0.83 | 0h 10m 0s | 34566 |
| | | | | | | 1h | 12:56 | -0.67 | 0h 56m 0s | 3452 |
| | | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |
| | | 33/<br>M/<br>Mixed Race | 1/<br>50mg | | 1/1 | pre-dose | 11:58 | 0 | 0h 0m 0s | 2345 |
| | | | | | | 5m | 12:04 | -0.17 | 0h 4m 0s | 234 |
| | | | | | | 1h | 12:35 | 0.83 | 1h 0m 0s | NR |
| | | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK\_L1

Population: xxxxx

#### Listing x.x xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| {Inv./}<br>Subj. | {Age(y)/<br>Sex/<br>Race} | Parameter<br>(units) | Period/<br>Tmt. | Value |
|---|---|---|---|---|
| PPD | 36/<br>M/<br>Mixed Race | Parameter1(unit) | 1/<br>50mg<br>2/<br>100mg | xx.xx<br>xx.xx |
| | | Parameter2(unit) | 1/<br>50mg<br>2/<br>100mg | xx |
| | 29/<br>M/<br>Mixed Race | Parameter1(unit) | 1/<br>100mg<br>2/ | xx.xx<br>xx.xx |
| | | Parameter2(unit) | 50mg<br>1/<br>100mg | xx |

USER ID: directory/program.sas DDMMMYYYY hh:mm
# 11. REVISION HISTORIY

| Version | Date | Amendment |
|---------|-------------|-------------------|
| 00 | 11-Jul-2017 | Issued version 00 |

### The GlaxoSmithKline group of companies

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

Title

: Reporting and Analysis Plan for Study 206817: A Single
Centre, Double Blind (Sponsor Open), Placebo Controlled, 3Period Crossover, Ascending Dose Study in Japanese Healthy
Elderly Male Subjects to Evaluate the Safety, Tolerability and
Pharmacokinetics of Danirixin in the Fed State (Part1) and an
open label, 2-way crossover to evaluate food effect on the
pharmacokinetics of Danirixin (Part2).

Compound Number : GSK1325756

Effective Date : 26-JUL-2017

### **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in the clinical pharmacology study report for protocol 206817.
- This RAP is intended to describe the safety, pharmacokinetics analyses required for the study.
- This version includes amendments to the originally approved RAP.
- This document will be provided to the study team members to convey the content of the statistical analysis complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | |
|---|---|
| Biostatistics Group 2 Associate Manager, Biomedical Data Sciences Department, Japan. | 21-Jul-2017 |
| PPD | |
| Clinical Pharmacology & Science Promotion Office, Medicines Development, Japan. | 21-Jul-2017 |

### Approved:

| PPD | |
|----------------------------------------------------------|-------------|
| Department Manager, Biomedical Data Sciences Department, | 26-Jul-2017 |
| Japan. | |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | F | PAGE |
|---|---|---|---|
| 1. | | RTING & ANALYSIS PLAN SYNPOSISRAP Amendments | |
| 2. | 2.1. (2.2. Since 2.3. | ARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s) Study Design Statistical Hypotheses | 6<br>6<br>7 |
| 3. | 3.1. I | IED ANALYSESInterim AnalysesFinal Analyses | 9 |
| 4. | | SIS POPULATIONSProtocol Deviations | |
| 5. | | DERATIONS FOR DATA ANALYSES AND DATA HANDLING ENTIONS | 10 |
| 6. | | POPULATION ANALYSESOverview of Planned Analyses | |
| 7. | 7.1. 0<br>7.2. 0 | Y ANALYSES Overview of Planned Adverse Events Analyses Overview of Planned Clinical Laboratory Analyses Overview of Planned Other Safety Analyses | 12<br>12 |
| 8. | 8.1. 8.2. I<br>8.3. I | MACOKINETIC ANALYSES | 14<br>15<br>15<br>15 |
| 9. | REFER | RENCES | 20 |
| 10. | 10.1. //<br>10.2. //<br>10.3. //<br>10.4. // | Appendix 1: Protocol Deviation Management | 22<br>23<br>26<br>26<br>27<br>27<br>27 |


| | | | 206817 |
|---|---|---|---|
| 10.5. | Appendix | x 5: Derived and Transformed Data | 31 |
| | 10.5.1. | General | |
| | 10.5.2. | Study Population | 31 |
| | 10.5.3. | Safety | 32 |
| | 10.5.4. | Pharmacokinetics | 33 |
| 10.6. | Appendix | x 6: Premature Withdrawals & Handling of Missing Data | 34 |
| | 10.6.1. | Premature Withdrawals | |
| | 10.6.2. | Handling of Missing Data | 34 |
| | 10.6.3. | Handling of Partial Dates | |
| | 10.6.4. | Handling of Missing Data for Statistical Analysis | 34 |
| 10.7. | Appendix | x 7: Values of Potential Clinical Importance | 35 |
| | 10.7.1. | Laboratory Values (Healthy Volunteers) | 35 |
| | 10.7.2. | ECG (Healthy Volunteers) | |
| | 10.7.3. | Vital Signs (Healthy Volunteers) | 36 |
| 10.8. | Appendix | x 8 - Abbreviations & Trade Marks | |
| | 10.8.1. | Abbreviations | 37 |
| | 10.8.2. | Trademarks | 38 |
| 10.9. | Appendix | x 9: List of Data Displays | 39 |
| | 10.9.1. | Data Display Numbering | 39 |
| | 10.9.2. | Mock Example Referencing | 39 |
| | 10.9.3. | Deliverable [Priority] | 39 |
| | 10.9.4. | Study Population Tables | 40 |
| | 10.9.5. | Safety Tables | |
| | 10.9.6. | Pharmacokinetic Tables | |
| | 10.9.7. | Pharmacokinetic Figures | 46 |
| | 10.9.8. | ICH Listings | 48 |
| 10.10. | Appendix | x 10: Example Mock Shells for Data Displays | 54 |
| | 10.10.1. | Study population | 54 |
| | 10.10.2. | Safety population | 79 |
| | 10.10.3. | PK population | 100 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | <ul> <li>The purpose of this RAP is to describe the planned analyses and output to be included<br/>in the Clinical Study Report for Protocol 206817.</li> </ul> |
| Protocol | <ul> <li>Reporting and Analysis Plan is based on original protocol (Dated:11-Apr-2017) for study<br/>GSK1325756 / 206817 [GlaxoSmithKline Document Number:2016N309585_01]</li> </ul> |
| Objectives | Part 1 |
| | <ul> <li>To assess the safety, tolerability and PK following single doses of GSK1325756H 10,<br/>50 and 100 mg in the fed state in healthy Japanese subjects of over 65 years of age<br/>inclusive.</li> </ul> |
| | Part 2 |
| | <ul> <li>To investigate the safety, tolerability and food effect on PK of GSK1325756 following a<br/>single dose of 50 mg in the fed and fasted state, in healthy Japanese subjects of over<br/>65 years of age inclusive.</li> </ul> |
| Endpoints | Part 1 and 2. |
| | Adverse events (AEs) |
| | <ul> <li>Change from baseline of clinical laboratory values, vital signs, and electrocardiogram<br/>(ECG) parameters</li> </ul> |
| | Blood concentration of GSK1325756 |
| | <ul> <li>Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, tlag, tlast of the blood<br/>concentration of GSK1325756, as data permit</li> </ul> |
| Study | This study consists of two parts. |
| Design | <ul> <li>Part 1 is a double blind, placebo-controlled, 3-period crossover, ascending dose, single<br/>oral administration in the fed condition</li> </ul> |
| | Part 2 is an open label, 2-way crossover, single oral dose in the fed and fasted state. |
| Analysis | Screened: Consisting of all subjects screened in the study |
| Population | <ul> <li>Screening Failure: Subjects who screened in the study but are never subsequently<br/>randomized.</li> </ul> |
| | Safety: All randomized subjects who take at least one dose of study treatment. |
| | <ul> <li>Pharmacokinetic: This population is defined as all subjects administered at least one<br/>dose of study treatment and who have PK sample taken and analysed.</li> </ul> |
| Hypothesis | The objectives of this study are to evaluate safety and tolerability of GSK1325756 and to estimate GSK1325756 Pharmacokinetic parameters. No formal statistical hypotheses will be tested in Part 1 and Part 2. Descriptive statistics will be used to assess safety and tolerability objectives. An estimation approach will be used to address the pharmacokinetic study objectives, where point estimates and corresponding 90% confidence intervals will be constructed. |
| Safety<br>Analyses | <ul> <li>Safety data will be presented in tabular and/or graphical format and summarized<br/>descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.</li> </ul> |
| Pharmacoki<br>netic<br>Analyses | Individual GSK1325756 blood concentration-time profiles (by part, treatment and subject) and median/mean (±SD) profiles by part and treatment will be plotted and listed. Treatment indicates dose group in Part 1 and the fed and fasted condition in Part 2. |
| | Blood concentration time data for GSK1325756 will be analyzed by non-compartmental methods using WinNonlin and derived PK parameters graphically present, summarised |

- and listed. No formal statistical analyses will be conducted.
- Statistical analyses will be carried out to explore the dose proportionality of GSK1325756 as assessed by AUC(0-t) and Cmax using the Power Model (Part 1).
- Statistical analyses will be carried out to explore the food effect of GSK1325756 as assessed by AUC(0-t) and Cmax using a mixed effects mode (Part 2).

### 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_206817_Final [11-Jul-2017 | |
| Reporting and Analysis Plan_206817_Final_Amend 1 [DD-Jul-2017] | |
| 1.1 RAP Amendments • added the section | |
| 10.9.1. Data Display<br>Numbering | corrected number of ICH Listings |
| 10.9.3. Deliverable [Priority] | deleted "(Part 2 only)" for SAC [2] |
| 10.9.4. Study Population Tables | <ul> <li>deleted "(Yes or No)" in the Programing Notes for No. 1.7 and No. 1.8</li> </ul> |
| 10.9.6. Pharmacokinetic Tables | added unit in the title for No. 3.1 and No. 3.5 |
| 10.9.8. ICH Listings | <ul> <li>corrected "Deliverable [Priority]" column for No. 1, No. 18, and No. 26</li> </ul> |
| | <ul> <li>added "Listing of Relationship between ATC Level 1, Ingredient and<br/>Verbatim Text" as No. 21</li> </ul> |
| | <ul> <li>corrected the title for No. 44 and No. 46</li> </ul> |
| | corrected "IDSL / TST ID / Example Shell" column for No. 70 and No. 71 |
| 10.10.1. Study population | added CM6 |
| 10.10.3. PK population • deleted "(unit)" in "Parameter" column for PK_T1 | |
| | deleted PK_L1 |
| | added PK14 |
| 11. Revision History | deleted the section |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [Dated: 11/APR/2017].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Part 1 | Part 1 and Part 2 |
| <ul> <li>To assess the safety, tolerability and PK<br/>following single doses of GSK1325756H 10,<br/>50 and 100 mg in the fed state in healthy<br/>Japanese subjects of over 65 years of age<br/>inclusive.</li> </ul> | <ul> <li>Adverse events (AEs)</li> <li>Change from baseline of clinical laboratory values, vital signs, and electrocardiogram (ECG) parameters</li> <li>Blood concentration of GSK1325756</li> </ul> |
| <ul> <li>Part 2</li> <li>To investigate the safety, tolerability and food effect on PK of GSK1325756 following a single dose of 50 mg in the fed and fasted state, in healthy Japanese subjects of over 65 years of age inclusive.</li> </ul> | <ul> <li>Cmax, AUC(0-t), AUC(0-inf), AUC(0-24), tmax, t1/2, tlag, tlast of the blood concentration of GSK1325756, as data permit</li> </ul> |

# 2.3. Study Design

# **Overview of Study Design and Key Features**

Subjects will be divided into Part 1 and 2, and receive the following study treatment doses shown in Table below.

### Part 1:

| Group | n | Period 1 | Washout | Period 2 | Washout | Period 3 |
|---|---|---|---|---|---|---|
| Α | 6 | 10 mg | | 50 mg | | Placebo |
| В | 6 | 10 mg | at least 7<br>days | Placebo | at least 7<br>days | 100 mg |
| С | 6 | Placebo | | 50 mg | | 100 mg |

### Part 2:

| Group | n | Period 1 | Washout | Period 2 |
|-------|---|---------------|------------|---------------|
| D | 8 | 50 mg, fed | at least 7 | 50 mg, fasted |
| Е | 8 | 50 mg, fasted | days | 50 mg, fed |

| Design<br>Features | Part 1: This is a double blind, placebo-controlled, 3-period crossover, ascending dose, single oral administration in the fed condition. |
|---|---|
| | Part 2: This is an open label, 2-way crossover, single oral dose in the fed and fasted state study. |
| Dosing | Part 1: Subjects will have a screening visit within 30 days prior to the first dose of study. A minimum washout period of 7 days will be required between each treatment period. Subjects will receive three treatment periods in the study. Subjects will be housed in the Clinical Research Unit from Day -1 (the day before dosing) through Day 3 for Period 1 and 2, and from Day -1 (the day before dosing) through Day 4 for Period 3. Subjects will return to the clinic 7 days (at least) after the previous administration day for Period 1 and 2, and subjects will visit the unit on Day 8 (+/- 1 day) of the last dosing for Period 3 for follow-up. |
| | Part 2:<br>Subjects will have a screening visit within 30 days prior to the first dose of study treatment, two treatment periods separated by at least 7 days, and follow-up. Subjects will be housed in the Clinical Research Unit from Day -1 (the day before dosing) through Day 3 (for Period 1 and 2), and re-visit 7 (±1) days after the last dose of Period 2 for follow-up. |

## Overview of Study Design and Key Features Sufficient participants will be randomised such that approximately 18 Treatment in Part 1 and 16 in Part 2 evaluable participants complete the study of Assignment each part. If participants prematurely discontinue the study, additional participants may be enrolled as replacement participants and assigned to the same treatment sequence, if applicable, at the discretion of the sponsor in consultation with the investigator. On Day 1 of each Part, participants will be assigned a unique number (randomization number) in ascending numerical order. The randomization number encodes the participant's assignment to one of the 3 sequences in Part 1 and one of the 2 sequences in Part 2, according to the randomization schedule generated prior to the study by the Biomedical Data Sciences Department at GSK. Participants will be randomized in a 1:1:1 ratio to receive sequence (A:B:C) for Part 1, or will be randomized in a 1:1 ratio to receive sequence (D:E) for Part 2. Each participant will be dispensed blinded study treatment, labeled with his unique randomization number, throughout the study. Investigators, participants and sponsor will remain blinded to each participant's assigned study treatment throughout the course of the study. For the concentration evaluation after Period 2 of Part 1, the pre-specified sponsor's person who is responsible for the confirmation of the concentration will review blood drug concentration data under unblended. No formal statistical analysis is planned. Interim Analysis A blind review of preliminary safety data (AE, clinical laboratory values, vital signs, ECG) and blood concentration will be conducted between Period 2 and Period 3 in Part 1 and prior to Part 2. After completion of Part 1, formal analysis for Part 1 is to be conducted.

# 2.4. Statistical Hypotheses

The objectives of this study are to evaluate safety, tolerability and PK profile of single dose of GSK1325756H and to investigate food effect of PK profile of single dose of GSK1325756H in healthy Japanese elderly subjects. No formal statistical hypotheses will be tested in Part 1 and Part 2. Descriptive statistics will be used to assess safety and tolerability objectives. An estimation approach will be used to address the PK study objectives, where point estimates and corresponding 95% confidence intervals will be constructed, unless otherwise stated.

### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

No formal statistical analysis is planned. However, following Period 1 and Period 2 of Part 1, a blind review of preliminary safety data (AE, clinical laboratory values, vital signs, ECGs) will be conducted between Period 2 and Period 3 in Part 1 and prior to Part 2. Furthermore, the sponsor's person who is responsible for the confirmation of the concentration will review blood drug concentration data under unblended.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects in each part have completed the study as defined in the protocol.
- 2. All required database cleaning activities in each part have been completed and final database release and database freeze has been declared by Data Management for each part.
- 3. All criteria for unblinding the randomisation codes have been met for Part 1.
- 4. Randomisation codes have been distributed according to RandAll NG procedures. After completion of Part 1, formal analysis for Part 1 is to be conducted.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Screened | Consisting of all subjects screened in the study. | Study Population |
| | Note: This definition indicates the same meaning as 'All subjects who have subject number' in a programming point of view. | |
| Screening Failure | Subjects who screened in the study but are never subsequently randomized. All participants who sign the ICF have the screening test in the study. | Study Population |
| | Note: This definition indicates the same meaning as 'Subjects who have subject number but are never subsequently randomized' in a programming point of view. | |
| Safety | All randomized subjects who take at least<br>one dose of study treatment. Participants will | Study Population |
| | be analyzed according to the treatment they actually received. | Safety |

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Pharmacokinetic | This population is defined as all subjects administered at least one dose of study treatment and who have PK sample taken and analysed. Participants will be analyzed according to the treatment they actually received. | • PK |

### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - o This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided. This will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---------|--------------------------------------------------------------|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Treatment States and Phases |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Safety Population, unless otherwise specified. These analyses will be performed in each part.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition and Reason for Study Withdrawal | Y | | Υ |
| Screening Status and Reasons for Screen Failure | Y | | Υ |
| Subjects for Whom the Treatment Blind was Broken | | | Υ |
| Planned and Actual Treatments | | | Y |
| Protocol Deviations | | | |
| Important Protocol Deviations | Y | | Υ |
| Inclusion/Exclusion Criteria Deviations | | | Υ |
| Populations Analysed | · | | |
| Study Populations | Υ | | |
| Subjects Excluded from Any Population | | | Y |
| Demographic and Baseline Characteristics | · | | |
| Demographic Characteristics | Y | | Υ |
| Demographic Characteristics for Screening Failure | | | Y |
| Age Ranges | Y | | |
| Race and Racial Combinations | Y | | Υ |
| Race and Racial Combinations for Screening Failure | | | Y |
| Medical Conditions and Concomitant Medications | · | | |
| Medical Conditions | | | Υ |
| Concomitant Medications | | | Y |
| Exposure and Treatment Compliance | | • | |
| Exposure to Study Treatment | | | Υ |
| Meal | | • | |
| Meal start and end days/times on fed treatment | | | Υ |

### NOTES:

• Y = Yes display generated.

### 7. SAFETY ANALYSES

The safety analyses will be based on the Safety Population, unless otherwise specified. These analyses will be performed in each part.

Adverse events occurred in washout period will be included in adverse events analyses for previous period. Also adverse events occurred in follow up period will be included in safety analyses for the last period.

### 7.1. Overview of Planned Adverse Events Analyses

Table 3 provides an overview of the planned adverse events analyses with full details of data displays being presented in Appendix 9: List of Data Displays.

Table 3 Overview of Planned Adverse Event Analyses

| Display Type | | Absolute | |
|---|---|---|---|
| | Sumi | Summary | |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Υ | | Υ |
| All AEs by Maximum Intensity | Υ | | |
| Drug-Related AEs by SOC and PT | Υ | | |
| Drug-Related AEs by Maximum Intensity | Υ | | |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Serious AEs | | | Υ |
| AEs Leading to Withdrawal from Study | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.2. Overview of Planned Clinical Laboratory Analyses

Table 4 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

Table 4 Overview of Planned Clinical Laboratory Analyses

| Display Type | | Abs | olute | Ch | Change from BL | |
|---|---|---|---|---|---|---|
| | <del>- </del> | | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Chemistry Data | Υ | | Υ | Υ | | Υ |
| Chemistry Results Relative to Normal Range | | | | Υ | | |
| All Chemistry Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | Y |
| Hematology | | • | | | • | |
| Hematology Data | Υ | | Υ | Υ | | Υ |
| Hematology Results Relative to Normal Range | | | | Υ | | |
| All Hematology Data for Subjects with any Value of Potential Clinical Concern/PCI | | | Y | | | Y |
| Urinalysis | | • | | | • | |
| Dipstick Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) | Υ | | Y* | | | |
| Gravity and pH | Υ | | Υ | | | |
| Hepatobiliary (Liver) | | | | | | |
| Liver Monitoring/Stopping Event Reporting | | | Υ | | | |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y | | | |
| Substance Use for Subjects with Liver Stopping Events | | | Y | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.3. Overview of Planned Other Safety Analyses

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 9: List of Data Displays.

<sup>\*:</sup> If blood or protein is abnormal, microscopic examination will be included.

Table 5 Overview of Planned Other Safety Analyses

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Summary | | Individual | Sumn | nary | Individual |
| | Т | F | L | Τ | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Y | | | |
| ECG Values | Υ | | Y | Υ | | Υ |
| All ECG Values for Subjects with any Value of PCI | | | Y | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Y | Υ | | Υ |
| All Vital Signs for Subjects with any Value of PCI | | | Y | | | |
| Ophthalmic examinations | | | | | | |
| Ophthalmic examinations | | | Υ | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8. PHARMACOKINETIC ANALYSES

# 8.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic population, unless otherwise specified. These analyses will be performed in each part.

Table 6 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 6 Overview of Planned Pharmacokinetic Analyses

| Display Type | l | Intrans | sformed | | Log-Transformed | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Stats<br>analysis | Summary | | Indiv | ridual |
| | F | T | F | L | | F | T | F | L |
| Descriptive statistics | | | | | | | | | |
| Blood Drug Concentrations | Y [1] [2] | Υ | Υ [1] | Υ | | | | | |
| Derived PK Parameters | Υ | Υ | | Υ | | | Υ | | |
| Statistical Analysis of PK Para | Statistical Analysis of PK Parameters | | | | | | | | |
| Power model (Part 1) | | | | | Υ | | | | |
| Food effect (Part 2) | | | | | Υ | | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (+ SD) and Median plots will be generated.

### 8.2. Drug Concentration Measures

Blood concentrations of GSK1325756 will be listed and summarised by part, treatment and nominal time. Standard summary statistics will be calculated (i.e. mean, standard deviation, median, minimum and maximum).

Individual blood concentration-time profiles and median/mean profiles by treatment will be plotted. Each of the figures will contain one plot on the untransformed scale (i.e. a linear plot) and one plot on the log transformed scale (i.e. log-linear plot).

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.4 Reporting Process & Standards).

### 8.3. Pharmacokinetic Parameters

### 8.3.1. Deriving Pharmacokinetic Parameters

- Derivation of pharmacokinetic parameters will be performed by, or under the direct auspices of, Clinical Pharmacology & Science Promotion Office, GlaxoSmithKline K.K.
- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.4 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis using WinNonlin (version 6.3 or higher)
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.
- Pharmacokinetic parameters described in Table 7 will be determined from blood GSK1325756 concentration-time data, as data permits.

 Table 7
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-24)<br>(h*ng/mL) | Area under the concentration-time curve will be calculated to fixed nominal time 24 hours after administration (AUC(0-24)),using the combination of linear and logarithmic trapezoidal methods (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| | If a sampling time deviation occurred at nominal time 24 hours after administration (and 24 < t), AUC(0-24) will be calculated using the concentration at time 24 hours after administration post-dose estimated by the method of interpolation. |
| | If nominal time 24 hours after administration > t (or if the concentration at time 24 hours after administration was below then limit of quantification), then the concentration (y) at time 24 hours after administration is estimated using lambda_z and last observed Ct according to the formula: |
| | y=Ct(obser) x e-lambda_z(24-t) |
| | Then the following equation will be used to calculate (AUC(0-24)) where t is the time of last quantifiable blood concentration. |
| | AUC(0-24) = AUC(0-t) + AUC(t-24) |
| | If lambda_z is not estimable, a partial AUC is not calculated (when 24 > t). |
| AUC(0-t)<br>(h*ng/mL) | Area under the concentration-time curve from zero time (pre-dose) to the time of the last quantifiable concentration (AUC(0-t)) will be calculated by a combination of linear and logarithmic trapezoidal methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). |
| AUC(0-inf)<br>(h*ng/mL) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite time (AUC(0-inf)) will be calculated as follows: |
| | $AUC(0-inf) = AUC(0-t) + Ct / lambda_z$ |
| Cmax (ng/mL) | Maximum observed concentration will be obtained directly from the concentration-time data. |
| Tmax (h) | Time to first occurrence of Cmax will be obtained directly from the concentration-time data. |
| t1/2 (h) | Terminal phase half-life will be calculated as follows: |
| | t1/2 = ln2 / lambda_z |
| tlag (h) | Lag time before observation of drug concentrations in sampled matrix. |

| Parameter | Parameter Description |
|---|---|
| tlast (h) | The time of the last measurable (positive) concentration. |
| %AUCex (%) | The area under the curve (AUC) from the last predicted non-zero concentration value to infinity as a percentage of the area under the curve extrapolated to infinity. |
| lambda_z (/h) | The first order rate constant associated with the terminal (log-linear) portion of the curve. |
| lambda_z_lower (h) | The lower limit on time for values to be included in the calculation of Lambda z. |
| lambda_z_upper (h) | The upper limit on time for values to be included in the calculation of Lambda z. |
| #pts | The number of time points used in computing Lambda z. |
| R2 | The goodness of fit statistic for the terminal elimination phase. |

- Additional parameters may be included as required.
- Lambda z is the terminal phase rate constant.
- Ct is the last observed quantifiable concentration.

### 8.3.2. Summary of Pharmacokinetic Parameters

- For each of these parameters, except for tmax, tlag and tlast, the following summary statistics will be calculated for each treatment:
  - o Non-transformed: arithmetic mean, median, maximum, minimum, 95% confidence interval for the arithmetic mean and standard deviation
  - Loge-transformed: geometric mean, 95% confidence interval for the geometric mean, standard deviation of logarithmically transformed data and between geometric coefficient of variation (CVb (%))
- Median, maximum, minimum, arithmetic mean, 95% confidence interval and standard deviation will be calculated for tmax, tlag and tlast.

### 8.3.3. Statistical Analysis of Pharmacokinetic Parameters

### 8.3.3.1. Dose proportionality

For Part 1, the PK-dose relationship will be investigated graphically in order to assess dose proportionality of GSK1325756. Plots of AUC (0-t) and Cmax versus dose will be plotted.

Also statistical analyses will be carried out to explore the dose proportionality of GSK1325756 as assessed by AUC(0-t) and Cmax, using the Power Model:

$$\log_{e}(Y_{ij}) = \mu + S_{i} + \beta * \log_{e}(D_{j}) + \varepsilon_{ij}$$

 $Y_{ij}$ : PK parameter (AUC(0-t), Cmax) on the *j*th dose for *i*th subject

μ: Overall mean (Intercept)

S<sub>i</sub>: Random effect for subject i following normal distribution  $N(0, \sigma_b^2)$ 

β: Slope for loge transformed dose

D<sub>j</sub>: Dose (j=1:10mg, 2:50mg, 3:100mg)

 $\epsilon_{ij}$ : Random error following normal distribution N(0,  $\sigma_w^2$ )

Following loge-transformation, AUC (0-t) and Cmax will be separately analyzed, if data permitted. A mixed effect model will be fitted with the loge transformed dose and period as fixed effects. Subject will be fitted as a random effect. The Kenward & Roger (KR) degrees of freedom approach will be used. Point estimates and their associated 90% confidence intervals will be constructed.

#### 8.3.3.2. Food effect

For Part 2, statistical analyses will be carried out to assess treatment (food effect) of GSK1325756 for AUC(0-t) and Cmax using Mixed effect model:

$$\log_e(Y_{ij}) = \mu + S_i + t_j + p_k + \varepsilon_{ij}$$

 $Y_{ij}$ : PK parameter (AUC(0-t), Cmax) on the *j*th treatment for *i*th subject

μ: Overall mean (Intercept)

S<sub>i</sub>: Random effect for subject i following normal distribution  $N(0, \sigma_b^2)$ 

t<sub>i</sub>: Treatment effect (j=fasted, fed)

pk: Period effect (k=period 1, period 2)

 $\epsilon_{ij}$ : Random error following normal distribution N(0,  $\sigma_w^2$ )

Following loge-transformation, AUC (0-t) and Cmax will be separately analysed using a mixed effects model fitting terms for treatment and period as fixed effects, and subject as a random effect in order to assess food effect of GSK1325756 (Fed vs. Fasted). The Kenward & Roger (KR) degrees of freedom approach will be used.

Point estimates for the adjusted means on the loge scale, the mean difference between treatments and associated 90% confidence interval will be constructed using the residual variance. The point estimate and confidence interval will then be exponentially backtransformed to obtain adjusted (least square) geometric means for each treatment, and point estimates and associated 90% confidence interval for the ratio of fasted/fed.


206817

Estimates of within-subject variability (CVw (%)) for AUC (0-t) and Cmax will also be provided. CVw (%) will be calculated based on the loge-normal distribution where:

CVw (%)= SQRT(exp(MSE)-1) \* 100. (MSE is the residual mean squared error from the model)

# 9. REFERENCES

GlaxoSmithKline Document Numbers 2016N309585\_01: Study Protocol of 206817. A Single Centre, Double Blind (Sponsor Open), Placebo Controlled, 3-Period Crossover, Ascending Dose Study in Japanese Healthy Elderly Male Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of Danirixin in the Fed State (Part1) and an open label, 2-way crossover to evaluate food effect on the pharmacokinetics of Danirixin (Part2).

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5 | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General |
| | Study Population |
| | Safety |
| | Pharmacokinetics |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | General |
| | Study Population & Safety |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Other RAP App | endices |
| Section 10.8 | Appendix 8: Abbreviations & Trade Marks |
| Section 10.9 | Appendix 9: List of Data Displays |
| Section 10.10 | Appendix 10: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management

Details will be referred latest Protocol Deviation Management Plan and data handling will be decided prior to final data base release.

# 10.2. Appendix 2: Time & Events

# Part 1, Period 1-2

| Day | | | | | | | Day 1 | | | | | | | | Day 2 | Day 3 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose | Screening | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5 h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Subject demography<br>/Medical history | X | | | | | | | | | | | | | | | | |
| Height, Weight, BMI | X | | | | | | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | | | | | | | |
| Serological test | X | | | | | | | | | | | | | | | | |
| Physical examination | X | Х | Х | | | | | | | | Х | | | | | Х | Х |
| Vital signs (PR, BP, temp) | X | Х | Х | | | | | | | | Х | | | | | Х | X |
| 12-lead ECG | X | Х | Х | | | | | | | | Х | | | | | Х | Х |
| Ophthalmic examination | X3 | | | | | | | | | | | | | | | | |
| SAEs <sup>2</sup> | <====== | | | | | | | | | | | | | | | | ====> |
| AEs <sup>2</sup> | | | | <==: | | | | | | | | | | | | | ====> |
| Con Med review | <====== | | | | | | | | | | | | | | | | ====> |
| Hematology, clinical<br>chemistry and urinalysis | X | Х | | | | | | | | | | | | | | | X |
| Administration | | | | Χ | | | | | | | | | | | | | |
| PK sampling | | | X | | X | X | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | Χ | Χ | X |
| Admission | | Χ | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | X |

Screening visit will occur only prior to the first dosing. Treatment Period 2 will occur after at least 7-days wash-out period. High fat meal will be started and completed before within 30 minutes of GSK1325756H/Placebo dosing.

<sup>2.</sup> All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified (see Section 9.1 Adverse Events).

<sup>3.</sup> Ophthalmic examinations are conducted on the day between Screening and Day-1. However, it is not carried out for those who are ineligible due to other screening criteria.

# Part 1, Period 3

| Day | | | | | | | | Day 1 | | | | | | | Day 2 | Da | y 3 | Day 4 | Falleni |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5<br>h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h | 60 h | 72 h | Follow<br>up <sup>2,3</sup> |
| Physical examination | Х | Х | | | | | | | | Х | | | | | X | Х | | Х | Х |
| Vital signs (PR,<br>BP, temp) | Х | Х | | | | | | | | Х | | | | | Х | Х | | Х | Х |
| 12-lead ECG | X | Х | | | | | | | | Х | | | | | Х | Х | | Х | X |
| Ophthaimic<br>examination | | | | | | | | | | | | | | | | | | | X |
| SAEs | <=== | | | | | | | | | | | | | | | | | | ====> |
| AEs | <=== | | | | | | | | | | | | | | | | | | ====> |
| Con Med review | <=== | ====== | ===== | ===== | ===== | | ===== | | ===== | ===== | ===== | | | | | | | .===== | ===> |
| Hematology,<br>clinical chemistry<br>and urinalysis | x | | | | | | | | | | | | | | | | | х | X |
| Administration | | | Х | | | | | | | | | | | | | | | | |
| PK sampling | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X | X | X | Χ | Χ | |
| Admission | X | | | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | | X | |

- Treatment Period 3 will occur after at least 7-days wash-out period. High fat meal will be started and completed before within 30 minutes of GSK1325756/Placebo dosing.
   Follow up visit will occur after 7 days (+/- 1day) of the last dosing.
   In the case where the subject has discontinued the study prematurely, the assessments for follow up will be carried out.

## Part 2, Period 1-2

| Day | | | | | | | | | Day 1 | | | | | | | Day 2 | Day 3 | Follow |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time post-dose | Screening | Day-1 | Pre-<br>dose | 0 h | 0.25<br>h | 0.5<br>h | 0.75<br>h | 1 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 48 h | up <sup>3,5</sup> |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Subject demography<br>/Medical history | Х | | | | | | | | | | | | | | | | | |
| Height, Weight, BMI | X | | | | | | | | | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | | | | | | | | | |
| Serological test | X | | | | | | | | | | | | | | | | | |
| Physical examination | х | Х | Х | | | | | | | | Х | | | | | Х | X | Х |
| Vital signs (PR, BP, temp) | Х | х | Х | | | | | | | | Х | | | | | Х | X | Х |
| 12-lead ECG | X | Х | Х | | | | | | | | Х | | | | | Х | Х | Х |
| Ophthalmic examination | Хе | • | | | | | | | | | | | | | | | | Х |
| SAEs4 | <====== | | | | | | | | ===== | ===== | | | | | | | | ====> |
| AEs4 | | | | <== | | | | | | | | | | | | | | ====> |
| Con Med review | <====== | | | | | | | | | | | | | | | | | ====> |
| Hematology, clinical<br>chemistry and<br>urinalysis | х | х | | | | | | | | | | | | | | | х | х |
| Administration | | | | Χ | | | | | | | | | | | | | | |
| PK sampling | | | Х | | X | Χ | Х | Χ | Х | Χ | Χ | Х | Χ | Х | Х | Х | Х | |
| Admission | | X | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | Х | |

- 1. Screening visit will occur only prior to the first dosing. Treatment Period 2 will occur after at least 7-days wash-out period.
- 2. For the fed condition, meal will be started and completed before within 30 minutes of GSK1325756H dosing.
- 3. Follow up visit will occur after 7-days (+/- 1day) of the last dosing.
- 4. All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified (see Section 9.1.Adverse Events).
- 5. In the case where the subject has discontinued the study prematurely, the assessments for follow up will be carried out.
- 6. Ophthalmic examinations are conducted on the day between Screening and Day-1. However, it is not carried out for those who are ineligible due to other screening criteria.

# 10.3. Appendix 3: Treatment States and Phases

### 10.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the assessment date.

| Treatment Phase | Definition |
|---|---|
| Part 1: Period 1 | Assessment Date < Previous Day of Dosing Start Date in Period 2 (Part 1) |
| Part 1: Period 2 | Previous Day of Dosing Start Date in Period 2 ≤ Assessment Date < Previous Day |
| | of Dosing Start Date in Period 3 (Part 1) |
| Part 1: Period 3 | Previous Day of Dosing Start Date in Period 3 ≤ Assessment Date (Part 1) |
| Part 2: Period 1 | Assessment Date < Previous Day of Dosing Start Date in Period 2 (Part 2) |
| Part 2: Period 2 | Previous Day of Dosing Start Date in Period 2 ≤ Assessment Date (Part 2) |

### 10.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

### 10.3.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date and Time < Dosing Start Date and Time |
| Part 1: Period 1 | Dosing Start Date and Time in Period 1 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 2 (Part 1) |
| Part 1: Period 2 | Dosing Start Date and Time in Period 2 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 3 (Part 1) |
| Part 1: Period 3 | Dosing Start Date and Time in Period 3 ≤ AE Start Date and Time (Part 1) |
| Part 2: Period 1 | Dosing Start Date and Time in Period 1 ≤ AE Start Date and Time < Dosing Start Date and Time in Period 2 (Part 2) |
| Part 2: Period 2 | Dosing Start Date and Time in Period 2 ≤ AE Start Date and Time (Part 2) |
| 0 17 0 | If Dosing Start Date and Time > AE Onset Date and Time = AE Onset Date and Time – Dosing Start Date and Time |
| Onset Time Since<br>First Dose (Minute) | If dosing Start Date and Time ≤ AE Onset Date and Time = AE Onset Date and Time - Dosing Start Date and Time +1 |
| | Missing otherwise |
| Onset Time Since<br>Last Dose (Minute) | AE Start Date and Time – Most Recent Treatment Start Date and Time + 1 |
| Duration (Minute) | AE Resolution Date and Time – AE Onset Date and Time + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF |

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

### 10.4.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | Part1 (So | cedule1) | |
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description | Order [1] |
| Р | Placebo, Fed | Placebo, Fed | 1 |
| X1 | GSK1325756H 10 mg, Fed | GSK1325756H 10 mg, Fed | 2 |
| X2 | GSK1325756H 50 mg, Fed | GSK1325756H 50 mg, Fed | 3 |
| Х3 | GSK1325756H 100 mg, Fed | GSK1325756H 100 mg, Fed | 4 |
| | Part2 (Scedule2) | | |
| X2 | GSK1325756H 50 mg, Fed | GSK1325756H 50 mg, Fed | 1 |
| X4 | GSK1325756H 50 mg, Fasted | GSK1325756H 50 mg, Fasted | 2 |

#### NOTES:

# 10.4.2. Sequence group Display Descriptors

| | Sequence Group Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Description [1] | Order |
| Α | X1/X2/P | A | 1 |
| В | X1/P/X3 | В | 2 |
| С | P/X2/X3 | С | 3 |
| D | X2/X4 | D | 4 |
| E | X4/X2 | Е | 5 |

### NOTES:

Footnote will be added in displays as follows.
 A: 10mg (Fed) / 50mg (Fed) / Placebo (Fed), B: 10mg (Fed) / Placebo (Fed) / 100mg (Fed), C: Placebo (Fed) / 50mg (Fed) / 100mg (Fed), D: 50mg (Fed) / 50mg (Fasted) , E: 50mg (Fasted) / 50mg (Fed)

<sup>1.</sup> Order in which treatments are to be presented in Listings. Note that the order in which treatments are to be presented in Tables, active treatment (X1, X2, X3 in Part 1, X2, X4 in Part 2) is shown in the first and placebo (P in Part 1) in the second.

### 10.4.3. Baseline Definition & Derivations

#### 10.4.3.1. Baseline Definitions

| Parameter | Study Asse | essments<br>as Baselin | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| Parameter | Screening | Screening Day -1 | | |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | Х | Х | Day 1<br>(Pre Dose) |
| Haematology | Х | Х | | Day -1 |
| Clinical Chemistry | X | Χ | | Day -1 |

#### NOTES:

• The baseline will be defined for each period in Part 1 and Part 2.

### 10.4.3.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.3.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.4.4. Reporting Process & Standards

| Reporting Pr | ocess |
|---|---|
| Software | |
| The curre | ntly supported versions of SAS software will be used. |
| Reporting Ar | ea |
| HARP<br>Server | : uk1salx00175 |
| HARP Area | Part1:/arenv/arprod/gsk1325756/mid206817/primary_01 |
| | Part2:/arenv/arprod/gsk1325756/mid206817/final_01 |
| QC | Part1:/arenv/arprod/gsk1325756/mid206817/primary_01/qc |
| Spreadsheet | Part2:/arenv/arprod/gsk1325756/mid206817/final_01/qc |
| Analysis Data | Analysis Datasets |
| Analysis of | Analysis datasets will be created according to GSK IDSL A&R dataset standards |
| Generation of RTF Files | |
| • N/A | • N/A |

### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (4.24) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | gorical Data N, n, frequency, % |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive Summary | Refer to IDSL Statistical Principle 6.06.1 |
| Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |


| Reporting Standards | |
|---|---|
| Reporting of Pharmac | okinetic Parameters |
| Descriptive Summary<br>Statistics.<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb/w (%)) will be reported. |
| | CVb (%) = SQRT (exp(SD <sup>2</sup> ) - 1) * 100 |
| | (SD = SD of loge-transformed data) |
| | CVw (%) =SQRT (exp(MSE) - 1) * 100 |
| | (MSE = mean square error from mixed effect model of loge-transformed data). |
| Parameters Not Being Log Transformed | tmax, tlag, tlast |
| Parameters Not Being<br>Summarised | The following PK parameters will not be summarised but listed: %AUCex, lambda_z, lambda_z_lower, lambda_z_upper, #pts, R2. |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

### **Reporting Standards**

### 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from start of dosing date:
  - Ref Date = Missing
- → Study Day = Missing
- o Ref Date < of start of dosing Date → Study Day = Ref Date of start of dosing Date
- Ref Data ≥ of start of dosing Date → Study Day = Ref Date (of start of dosing Date) + 1

### 10.5.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Reference will be Randomization date for Part 1 and Part 2
- Reference date for calculation of age at screening will be from visit 1 (Screening visit) date, however this will be from screen failure date for a screen failure subject.
- Analysis age group will be categorized (Years):
  - <=18, 19-64, 65-74, >=75
- Age will be categorized for EudraCT:
  - <=17 years, 18-64 years, 65-84 years, >=85 years

### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

### 10.5.3. Safety

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

| Laboratory Assess | Laboratory Assessments |
|---|---|
| Haematology | Platelet Count, RBC Count, Haemoglobin, Hematocrit, RBC Indices (MCV, MCH, %Reticulocytes), WBC count with Differential (Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils) |
| Clinical Chemistry | BUN, Creatinine, Glucose (fasting), Uric acid, HDL-cholesterol, Amylase, Potassium, Sodium, Calcium, TG, LDH, Chloride, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatise, Total Cholesterol, GGT, Phosphorus, Total and direct bilirubin, Total Protein, Albumin, LDL-cholesterol, CK (CPK) |
| Routine Urinalysis | <ul> <li>Specific gravity, pH (assessed by dipstick)</li> <li>glucose, protein, blood, ketones, bilirubin, urobilinogen by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> |

### ECG (12-lead ECG)

ECG findings, ECG values (Heart rate, PR interval, QRS duration, QT interval and QTcF intervals)

### **Vital Signs**

Pulse rate, Blood pressure (Systolic, Diastolic), Temperature

### **Ophthalmic examinations**

Ophthalmic examinations

#### 10.5.4. Pharmacokinetics

#### **PK Parameters**

- If one or more non-quantifiable (NQ) values occur in a profile before the first measurable
  concentration, they will be assigned a value of zero concentration. For linear plots, zero
  concentration value(s) before the first measurable concentration will be included in the plot. For
  log-linear plots, zero concentration value(s) before the first measurable concentration will be
  assigned a missing value.
- If a single NQ value occurs between measurable concentrations in a profile, the NQ should generally be set to missing in the derivation of pharmacokinetic parameters, statistical analysis, and the individual subject plots.
- If two or more NQ values occur in succession between measurable concentrations, the profile
  will be deemed to have terminated at the last measurable concentration prior to these NQs.
  For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent
  measurable concentrations will be retained. For the derivation of pharmacokinetic parameters,
  these NQs and any subsequent measurable concentrations will be set to missing.
- NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters and from the individual subject plots.
- Individual's PK parameters reported as 'NC' (Not Calculable) or 'ND' (Not Determined) will be
  included in listings but omitted (set to missing) from figures, summaries and statistical
  analyses.

# 10.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

### 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion was defined as a participant has completed all periods of the study including the last visit or the last scheduled procedure (Follow-up) for each period as described in the protocol. |
| | Withdrawn subjects maybe replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |

# 10.6.3. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 10.6.4. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|------------|--------------------------------------------------|
| Imputation | No imputation will be performed for missing data |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. Laboratory Values (Healthy Volunteers)

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | -// | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |
## 10.7.2. ECG (Healthy Volunteers)

| ECG Parameter | Units | Clinical Cor | ncern Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | > 450 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | > 60 [1] | |

### NOTES:

## 10.7.3. Vital Signs (Healthy Volunteers)

| Vital Sign Parameter Units | | Clinical Concern Range | |
|----------------------------|------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>1.</sup> Represent standard ECG values of PCI for HV studies

# 10.8. Appendix 8 - Abbreviations & Trade Marks

### 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| AUC(0-24) | Area under the concentration-time curve from pre-dose to 24 hours |
| AUC(0-inf) | Area under the concentration-time curve from time zero (pre-dose) |
| | extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to |
| () | last time of quantifiable concentration within a subject across all |
| | treatments |
| BMI | Body mass index |
| BP | Blood pressure |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CSR | Clinical Study Report |
| CVb | Coefficient of variation (Between) |
| CVw | Coefficient of Variation (Within) |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| GSK | GlaxoSmithKline |
| HR | Heart rate |
| hrs | Hours |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| LLN | Lower Limit of Normal |
| LLQ | Lower Limit of Quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MG | Milligrams |
| msec | Milliseconds |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event(s) |
| SAS | Statistical Analysis Software |
| SD | Standard Deviation |
| ULN | Upper Limit of Normal |
| SOP | Standard Operation Procedure |
| t1/2 | Terminal half-life |
| Tmax | Time to maximum observed blood drug concentration |
| TFL | Tables, Figures & Listings |

### 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| None | SAS |
| | WinNonlin |

### 10.9. Appendix 9: List of Data Displays

### 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------------------|---------|
| Study Population | 1.1 to 1.14 | N/A |
| Safety | 2.1 to 2.34 | N/A |
| Pharmacokinetic | 3.1 to 3.8 3.1 to 3.10 | |
| Section | Listings | |
| ICH Listings | 1 to 71 | |
| Other Listings | N/A | |

### 10.9.2. Mock Example Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

• Indicate display is Non-Standard in the 'IDSL/TST ID / Example Shell' or 'Programming Notes' column.

### 10.9.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------|
| PR [1] | Primary Report (Part 1 only) |
| SAC [2] | Statistical Analysis Complete |

### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

## 10.9.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | CP_ES1 | Summary of Subject Disposition (Part 1) | Completed or withdrawn and the reason for withdrawal. | PR [1] |
| 1.2. | Safety | ES4 | Summary of Subject Disposition at each period (Part 1) | Completed or withdrawn at each period. | PR [1] |
| 1.3. | Safety | CP_ES1 | Summary of Subject Disposition (Part 2) | Completed or withdrawn and the reason for withdrawal. | SAC [2] |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | The number (%) of Randomized or screening failure subjects as the screening status, and the reason for screening failure. | SAC [2] |
| Protoc | ol Deviation | | | | |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations (Part 1) | Data is from DV1 dataset. | PR [1] |
| 1.6. | Safety | DV1 | Summary of Important Protocol Deviations (Part 2) | Data is from DV1 dataset. | SAC [2] |
| Popula | tion Analysed | | | | |
| 1.7. | Safety | SP1 | Summary of Study Populations (Part 1) | Only PK population is summarized. | PR [1] |
| 1.8. | Safety | SP1 | Summary of Study Populations (Part 2) | Only PK population is summarized. | SAC [2] |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.9. | Safety | DM3 | Summary of Demographic Characteristics (Part 1) | | PR [1] |
| 1.10. | Safety | DM3 | Summary of Demographic Characteristics (Part 2) | | SAC [2] |
| 1.11. | Screened | DM11 | Summary of Age Ranges (Part 1) | <=17 years, 18-64 years, 65-84 years, >=85 years | PR [1] |
| 1.12. | Screened | DM11 | Summary of Age Ranges (Part 2) | <=17 years, 18-64 years, 65-84 years, >=85 years | SAC [2] |

| Study F | Study Population Tables | | | |
|---|---|---|---|---|
| No. Population Little Programming Notes | | | | Deliverable<br>[Priority] |
| 1.13. | Safety | DM5 | Summary of Race and Racial Combinations (Part 1) | PR [1] |
| 1.14. | Safety | DM5 | Summary of Race and Racial Combinations (Part 2) | SAC [2] |

# 10.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 1) | | PR [1] |
| 2.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity (Part 1) | | PR [1] |
| 2.3. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term (Part 1) | | PR [1] |
| 2.4. | Safety | AE5A | Summary All Drug-Related Adverse Events by Maximum Intensity (Part 1) | | PR [1] |
| 2.5. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term (Part 2) | | SAC [2] |
| 2.6. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity (Part 2) | | SAC [2] |
| 2.7. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term (Part 2) | | SAC [2] |
| 2.8. | Safety | AE5A | Summary All Drug-Related Adverse Events by Maximum Intensity (Part 2) | | SAC [2] |
| Labora | tory: Chemistry | / | | | |
| 2.9. | Safety | LB1 | Summary of Chemistry (Part 1) | | PR [1] |
| 2.10. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 1) | | PR [1] |
| 2.11. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 1) | | PR [1] |
| 2.12. | Safety | LB1 | Summary of Chemistry (Part 2) | | SAC [2] |
| 2.13. | Safety | LB1 | Summary of Chemistry Changes from Baseline (Part 2) | | SAC [2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline with Respect to the Normal Range (Part 2) | | SAC [2] |
| Labora | tory: Hematolo | gy | | | |
| 2.15. | Safety | LB1 | Summary of Hematology (Part 1) | | PR [1] |
| 2.16. | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 1) | | PR [1] |
| 2.17. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 1) | | PR [1] |
| 2.18. | Safety | LB1 | Summary of Hematology (Part 2) | | SAC [2] |
| 2.19. | Safety | LB1 | Summary of Hematology Changes from Baseline (Part 2) | | SAC [2] |
| 2.20. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline with Respect to the Normal Range (Part 2) | | SAC [2] |
| Labora | tory: Urinalysis | <b>5</b> | | | |
| 2.21. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 1) | | PR [1] |
| 2.22. | Safety | LB1 | Summary of Urinalysis Data (Specific Gravity and pH) (Part 1) | | PR [1] |
| 2.23. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) (Part 2) | | SAC [2] |
| 2.24. | Safety | LB1 | Summary of Urinalysis Data (Specific Gravity and pH) (Part 2) | | SAC [2] |
| ECG | | | | | |
| 2.25. | Safety | EG1 | Summary of ECG Findings (Part 1) | | PR [1] |
| 2.26. | Safety | EG2 | Summary of ECG Value (Part 1) | | PR [1] |
| 2.27. | Safety | EG2 | Summary of Change from Baseline in ECG Values (Part 1) | | PR [1] |
| 2.28. | Safety | EG1 | Summary of ECG Findings (Part 2) | | SAC [2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.29. | Safety | EG2 | Summary of ECG Value (Part 2) | | SAC [2] |
| 2.30. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit (Part 2) | | SAC [2] |
| Vital Si | gns | | | | |
| 2.31. | Safety | VS1 | Summary of Vital Signs (Part 1) | | PR [1] |
| 2.32. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 1) | | PR [1] |
| 2.33. | Safety | VS1 | Summary of Vital Signs (Part 2) | | SAC [2] |
| 2.34. | Safety | VS1 | Summary of Change from Baseline in Vital Signs (Part 2) | | SAC [2] |

### 10.9.6. Pharmacokinetic Tables

| Pharma | acokinetic: Tabl | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part 1 | | | | | |
| 3.1. | PK | PK01: pkct1 | Summary of GSK1325756 Blood Concentration (ng/mL) (Part 1) | | PR [1] |
| 3.2. | PK | PK03: pkpt1 | Summary of GSK1325756 Pharmacokinetic Parameters (non-transformed) (Part 1) | | PR [1] |
| 3.3. | PK | PK05: pkpt3 | Summary of GSK1325756 Pharmacokinetic Parameters (loge-transformed) (Part 1) | | PR [1] |
| 3.4. | PK | Study Specific (PK_T1) | Analysis of Power Model Analysis for GSK1325756 Dose<br>Proportionality of Pharmacokinetic Parameters (AUC(0-t),<br>Cmax) (Part 1) | Parameter, Effect, n, Point estimate of Slope, SE, 90% CI | PR [1] |
| Part 2 | | | | | |
| 3.5. | PK | PK01: pkct1 | Summary of GSK1325756 Blood Concentration (ng/mL) (Part 2) | | SAC [2] |
| 3.6. | PK | PK03: pkpt1 | Summary of GSK1325756 Pharmacokinetic Parameters (non-transformed) (Part 2) | | SAC [2] |
| 3.7. | PK | PK05: pkpt3 | Summary of GSK1325756 Pharmacokinetic Parameters (loge-transformed) (Part 2) | | SAC [2] |
| 3.8. | PK | Study Specific (PK_T2) | Analysis of food effect for Pharmacokinetic Parameters (AUC(0-t), Cmax) (Part 2) | n, Geometric mean of Fasted and Fed, ratio (Fasted/Fed), 90% Cl and CVw(%) | SAC [2] |

# 10.9.7. Pharmacokinetic Figures

| Pharma | acokinetic: Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Part 1 | 1 | | | | |
| 3.1. | PK | PK16b: pkcf1x | Individual GSK1325756 Blood Concentration-Time Plots by Subject (Part 1) | By Subject (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | PR [1] |
| 3.2. | PK | PK24: pkcf6 | Individual GSK1325756 Blood Concentration-Time Plots by treatment (Part 1) | By Treatment (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | PR [1] |
| 3.3. | PK | Study Specific (PK_F1) | Mean (+SD) GSK1325756 Blood Concentration-Time Plots (Part 1) | Unit of x-axis is Hours | PR [1] |
| 3.4. | PK | PK18: pkcf3 | Median GSK1325756 Blood Concentration-Time Plots (Part 1) | Unit of x-axis is Hours | PR [1] |
| 3.5. | PK | PK28 | Plot of GSK1325756 Treatment and PK Parameters (AUC (0-t), Cmax) (Part 1) | | PR [1] |
| Part 2 | | | | | |
| 3.6. | PK | PK16b: pkcf1x | Individual GSK1325756 Blood Concentration-Time Plots by Subject (Part 2) | By Subject (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | SAC [2] |
| 3.7. | PK | PK24: pkcf6 | Individual GSK1325756 P Blood Concentration-Time Plots by Treatment (Part 2) | By Treatment (Linear and Semi-Log). Actual time is used. Unit of x-axis is Hours. | SAC [2] |
| 3.8. | PK | Study Specifics (PK_F1) | Mean (+SD) GSK1325756 Blood Concentration-Time Plots (Part 2) | Unit of x-axis is Hours | SAC [2] |
| 3.9. | PK | PK18: pkcf3 | Median GSK1325756 Blood Concentration-Time Plots (Part 2) | Unit of x-axis is Hours | SAC [2] |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | PK | PK28 | Plot of GSK1325756 Treatment and PK Parameters (AUC(0-t), Cmax) (Part 2) | | SAC [2] |

# 10.9.8. ICH Listings

Note: 'Inv.' in the standard displays will be replaced to 'Centre'.

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1. | Screening<br>Failure | ES7 | Listing of Reasons for Screen Failure | | SAC [2] |
| 2. | Safety | CP-ES10x | Listing of Reasons for Study Withdrawal (Part 1) | | PR [1] |
| 3. | Safety | CP-ES10x | Listing of Reasons for Study Withdrawal (Part 2) | | SAC [2] |
| 4. | Safety | BL2 | Listing of Subjects for Whom the Treatment Blind was Broken (Part 1) | | PR [1] |
| 5. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 1) | | PR [1] |
| 6. | Safety | TA2 | Listing of Planned and Actual Treatments (Part 2) | | SAC [2] |
| Protoco | ol Deviations | | | | |
| 7. | Safety | DV2 | Listing of Important Protocol Deviations (Part 1) | Column for Treatment Sequence/Period of Protocol deviation will be displayed after Centre./Subj. Period day will be displayed in the same column of Date of Deviation/Study day. | PR [1] |
| 8. | Safety | DV2 | Listing of Important Protocol Deviations (Part 2) | | SAC [2] |
| 9. | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [2] |
| Popula | tions Analysed | | | | |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10. | Safety | Study Specifics (POP_L1) | Listing of Subjects Excluded from PK Population (Part 1) | | PR [1] |
| 11. | Safety | Study Specifics (POP_L1) | Listing of Subjects Excluded from PK Population (Part 2) | | SAC [2] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 12. | Safety | DM4 | Listing of Demographic Characteristics (Part 1) | "Age at Screening" is added. | PR [1] |
| 13. | Safety | DM4 | Listing of Demographic Characteristics (Part 2) | "Age at Screening" is added. | SAC [2] |
| 14. | Screening<br>Failure | DM4 | Listing of Demographic Characteristics for Screening Failure Subjects | | SAC [2] |
| 15. | Safety | DM10 | Listing of Race (Part 1) | | PR [1] |
| 16. | Safety | DM10 | Listing of Race (Part 2) | | SAC [2] |
| 17. | Screening<br>Failure | DM10 | Listing of Race for Screening Failure Subjects | Treatment is not needed to display. | SAC [2] |
| Medica | l Conditions ar | d Concomitant M | edications | | • |
| 18. | Screened | MH3 | Listing of Medical Conditions | | SAC [2] |
| 19. | Safety | CM5 | Listing of Concomitant Medications (Part 1) | | PR [1] |
| 20. | Safety | CM5 | Listing of Concomitant Medications (Part 2) | | SAC [2] |
| 21. | Screened | CM6 | Listing of Relationship between ATC Level 1, Ingredient and Verbatim Text | | SAC [2] |
| Expos | ure and Treatmo | ent Compliance | | <u> </u> | |
| 22. | Safety | EX4 | Listing of Exposure Data (Part 1) | | PR [1] |
| 23. | Safety | EX4 | Listing of Exposure Data (Part 2) | | SAC [2] |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Meal | | | | | |
| 24. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days (Part 1) | | PR [1] |
| 25. | Safety | CP_ML1x | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days (Part 2) | | SAC [2] |
| Advers | e Events | | | • | • |
| 26. | Safety | AE9CP | Listing of All Adverse Events (Part 1) | | PR [1] |
| 27. | Safety | AE9CP | Listing of All Adverse Events (Part 2) | | SAC [2] |
| 28. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 1) | | PR [1] |
| 29. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events (Part 2) | | SAC [2] |
| 30. | Screened | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC [2] |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 31. | Safety | AE9CP | Listing of Serious Adverse Events (Part 1) | | PR [1] |
| 32. | Safety | AE9CP | Listing of Serious Adverse Events (Part 2) | | SAC [2] |
| 33. | Screening<br>Failure | AE9CP | Listing of Serious Adverse Events for Screening Failure Subject | Treatment is not needed to display. | SAC [2] |
| 34. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 1) | | PR [1] |
| 35. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study (Part 2) | | SAC [2] |
| Labora | tory (Chemistry | / Data) | | | |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 36. | Safety | CP_LB6 | Listing of All Chemistry Data (Part 1) | Listing of All Chemistry Data (Part 1) Change from baseline is included. | |
| 37. | Safety | CP_LB6 | Listing of All Chemistry Data (Part 2) | Change from baseline is included. | SAC [2] |
| 38. | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 39. | Safety | CP_LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Labora | tory (Hematolo | gy Data) | | | |
| 40. | Safety | CP_LB6 | Listing of All Hematology Data (Part 1) | Change from baseline is included. | PR [1] |
| 41. | Safety | CP_LB6 | Listing of All Hematology Data (Part 2) | Change from baseline is included. | SAC [2] |
| 42. | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 43. | Safety | CP_LB6 | Listing of All Hematology Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Labora | tory (Urinalysis | Data) | | | |
| 44. | Safety | UR2b | Listing of All Urinalysis Dipstick and Microscopy Data(Part 1) | Time will be displayed after 'Date'. | PR [1] |
| 45. | Safety | CP_LB6 | Listing of Urinalysis Data (Gravity and pH) (Part 1) | | PR [1] |
| 46. | Safety | UR2b | Listing of All Urinalysis Dipstick and Microscopy Data (Part 2) | Time will be displayed after 'Date'. | SAC [2] |
| 47. | Safety | CP_LB6 | Listing of Urinalysis Data (Gravity and pH) (Part 2) | | SAC [2] |
| Hepato | biliary (Liver) | | | | |
| 48. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 1) | Column for Treatment/Period will be displayed after the column for Age/Sex/Race Detail. | PR [1] |
| 49. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting (Part 2) | | SAC [2] |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 50. | Safety | МН3 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part 1) | | PR [1] |
| 51. | Safety | МН3 | Listing of Medical Conditions for Subjects with Liver Stopping Events (Part 2) | | SAC [2] |
| 52. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 1) | | PR [1] |
| 53. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events (Part 2) | | SAC [2] |
| ECG | | | | | • |
| 54. | Safety | CP_EG4 | Listing of All ECG Values (Part 1) | | PR [1] |
| 55. | Safety | CP_EG4 | Listing of All ECG Values (Part 2) | | SAC [2] |
| 56. | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 1) | | PR [1] |
| 57. | Safety | CP_EG4 | Listing of Change from Baseline in ECG Values (Part 2) | | SAC [2] |
| 58. | Safety | CP_EG6 | Listing of ECG Findings (Part 1) | | PR [1] |
| 59. | Safety | CP_EG6 | Listing of ECG Findings (Part 2) | | SAC [2] |
| 60. | Safety | CP_EG4 | Listing of All ECG Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |
| 61. | Safety | CP_EG4 | Listing of All ECG Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Vital Si | gns | | | | |
| 62. | Safety | CP_VS5 | Listing of All Vital Signs (Part 1) | Change from baseline is included. | PR [1] |
| 63. | Safety | CP_VS5 | Listing of All Vital Signs (Part 2) | Change from baseline is included. | SAC [2] |
| 64. | Safety | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 1) | | PR [1] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 65. | Safety | CP_VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance (Part 2) | | SAC [2] |
| Others | | | | | |
| 66. | Safety | Study Specifics<br>(SAFE_L1) | Listing of Ophthalmic examinations (Part 1) | | PR [1] |
| 67. | Safety | Study Specifics (SAFE_L1) | Listing of Ophthalmic examinations (Part 2) | | SAC [2] |
| PK | | | | | |
| 68. | PK | PK08: pkcl1x | Listing of GSK1325756 Blood Concentration (Part 1) | | PR [1] |
| 69. | PK | PK08: pkcl1x | Listing of GSK1325756 Blood Concentration (Part 2) | | SAC [2] |
| 70. | PK | PK14: pkpl1x | Listing of GSK1325756 Pharmacokinetic Parameters (Part 1) | | PR [1] |
| 71. | PK | PK14: pkpl1x | Listing of GSK1325756 Pharmacokinetic Parameters (Part 2) | | SAC [2] |

206817

- 10.10. Appendix 10: Example Mock Shells for Data Displays
- 10.10.1. Study population

206817


Example CP\_ES1 (XO studies)
Protocol: GSK123456

Population: xxxxx

### Table x.x

| | Tota | al |
|-----------------------------------------|------|-------|
| | (N=) | 100) |
| Completion Status | | |
| Completed | 50 | (50%) |
| Withdrawn | 50 | (50%) |
| Primary*/subreason^ for withdrawal | | |
| Adverse event | 10 | (10%) |
| Elevated ALT levels | 2 | (2%) |
| Severe vomiting | 5 | (5%) |
| Lack of efficacy | 0 | |
| Protocol deviation | 0 | |
| Subject reached stopping criteria | 10 | (10%) |
| CD4 levels below continuation threshold | 10 | (10%) |
| Study closed/terminated | 0 | |
| Lost to follow-up | 0 | |
| Investigator discretion | 0 | |
| Withdrew consent | 30 | (30%) |
| Burden of procedures | 10 | (10%) |
| Pursue alternative treatment | 20 | (20%) |
| Other | 0 | |

206817

Example: ES4


Population: xxxxx

### 

| Phase | | Not Randomized (N=10) | Placebo<br>(N=100) | Curitol<br>10mg<br>(N=100) |
|---|---|---|---|---|
| Screening | Entered<br>Completed | 10 (100%)<br>0 | 100 (100%)<br>100 (100%) | 100 (100%)<br>100 (100%) |
| | Withdrawn | 10(100%) | 0 | 0 |
| Double blind | Entered | | 100 (100%) | 100 (100%) |
| | Completed | | 50 (50%) | 50 (50%) |
| | Withdrawn | | 50 (50%) | 50 (50%) |
| Follow-up | Entered | | 50 (50%) | 50 (50%) |
| | Completed | | 50 (50%) | 50 (50%) |
| | Withdrawn | | 0 | 0 |

206817


Example: ES6 (SF for CONSORT)

Protocol: GSK123456

Population: xxxxx

### 

| | Screened<br>Subjects<br>(N=100) |
|---|---|
| Screening Status | |
| ENROLLED | 50 (50%) |
| FAILED | 50 (50%) |
| Reason(s) for Failure DID NOT MEED INCLUSION/EXCLUSION CRITERIA | 25 (25%) |
| STUDY CLOSED/TERMINATED | 25 (25%)<br>5 (5%) |
| • | ` ' |
| PHYSICIAN DECISION | 10 (10%) |
| PROTOCOL DEVIATION | 10 (10%) |

206817

Example: CP\_ES10x Protocol: GSK123456 Population: xxxxx


### Listing x.x

### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| | Treatment | Last | Date of Withdrawal/ Study Day of Withdrawal/ | | | Date of Last |
|---|---|---|---|---|---|---|
| Centre | Sequence/ | Treatment | Period Day | | | Contact/ |
| ID/ | Period of | Before | of | Primary Reason | Subreason for | Study Day of |
| Subj. | Withdrawal | Withdrawal | Withdrawal | for Withdrawal | Withdrawal | Last Contact |
| xxxxxx/ | PAB/ | А | DDMMMYYYY/ | Adverse Event | Elevated ALT levels | DDMMMYYYY/ |
| XXX | Period 1 | | xx/ | | | X |
| | | | X | | | |
| xxxxxx/ | BPC/ | В | DDMMMYYYY/ | | | DDMMMYYYY/ |
| XXX | Period 2 | | x/ | | | X |
| | | | X | | | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: ES7 (for SF)
Protocol: GSK123456
Population: xxxxx


### Listing x.x

### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID/ | Date of<br>Screen | |
|---|---|---|
| Subj. | Failure | Reason Term(s) for Screen Failure |
| xxxxxx/<br>xxx | DDMMMYYYY | DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| xxxxxx/<br>xxx | DDMMMYYYY | PHYSICIAN DECISION DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| xxxxxx/<br>xxx | DDMMMYYYY | DID NOT MEED INCLUSION/EXCLUSION CRITERIA |
| | DDMMMYYYY | PHYSICIAN DECISION |

206817

Example: BL2 (for XO studies)


# Population: xxxxx Listing x.x

### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID | Subj. | Sequence/<br>Treatment<br>when Blind<br>broken | Date<br>Blind<br>Broken | Time<br>Blind<br>Broken | Study<br>Day | Period<br>Day | Reason |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | PBC/<br>Treatment A | DDMMMYYYY | hh:ss | XX | X | Other: PT REQUESTED TO KNOW<br>FOR MEDICAL REASONS |
| XXXXXX | XXXX | APC/<br>Treatment C | DDMMMYYYY | hh:ss | XX | XX | Medical Emergency |

206817

Example: TA2 (for XO studies)

Population: xxxxx

### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

Country: Canada
Centre ID: PPD
Investigator: PPD

| Subject<br>ID | Randomization<br>Number | Randomization Date | Period | Randomization<br>Treatment | Actual Treatment | Deviation |
|---|---|---|---|---|---|---|
| PPD | | 01JAN08 | 1 | Curital 10mg | Curital 10mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Placebo | No treatment | Y |
| | | | 4 | Curital 20mg | No treatment | Y |
| | | 03JAN08 | 1 | Curital 20mg | Curital 20mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Curital 10mg | Curital 10mg | |
| | | | 4 | Placebo | Placebo | |
| | | 01FEB08 | 1 | Placebo | Placebo | |
| | | OIFEBOO | | | | |
| | | | 2 | Curital 10mg | Curital 10mg | |
| | | | 3 | Placebo | Placebo | |
| | | | 4 | Curital 20mg | Curital 10mg | Y |
| | | 15FEB08 | 1 | Curital 10mg | Curital 10mg | |
| | | | 2 | Placebo | Placebo | |
| | | | 3 | Placebo | Placebo | |
| | | | 4 | Curital 10mg | Curital 20mg | Y |

206817

Example: IE4 (for XO studies)

Population: xxxxx

Listing x.x

### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID | Subj. | Treatment sequence | Type | Criterion |
|---|---|---|---|---|
| xxxxxx | XXX | APC | INCLUSION | Is the subject 18 years of age or older? |
| xxxxx | XXX | PAB | EXCLUSION | Has the subject had an asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to Visit 1? |

206817

Example: DV1


Population: xxxxx

### 

| Category/Coded Term | _ | tal<br>=200) |
|---|---|---|
| Any important protocol deviations | 60 | (30%) |
| Informed consent WRONG INFORMED CONSENT/ASSENT VERSION SIGNED | | (5%)<br>(5%) |
| Eligibility criteria not met | 14 | (7%) |
| Not withdrawn after developing withdrawal criteria Not discontinued from study treatment Not withdrawn from study | 10 | (9%)<br>(5%)<br>(4%) |
| EXCLUDED MEDICATION, VACCINE OR DEVICE MEDICATION, EXCLUDED BY THE PROTOCOL, WAS ADMINISTERED | | (2%)<br>(2%) |
| Assessment or time point completion OUT OF WINDOW EFFICACY ASSESSMENT | | (1응)<br>(1응) |
| WRONG STUDY TREATMENT/ADMINISTRATION/DOSE<br>STUDY TREATMENT NOT ADMINISTERED PER PROTOCOL<br>EXPIRED STUDY TREATMET ADMINISTERED | 2 | (2%)<br>(1%)<br>(1%) |
| Failure to report SAFETY EVENTS PER Protocol<br>SAE NOT REPORTED WITHIN THE EXPECTED TIME FRAME<br>LIVER FUNCTION ABNORMALITIES PER PROTOCOL | 4 | (5%)<br>(2%)<br>(2%) |

206817

Example: DV2

Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
|---|---|---|---|---|---|---|
| | | | Deviation Requires Exclusion from | | | |
| Site Id./ | Date of<br>Deviation/ | Category/<br>Coded Term | Term | Intent to Treat Population | Safety<br>Population | Per<br>Protocol<br>Population |
| PPD | PPD 28 | ILURE TO REPORT SAFETY EVENTS PER PROTOCOL / SAE NOT REPORTED WITHIN THE EXPECTED TIME FRAME | SAE OF FEVER WITH SEVERE CHILLS REQUIRING IV HYDRATION WAS NOT REPORTED TO GSK WITHIN 24 HOURS. | | | |
| | 31 | ELIGIBILITY CRITERIA<br>NOT MET / ELIGIBILITY<br>CRITERIA NOT MET | SUBJECT SCREEN<br>FAILED BUT WAS<br>RANDOMIZED IN<br>ERROR. | | Y | Y |
| | PPD<br>1 | WRONG STUDY TREATMENT/ ADMINISTRATION/DOSE / STUDY TREATMENT NOT ADMINISTERED PER PROTOCOL | SUBJECT MISSED<br>WEEK 8<br>TREATMENT | | | |
| | <b>PPD</b> 2 | WRONG STUDY TREATMENT/<br>ADMINISTRATION/DOSE /<br>STUDY TREATMENT NOT<br>ADMINISTERED PER<br>PROTOCOL | INTERRUPTION OF IP FOR GREATER THAN 20 PERCENT OF TIME | | | Y |

206817

Example: SP1


Population: xxxxx

### 

| Population | No Treatment (N=50) | Placebo<br>(N=xxx) | Treatment 1 (N=200) | Treatment 2 (N=250) | Total<br>(N=500) |
|---|---|---|---|---|---|
| Screened | 50 (100%) | xx (xxx%) | 200 (100%) | 250 (100%) | 500 (100%) |
| Enrolled | 10 (20%) | xx (xxx%) | 200 (100%) | 250 (100%) | 460 (92%) |
| Randomized | 5 (10%) | xx (xx%) | 200 (100%) | 250 (100%) | 455 (91%) |
| Safety | | xx (xx%) | 195 (98%) | 245 (98%) | 440 (88%) |
| PK | | xx (xx%) | 200 (100%) | 250 (100%) | 455 (91%) |

206817


Example: POP\_L1
Protocol: GSK123456

Population: xxxxx (Randomised subjects)

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Centre ID/<br>Subj. | Treatment sequence | PK<br>population |
|---------------------|--------------------|------------------|
| xxxxxx/<br>xxx | ABC | Y |
| xxxxxx/<br>xxx | СВА | Υ |
| xxxxxx/<br>xxx | BAC | Y |

206817

Example: DM3 (for XO studies)

Protocol: GSK123456
Population: xxxxx


### 

| | Total<br>(N=100) |
|------------------------|------------------|
| Sex | |
| n | 100 |
| F | 50 (50%) |
| M | 50 (50%) |
| Age (YEARS)[1] | |
| n | 100 |
| Mean | 50.0 |
| SD | 10.00 |
| Median | 50.0 |
| Min. | 18 |
| Max. | 65 |
| Age Group(YEARS)[1] | |
| <=18 | 5 (5%) |
| 19-64 | 50 (50%) |
| >=65 | 45 (45%) |
| Ethnicity | |
| n | 100 |
| HISPANIC OR LATINO | 10 (10%) |
| NOT HISPANIC OR LATINO | 90 (90%) |


Example: DM3 (continued) Protocol: GSK123456

Population: xxxxx

#### Table x.x XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX

Total (N=100)Race Detail AMERICAN INDIAN OR ALASKA NATIVE 1 (1%) ASIAN - CENTRAL/SOUTH ASIAN HERITAGE 3 (3%) ASIAN - EAST ASIAN HERITAGE 4 (4%) ASIAN - JAPANESE HERITAGE 3 (3%) ASIAN - SOUTH EAST ASIAN HERITAGE (1%) BLACK OR AFRICAN AMERICAN (2%) NATIVE HAWAIIAN OR OTHER PACIFIC 59 (59%) ISLANDER WHITE - ARABIC/NORTH AFRICAN HERITAGE 26 (26%) WHITEWHITE/CAUSASIAN/EUROPEAN 1 (1%) *HERITAGE* MIXED ASIAN RACE 1 (1%) 1 (1%) MIXED WHITE RACE MULTIPLE1 (1%) Height (cm) 100 n Mean 150.0 10.00 SD Median 50.0 Min. 18 65

USER ID: directory/program.sas DDMMMYYYY hh:mm

Max.

206817


Example: DM3 (continued)

Protocol: GSK123456
Population: xxxxx

### 

USER ID: directory/program.sas DDMMMYYYY hh:mm

Options (units)

206817

Example: DM4 (for XO studies)


Population: xxxxx

### 

| Centre ID/<br>Subj. | Treatment<br>Sequence | Partial<br>Date of<br>Birth | Age<br>(YEARS)<br>[1] | Sex | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Option (unit) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx/<br>xxx | ABC | MMYYYY | xx | F | HISPANIC OR LATINO | xxx | XX | |
| xxxxxx/<br>xxx | BCA | MMYYYY | xx | М | NOT HISPANIC OR LATINO | XXX | xx | |
| xxxxxx/<br>xxx | CAB | | xx | М | NOT HISPANIC OR LATINO | xxx | xx | |

206817

Example: DM5


Population: xxxxx

# Table x.x Xxxxxxxxxxxxxxxxxxxxxxxx

| | | Treatment A (N=XXX) | | Treatment B (N=XXX) | | Total<br>(N=XXX) | |
|---|---|---|---|---|---|---|---|
| Race | n | 100 | | 100 | | 200 | |
| | African American/African Heritage | 30 | (30%) | 30 | (30%) | 60 | (30%) |
| | American Indian or Alaskan Native | 0 | | 0 | | 0 | |
| | Asian | 15 | (15%) | 15 | (15%) | 30 | (15%) |
| | Central/South Asian Heritage | 3 | (3%) | 3 | (3%) | 6 | (3%) |
| | Japanese/East Asian Heritage/South | 11 | (11%) | 11 | (11%) | 22 | (11%) |
| | East Asian Heritage | | | | | | |
| | Mixed Asian Heritage | 1 | (1%) | 1 | (1%) | 2 | (1%) |
| | Native Hawaiian or other Pacific | 10 | (10%) | 10 | (10%) | 20 | (10%) |
| | Islander | | | | | | |
| | White | 35 | (35%) | 35 | (35%) | 70 | (35%) |
| | Native Hawaiian or other Pacific | 2 | (2%) | 2 | (2%) | 4 | (4%) |
| | Islander & American Indian or Alaskan | | | | | | |
| | Native | | | | | | |
| | White & African American/African | 3 | (3%) | 3 | (3%) | 6 | (3%) |
| | Heritage | | | | | | |
| | White & Asian | 5 | (5%) | 5 | (5%) | 10 | (5%) |
206817

Example: DM11


Population: xxxxx

#### 

| | No Treatment | Total |
|---|---|---|
| | (N=1) | (N=201) |
| Age Ranges [1] In utero Preterm newborn infants (gestational age <37 weeks) | 0 0 | 4 (2%)<br>2 (1%) |
| Newborns (0-27 days) Infants and toddlers (28 days-23 months) Children (2-11 years) | 0<br>0<br>0 | 6 (3%)<br>8 (4%)<br>6 (3%) |
| Adolescents (12-17 years) Adult (18-64 years) >=65-84 years | 0 0 0 | 2 (1%)<br>118 (59%)<br>52 (26%) |
| >=85 years | 1 (100%) | 3 (1%) |

206817

Example: DM10 (for XO studies)

Protocol: GSK123456
Population: xxxxx

# Page 1 of n

#### 

| Centre<br>ID | Subj. | Treatment sequence | Race | Race Detail |
|---|---|---|---|---|
| xxxxxx | XXX | ABC<br>BCA | BLACK OR AFRICAN AMERICAN<br>Mixed race | BLACK OR AFRICAN AMERICAN<br>ASIAN - EAST ASIAN HERITAGE<br>ASIAN - JAPANESE HERITAGE |
| | XXX | CAB | WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE | WHITE - ARABIC/NORTH AFRICAN HERITAGE |
| | XXX | ABC | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE |
| xxxxxx | XXX | ABC | Mixed race | WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAG<br>ASIAN - JAPANESE HERITAGE |
| | XXX | BCA | NATIVE HAWAIIAN OR OTHER PACIFIC<br>ISLANDER | NATIVE HAWAIIAN OR OTHER PACIFIC<br>ISLANDER |
| | XXX | CAB<br>ABC | BLACK OR AFRICAN AMERICAN<br>WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE | BLACK OR AFRICAN AMERICAN<br>WHITE - ARABIC/NORTH AFRICAN<br>HERITAGE |
| xxxxx | xxx<br>xxx | BCA<br>CAB | AMERICAN INDIAN OR ALASKA NATIVE<br>Mixed race | AMERICAN INDIAN OR ALASKA NATIVE<br>BLACK OR AFRICAN AMERICAN<br>WHITE - WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE |

206817

Example: MH3


Population: xxxxx Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv. | Subject | Treatment<br>Sequence | Classification | Condition | Status |
|---|---|---|---|---|---|
| PPD | | AB | Hepatobiliary<br>Psychiatric | HEPATITIS A PARANOIA COMBINED WITH MANIA. | Current<br>Past |
| | | AB | Eye | ASTIGMATISM | Current |
| | | BA | Metabolism and nutrition | RICKETS | Current |

206817

Example: CM5

Population: xxxxx

Listing x.x

| Inv./<br>Subj./<br>Seq | Treat-<br>ment/<br>Period | ATC Level 1/<br>Ingredient/<br>Verbatim Text/<br>Indication | Dose/<br>Units/<br>Freq/<br>Route | Start<br>Date/Time<br>Study Day/<br>Period Day | Stop<br>Date/Time<br>Study Day/<br>Period Day | Started<br>Pre-<br>Trial? | Ongoing<br>Medi-<br>cation? |
|---|---|---|---|---|---|---|---|
| PPD | Tmt A/<br>Per 1 | Endocrine & metabolic/<br>Fluticasone propionate/ | 2/<br>MG/ | PPD<br>12:30/ | | | Y |
| ABC | | FLIXOTIDE/ Asthma | 2XD/<br>IH | 15/<br>7 | | | |

206817

Example: CM6

Population: xxxxx

Listing x.x

| ATC Level 1 | Ingredient | Verbatim Text |
|---|---|---|
| Endocrine & metabolic | Fluticasone Propionate<br>Prednisolone | FLIXOTIDE<br>PREDNISOLONE |
| Drugs acting via the nervous system | Paracetamol | PANADOL<br>CHILDREN'S PANADOL 1-5YERS |

USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: EX4


#### 

| Centre<br>ID | Subj. | Treatment | Start<br>Date/<br>Start Time<br>of Dose | Stop Date/<br>Stop Time<br>of Dose | Duration<br>(days) | Dose | | Formulat ion/Route | Freque<br>ncy | Cumulat<br>ive<br>Dose |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | Treatment A | DDMMMYYYY/ hh:ss DDMMMYYYY/ | DDMMMYYYY/<br>hh:ss | xx | xx<br>xx | mg<br>mg | Tablet/<br>Oral<br>Tablet/ | 1xday<br>1xday | |
| | | Treatment C | hh:ss<br>DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Oral<br>Tablet/<br>Oral | 1xday | |
| | PPD | Placebo Treatment B | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Treatment C | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Treatment A Placebo | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |
| | | Treatment B | DDMMMYYYY/<br>hh:ss | DDMMMYYYY/<br>hh:ss | XX | XX | mg | Tablet/<br>Oral | 1xday | |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_ML1x Protocol: GSK123456 Population: xxxxx


# Listing x.x Xxxxxxxxxxxxxxxxxxxxx

| Cohort<br>(Optional) | Investigator OR Centre ID (Optional) | Subj. | Treatment | Meal type (Optional) | Period<br>(Optional)<br>/Visit | <u>Visit</u><br>Date | <u>Dose</u><br>Time | Meal<br>Start<br>Time | Meal End Time<br>(Optional) | mir<br>Mea<br>(Op |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 50mg | High-fat | Period | | | | | |
| 1 | PPD | | GSK123456<br>25mg | breakfast<br>High-fat | 2/Day 4<br>Period | PPD | 8:13 | 7:30 | 7:41 | Y |
| | | | GSK123456 | breakfast | 2/Day 4 | | 8:12 | 7:28 | 7:42 | Y |
| | | | 10mg<br>GSK123456 | High-fat<br>breakfast | Period<br>2/Day 4 | | 8:10 | 7:27 | 7:35 | Y |
| | | | 50mg | High-fat | Period | | | | | |
| 2 | | | GSK123456<br>50mg | breakfast<br>High-fat | 2/Day 4<br>Period | | 8:09 | 7:28 | 7:50 | N |
| | | | GSK123456 | breakfast | 2/Day 4 | | 8:11 | 7:30 | 7:41 | Y |
| | | | 25mg<br>GSK123456 | High-fat<br>breakfast | Period<br>2/Day 4 | | 8:09 | 7:25 | 7:42 | Y |
| | | | 10mg<br>GSK123456 | High-fat<br>breakfast | Period<br>2/Day 4 | | 8:10 | 7:27 | 7:36 | Y |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

### 10.10.2. Safety population

Example: AE1


Population: xxxxx

# Table x.x Xxxxxxxxxxxxxxxxxxxxxxxx

| System Organ Class | Placebo | Drug A | Drug B |
|----------------------------|----------|----------|----------|
| Preferred Term | (N=78) | (N=78) | (N=78) |
| ANY EVENT | 58 (74%) | 64 (82%) | 64 (85%) |
| Gastrointestinal disorders | | | |
| Any event | xx (xx%) | xx (xx%) | xx (xx%) |
| Dyspepsia | xx (xx%) | xx (xx%) | xx (xx%) |
| Nausea | xx (xx%) | xx (xx%) | xx (xx%) |
| Vomiting Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Constipation | xx (xx%) | xx (xx%) | xx (xx%) |
| Diarrhoea Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Toothache | xx (xx%) | xx (xx%) | xx (xx%) |
| Abdominal Pain Upper | xx (xx%) | xx (xx%) | xx (xx%) |
| Dry Mouth | xx (xx%) | xx (xx%) | xx (xx%) |
| Flatulence | xx (xx%) | xx (xx%) | xx (xx%) |
| Gastrointestinal Upset | xx (xx%) | xx (xx%) | xx (xx%) |
| Haemorrhoids | xx (xx%) | xx (xx%) | xx (xx%) |
| Loose Stools | xx (xx%) | xx (xx%) | xx (xx%) |
| Abdominal Pain Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Faecal Incontinence | xx (xx%) | xx (xx%) | xx (xx%) |
| Gastritis Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Lip Disorder Nos | xx (xx%) | xx (xx%) | xx (xx%) |
| Lip Dry | xx (xx%) | xx (xx%) | xx (xx%) |
| Stomach Discomfort | xx (xx%) | xx (xx%) | xx (xx%) |
| Nervous system disorders | | | |
| Any event | xx (xx%) | xx (xx%) | xx (xx%) |
| Headache | xx (xx%) | xx (xx%) | xx (xx%) |
| Dizziness | xx (xx%) | xx (xx%) | xx (xx%) |
| Extrapyramidal Disorder | xx (xx%) | xx (xx%) | xx (xx%) |

Extrapyramidal Disorder USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: AE5A


Population: xxxxx

#### 

Treatment: Treatment A (N=200)

| System Organ Class | | | | | | | 1 | MODERATE | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | | MILD | M | ODERATE | | SEVERE | | /SEVERE | UI | NKNOWN | | Total |
| ANY EVENT | 30 | (15%) | 40 | (20%) | 40 | (20%) | 80 | (40%) | 1 | (<1%) | 151 | (76%) |
| Cardiovascular | | | | | | | | | | | | |
| Any Event | 20 | (10%) | 40 | (20%) | 40 | (20%) | 80 | (40%) | 0 | | 140 | (70%) |
| Hypertension | 0 | | 20 | (10%) | 20 | (10%) | 20 | (10%) | 0 | | 40 | (20%) |
| Syncope | 0 | | 0 | | 0 | | 0 | | 0 | | 0 | |
| Hypotension | 20 | (10%) | 0 | | 0 | | 40 | (20%) | 0 | | 60 | (30%) |
| Nervous system | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |
| disorders | | | | | | | | | | | | |
| Any Event | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |
| _ | | | | | | | | | | | | |
| Dizziness | 10 | (5%) | 0 | | 0 | | 0 | | 1 | (<1%) | 11 | (6%) |

206817

Example: LB1


Population: xxxxx

#### 

| Test (units) | | | Planned | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | N | Time | n | Mean | SD | Median | Min. | Max. |
| Alkaline Phosphatase | Trt A | 202 | Week 8 | 150 | 2.1 | 7.95 | 1 | -25 | 32 |
| (IU/L) | | | Week 12 | 133 | 0.4 | 10.05 | 1 | -64 | 33 |
| | | | Week 24 | 55 | -1.6 | 18.22 | 0 | -339 | 44 |
| | Trt B | 220 | Week 8 | 150 | 2.1 | 7.95 | 1 | -25 | 32 |
| | | | Week 12 | 133 | 0.4 | 10.05 | 1 | -64 | 33 |
| | | | Week 24 | 55 | -1.6 | 18.22 | 0 | -339 | 44 |
| Alanine Aminotransferase (IU/L) | Trt A | 202 | Week 8 | 150 | -1.2 | 16.32 | 0 | -320 | 38 |
| | | | Week 12 | 133 | 0.7 | 10.55 | 1 | -64 | 32 |
| | | | Week 24 | 55 | -3.3 | 29.50 | 0 | -235 | 36 |
| | Trt B | 220 | Week 8 | 150 | -1.2 | 16.32 | 0 | -320 | 38 |
| | | | Week 12 | 133 | 0.7 | 10.55 | 1 | -64 | 32 |
| | | | Week 24 | 55 | -3.3 | 29.50 | 0 | -235 | 36 |

206817

Example: LB4


Population: xxxxx

#### 

Test= Alanine Aminotransferase (IU/L), Treatment=Treatment A

| Planned<br>Time | N | n | Baseline<br>Value | High | 1 | Norn | nal | Low | | Tota | al |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Week 1 | 100 | 100 | High<br>Normal<br>Low | 0<br>10<br>0 | (10%) | 1<br>84<br>0 | (1%)<br>(84%) | 3<br>2<br>0 | (3%)<br>(2%) | 4<br>96<br>0 | (4%)<br>(96%) |
| Week 4 | 100 | 100 | Total<br>High<br>Normal | 0 10 | (10%) | 85<br>1<br>84 | (85%)<br>(1%)<br>(84%) | 5<br>3<br>2 | (5%)<br>(3%)<br>(2%) | 100<br>4<br>96 | (100%)<br>(4%)<br>(96%) |
| | | | Low<br>Total | 0<br>10 | (10%) | 0<br>85 | (85%) | 0<br>5 | (5%) | 100 | (100%) |
| Worst Case<br>Post-Baseline | 100 | 100 | High | 0 | | 1 | (1%) | 3 | (3%) | 4 | (4%) |
| | | | Normal<br>Low | 10 | (10%) | 84 | (84%) | 2 | (2왕) | 96<br>0 | (96%) |
| | | | Total | 10 | (10%) | 85 | (85%) | 5 | (5%) | 100 | (100%) |

Example: UR3b


Population: xxxxx

#### 

| | D ' . 1/D1 1 | | | atment A<br>N=100) | | atment B<br>N=100) |
|---|---|---|---|---|---|---|
| Test | Period/Planned<br>Relative Time | Result | | | | |
| Urine General<br>Dipstick | SCREENING/<br>SCREENING | Positive | 30 | (30%) | 60 | (60%) |
| | | Negative | 40 | (40%) | 30 | (30%) |
| | | No Result | 30 | (30%) | 10 | (10%) |
| | PERIOD 1/DAY 1 | Positive | 40 | (40%) | 50 | (50%) |
| | | Negative | 30 | (30%) | 40 | (40%) |
| | | No Result | 30 | (30%) | 10 | (10%) |
| Urine Occult Blood (Dipstick) | SCREENING/<br>SCREENING | None | 40 | (40%) | 40 | (40%) |
| | | Trace | 25 | (25%) | 25 | (25%) |
| | | 1+<br>2+<br>3+ | 10<br>0<br>0 | (10%) | 15<br>0<br>0 | (15%) |
| | | No Result | 10 | (10%) | 20 | (20%) |
| | PERIOD 1/DAY 1 | None<br>Trace | 40<br>30 | (40%)<br>(30%) | 40<br>30 | (40%)<br>(30%) |
| | | 1+<br>2+ | 5<br>2 | (5%)<br>(2%) | 5<br>4 | (5응)<br>(4응) |
| | | 3+ | 0 | | 0 | |

206817

Example: EG1


Population: xxxxx

#### 

| | Trea | atment A<br>(N=157) | Trea | atment B<br>(N=160) |
|---|---|---|---|---|
| Time Period 1 | | | | |
| n | 156 | | 160 | |
| Normal | 81 | (52%) | 90 | (56%) |
| Abnormal, not clinically significant | 75 | (48%) | 69 | (43%) |
| Abnormal, clinically significant | 0 | , , | 1 | (<1%) |
| Time Period 2 | | | | |
| n | 117 | | 123 | |
| Normal | 50 | (43%) | 67 | (54%) |
| Abnormal, not clinically significant | 64 | (55%) | 55 | (45%) |
| Abnormal, clinically significant | 2 | (2%) | 1 | (<1%) |
| n | 117 | | 122 | |
| Clinically significant change from baseline | 2 | (2%) | 1 | (<1%) |
| Not a clinically significant change | 115 | (98%) | 121 | (>99%) |
| Not applicable | 0 | | 0 | |

206817

Example: EG1 (continued)

Population: xxxxx

#### 

| | Treatment A<br>(N=157) | Treatment B (N=160) |
|---|---|---|
| Any time post-baseline | | |
| n | 117 | 123 |
| Normal | 50 (43%) | 67 (54%) |
| Abnormal, not clinically significant | 65 (56%) | 55 (45%) |
| Abnormal, clinically significant | 2 (2%) | 1 (<1%) |
| No result (not available) | 0 | 0 |
| n | 117 | 122 |
| Clinically significant change from baseline | 2 (2%) | 1 (<1%) |
| Not a clinically significant change | 115 (98%) | 121 (>99%) |
| Not applicable | 0 | 0 |

206817

Example: EG2

Population: xxxxx

#### Planned Relative

Time

| | Treatment | N | | n | Mean | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Heart Rate | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (bpm) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | IIC D | 200 | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| PR Interval | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (msec) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | | | TIME 2 | T 0 0 | 24.0 | 10.07 | 09.0 | 1 4 | 123 |

206817

Example: VS1

Population: xxxxx

Planned Relative Time

| | | | TOTACT OF TIME | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Treatment | N | | n | Mean | SD | Median | Min. | Max. |
| Systolic BP | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (mmHg) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| Diastolic BP | Trt A | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| (mmHg) | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| - | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |
| | Trt B | 200 | Time 1 | 200 | 91.6 | 11.32 | 90.0 | 68 | 140 |
| | | | Time 2 | 190 | 92.4 | 9.83 | 90.0 | 70 | 122 |
| | | | Time 3 | 186 | 92.6 | 10.87 | 89.0 | 72 | 125 |

206817

Example: AE7


Population: xxxxx

#### 

| System Organ Class<br>Preferred Term | Treatment | No.<br>with<br>Event | Unique Subject Id. |
|---|---|---|---|
| Gastrointestinal disorders<br>Dyspepsia | Placebo | 9 | PPD |
| | Treatment A | 11 | |
| | Treatment B | 4 | |
| Nausea | Placebo | 6 | |
| | Treatment A | 8 | |
| | Treatment B | 4 | |

206817

Example: AE9CP


Population: xxxxx

#### 

| Site Id./ Unique Subject Id./ /Arm | Treatme nt/ Period | Age(YEARS)/<br>Sex/<br>Race<br>Detail/<br>Weight<br>(kg) | System Organ Class/<br>Preferred Term/<br>VERBATIM TEXT | Outcome/<br>Onset Datetime/<br>Datetime of<br>Resolution/<br>Duration | Time since<br>Study 1st<br>Dose/<br>Period 1st<br>Dose/<br>Last Dose | Maximum Intensity/ Maximum Grade/ Serious/ Withdrawal | Frequency/<br>Action Taken/<br>Relation to<br>Study<br>Treatment |
|---|---|---|---|---|---|---|---|
| AB-BA-BA | Tmt A/<br>Per 1 | 57/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE/<br>62.0 | Gastrointestinal<br>Disorders/<br>Internal spasm/<br>ENTERO - SPASM | PPD T06:05/T09:35/22d 13h 6m | 31d 26h 4m/ | MILD/<br>1<br>N/<br>N | INTERMITTENT/<br>DOSE REDUCED/<br>Y |
| | Tmt B/<br>Per 2 | 65/<br>M/<br>MIXED WHITE<br>RACE/<br>75.0 | Musculoskeletal and<br>connective tissue<br>disorders/<br>Arthralgia/<br>PAIN IN RIGHT<br>SHOULDER | PPD T05:50/T21:55/71d 9h 45m | 83d 1h 12m/ | MODERATE/<br>2/<br>N/<br>N | SINGLE EVENT/<br>DOSE NOT<br>CHANGED/<br>N |

206817

Example: AE2

Population: xxxxx

Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| System Organ Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system disorders | Lymphadenopathy | ENLARGED LYMPH NODE |
| Cardiac disorders | Palpitations<br>Ear pain | CLOGGED EARS WITH EAR WAX EARACHES IN BOTH EARS |
| | Lat Pari | RIGHT EAR PAIN |
| | Tinnitus | RINGING IN RIGHT EAR |
| Eye disorders | Asthenopia | TIRED EYES |
| | Conjunctivitis | BILATERAL ACUTE CONJUNCTIVITIS |
| | | CONJUNCTIVITIS |
| | Dry eye nos | DRY EYES |
| | Eye redness | REDDENED EYES |
| | Vision blurred | BLURRED VISION |
| | | BLURRY VISION |
| | | WORSENING OF BLURRED VISION |
| Gastrointestinal disorders | Abdominal pain nos | ABDOMEN PAIN |
| | Abdominal pain upper | MID-EPIGASTRIC AREA PAIN |
| | | STOMACH ACHE |
| • | • | • |
| • | • | • |

206817

Example: CP\_LB6
Protocol: GSK123456

Population: xxxxx

### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./<br>Subj./ | Age(y)/<br>Sex/ | Treat-<br>ment/ | Lab test | Planned<br>Relative | | Study<br>Day/<br>Period | Co | nverted Data | Fl | ag[1 | ] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Seq | Race | Period | (units) | Time | Date/Time | Day | Value | Normal Range | NR | . CI | BL |
| PPD | 63/ | Trt A/ | Alk Phos | Screening | PPD<br>12:05 | -1/-1 | 64.00 | 32.0- 92.0 | | | |
| | Male/ | Per 1 | ( - / - / | Week 12 | PPD | 85/85 | 84.00 | 32.0- 92.0 | | | |
| | | | | | 13:45 | | | | | | |
| | White | | | | | | | | | | |
| | | | ALT (U/L) | Screening | PPD<br>13:32 | -1/-1 | 29.00 | 10.0- 40.0 | | | |
| | | | | Week 12 | PPD | 85/85 | 70.00 | 10.0- 40.0 | Н | Н | Н |
| | | | | | 09:55 | | | | | | |

206817

Example: UR2b


Population: xxxxx

#### 

| Inv. | Subject | Treatment | Period | Visit | Sample Date | Study<br>Day | Period<br>Day | Urinalysis<br>Test | Result |
|---|---|---|---|---|---|---|---|---|---|
| PPD | | Trt A | 1 | 1 | PPD | 1 | 1 | Blood | ++ or 2+ |
| | | Trt B | 2 | 8 | | 137 | 1 | Blood | + or 1+ |
| | | Trt B | 1 | 1 | | 1 | 1 | Blood | + or 1+ |
| | | Trt A | 2 | 8 | | 137 | 1 | Protein<br>Blood | +++ or 3+<br>+ or 1+ |

206817

Example: LIVER5

Population: xxxxx

#### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxxx

Treatment: Treatment A

| Site Id./<br>Unique Subject<br>Id. | Age(YEARS)/<br>Sex/<br>Race Detail | Maximum Status of<br>the Liver Event | Date First<br>Detected/<br>Study Day | Time<br>Since<br>First<br>Dose<br>(days) | Time<br>Since<br>Last<br>Dose<br>(days) | Restart/Re-<br>challenge After<br>Stopping Criteria<br>Was Met | Resolved?/<br>Date<br>resolved |
|---|---|---|---|---|---|---|---|
| PPD | 63/<br>M/<br>WHITE -<br>WHITE/CAUSAS<br>IAN/EUROPEAN<br>HERITAGE | LIVER MONITORING<br>CRITERIA | <b>PPD</b><br>101 | 101 | 1 | N | Y/<br>2010-02-19 |
| | 61/<br>F/<br>ASIAN -<br>JAPANESE<br>HERITAGE | LIVER EVENT<br>STOPPING CRITERIA | <b>PPD</b><br>68 | 68 | 1 | Y | Y/<br>2010-04-10 |
| | | LIVER EVENT<br>STOPPING CRITERIA | PPD<br>134 | 134 | 7 | N | N |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: SU2


Population: xxxxx

#### 

| | Inv./<br>Subj. | Visit | Study<br>Day | Assess-<br>ment<br>Date | Smoking<br>History | Cur-rently<br>Smoke | Last<br>Smoked | Smoked<br>Since<br>Last<br>Visit | Days<br>Smoked<br>Since<br>Last<br>Visit | Years<br>Smoked | Ciga-<br>rettes<br>/day | Smoki<br>ng<br>Pack<br>Years<br>* |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Trt A | PPD | Visit 1 | 1 | PPD | Never | No | | No | Zero | | | |
| | | Visit 1 | 1 | | Current | Yes | | Yes | A few | 5 | 20 | 5 |
| Trt B | | Visit 1 | 1 | | Former | No | 31DEC1<br>990 | No | Zero | 18 | 30 | 27 |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_EG4
Protocol: GSK123456
Population: xxxxx


#### 

| | | | | | Actual | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Inv./ | Age | Treat- Planned | | Study | Relative | Heart | PR | QRS | RR | QΤ | | |
| Subj. | (y)/ | ment/ Relative | ECG | Day | Time | Rate | Int. | Dur. | Int. | Int. | QTcB | QTcF |
| /Seq. | Sex/ | Period Time | Date/Time | /Period | (optional) | (bpm) | (msec | (mse | (msec) | (msec) | (msec) | (msec) |
| | Race | | | Day | | | ) | c) | | | | |
| PPD | 65/ | Trt A/ Time 1 | PPD | 1/1 | -30m | 60 L | 150 | 350 | 750 | 450 | 520 | 495 |
| | White/ | Per 1 | 14:00 | | | | | | | | | |
| /AB | Female | | | | | | | | | | | |
| | | Time 2 | PPD | 7/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 15:00 | | | | | | | | | |
| | | Trt B/ Time 1 | PPD | 14/1 | -30m | 80 | 150 | 390 | 750 | 450 | 520 | 495 |
| | | Per 2 | 19:00 | • | | | | Н | | | | |
| | | Time 2 | PPD | 21/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 20:00 | | | | | | | | | |
| PPD | 58 | Trt A/ Time 1 | PPD | 1/1 | -30m | 80 | 90 L | 350 | 800 н | 450 | 520 | 495 |
| | Male/ | Per 2 | 14:00 | , | | | | | | | | |
| /BA | White/ | | | | | | | | | | | |
| | | Time 2 | PPD | 7/7 | 26m | 80 | 150 | 350 | 750 | 450 | 520 | 495 |
| | | | 15:00 | _ | | | | | | | | |

206817

Example: CP\_EG6
Protocol: GSK123456


#### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./<br>Subj./<br>Seq. | Age (y)/<br>Sex/<br>Race | Treat-<br>ment/<br>Period | Planned<br>Relative<br>Time/ECG<br>Date/Time | Study<br>Day/<br>Period<br>Day | ECG Finding | Clinically<br>Significant<br>Change from<br>Baseline? | Clinically<br>Significant Abnormality |
|---|---|---|---|---|---|---|---|
| PPD<br>A/B | 65/<br>Female/<br>White | Trt A/<br>Per 1 | Visit 1/<br>PPD<br>/14:00 | 1/1 | Normal | | |
| | | | Visit 2/<br>PPD<br>/12:00 | 4/4 | Abnormal-not clinically significant | No | |
| | | Trt B/<br>Per 2 | Visit 3/<br>PPD<br>/19:00 | 8/1 | Abnormal-<br>clinically<br>significant | | Sinus tachycardia |
| | | | Visit 4/<br>PPD<br>/13:00 | 12/4 | No result (not available) | | |
| PPD<br>B/A | 58<br>Male/<br>White | Trt B/<br>Per 1 | Visit 1/<br>PPD<br>/14:00 | 16/1 | Abnormal-<br>clinically<br>significant | | Ectopic ventricular beats |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: CP\_VS5
Protocol: GSK123456
Population: xxxxx


#### 

| | | | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|---|---|
| Inv./ | Age(y)/ | Treat- | Planned | | | Blood | Blood | Vital Sign |
| Subj./ | Sex/ | ment/ | Relative | Actual | Study Day/ | Pressure | Pressure | 3 |
| Seq. | Race | Period | Time | Date/Time | Period Day | (mmHg) | (mmHg) | (units) |
| PPD | 23/ | Tmt B/ | Time 1 | PPD | 1/1 | 190 н | 60 | xx H |
| | Male/ | Per 1 | Time 2 | | 5/5 | 95 | 50 L | xx H |
| B/C/A | White | | Time 3 | | 10/10 | 95 | 60 | XX |
| | | Tmt C/ | Time 1 | | 15/1 | 185 Н | 90 н | xx H |
| | | Per 2 | Time 2 | | 20/5 | 95 | 50 | xx H |
| | | | Time 3 | | 25/10 | 95 | 60 | XX |
| | | Tmt A/ | Time 1 | | 30/1 | 200 Н | 45 L | xx H |
| | | Per 3 | Time 2 | | 35/5 | 95 | 60 | xx H |
| | | | Time 3 | | 40/10 | 95 | 85 H | XX |

206817

Example: SAFE\_L1
Protocol: GSK123456
Population: xxxxx


### Listing x.x

#### xxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Inv./ | Age(y)/ | Treat-ment/ | Planned | Actual | Study Day/ | Location/ | Test type | Side | Test |
|---|---|---|---|---|---|---|---|---|---|
| Subj./ | Sex/ | Period | Relative | Date/Time | Period Day | Category | | | Result |
| Seq. | Race | | Time | | | | | | |
| PPD | 23/ | Tmt B/ | Time 1 | PPD | 1/ | Eye/ | Indirect | Left | Normal |
| | | | | | | | fundoscopic | | |
| | | | | | | | exam | | |
| | Male/ | Period x | | | 1 | Ophthalmological | | Right | XXXXX |
| | | | | | | examination | | | |
| B/C/A | White | | | | | | Slit lamp | Left | XXXXXX |
| | | | | | | | | Right | XXXXXX |
| | | | Time 2 | | 5/ | | xxxxxxxxx | xxxxx | XXXXXX |
| | | | | | 5 | | | XXXXX | XXXXXXX |
| | | | | | | | xxxxxxxxx | XXXXX | xxxxxx |
| | | | | | | | | XXXXX | XXXXXXX |
| | | Tmt C/ | Time 1 | | 15/ | | xxxxxxxxx | xxxxx | XXXXXX |
| | | Period 2 | | | 1 | | | XXXXX | xxxxxxx |

USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

### 10.10.3. PK population

206817

Example: PK01


Population: xxxxx

#### 

| Treatmen<br>t | N | {Add.<br>time<br>var.} | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | {95% CI (Lower, Upper)} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 50mg | 24 | | Pre-dose | 24 | 20 | XXXX.X | (xxxx.x,xxxx.x) | | xxxx.x | XXXX | xxxx |
| Joney | 27 | | 30 min | 24 | 1 | XXXX.X | (XXXX.X, XXXX.X) | xx.xx | XXXX.X | XXXX | XXXX |
| | | | 1 hr | 23 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| | | | 2 hr | 24 | 0 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 100mg | 24 | | Pre-dose | 24 | 3 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 2 | | | 30 min | 21 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | xxxx.x | XXXX | XXXX |
| | | | 1 hr | 21 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | xxxx.x | XXXX | XXXX |
| | | | 2 hr | 21 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 200mg | 24 | | Pre-dose | 24 | 0 | xxxx.x | (xxxx.x,xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |
| 2 | | | 30 min | 23 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | xxxx.x | XXXX | XXXX |
| | | | 1 hr | 24 | 0 | XXXX.X | (xxxx.x,xxxx.x) | xx.xx | xxxx.x | XXXX | XXXX |
| | | | 2 hr | 24 | 0 | XXXX.X | (xxxx.x, xxxx.x) | XX.XX | XXXX.X | XXXX | XXXX |

206817

Example: PK03


Population: xxxxx

#### 

| Parameter | Treatment | N | {Additio<br>nal<br>time<br>variable<br>s} | n | Mean | {95% CI<br>(Lower,Upper)<br>} | SD | Median | Min. | Max. |
|---|---|---|---|---|---|---|---|---|---|---|
| AUC(0-t) (units) | 50mg | 24 | 1 | 24 | XXXX.XX | (xxxx.xx,xxxx<br>.xx) | xx.xx<br>x | xxxx.xx | xxxx.x | XXXX.X |
| | | | 14 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | XXXX.X |
| | 100mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | xx.xx<br>x | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 23 | xxxx.xx | (xxxx.xx, xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | xxxx.x |
| Cmax (units) | 50mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | xx.xx<br>x | xxxx.xx | xxxx.x | xxxx.x |
| | | | 14 | 23 | xxxx.xx | (xxxx.xx, xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | xxxx.x |
| | 100mg | 24 | 1 | 24 | xxxx.xx | (xxxx.xx,xxxx<br>.xx) | XX.XX | xxxx.xx | XXXX.X | xxxx.x |
| | | | 14 | 21 | xxxx.xx | (xxxx.xx, xxxx<br>.xx) | XX.XX<br>X | xxxx.xx | xxxx.x | xxxx.x |

(xxxx.xx,xxxx.xx)

(xxxx.xx,xxxx.xx)

XX.XXX

XX.XXX

XX.XX

XX.XX

Example: PK05


Population: xxxxx

#### 

#### {Additiona 1 Geom. 95% CI time {%CVb} Parameter Treatment Ν n Mean (Lower, Upper) SD variables} (logs) 24 AUC(0-t)50mg 1 24 (xxxx.xx,xxxx.xx)XXXX.XX XX.XXX XX.XX (units) 14 24 XXXX.XX (xxxx.xx,xxxx.xx)XX.XXX XX.XX 100mg 24 1 24 XXXX.XX (xxxx.xx, xxxx.xx)XX.XX XX.XXX 14 23 XXXX.XX (xxxx.xx, xxxx.xx) ${\tt XX.XXX}$ XX.XX 200mg 24 1 24 XXXX.XX (xxxx.xx, xxxx.xx)XX.XXX XX.XX 21 14 XXXX.XX (xxxx.xx, xxxx.xx)xx.xx XX.XXX Cmax 50mg 24 1 24 XXXX.XX (xxxx.xx, xxxx.xx)XX.XXX XX.XX (units) 14 24 (xxxx.xx, xxxx.xx)XXXX.XX XX.XXX XX.XX 100mg 24 1 24 (xxxx.xx, xxxx.xx)XXXX.XX XX.XXX XX.XX 14 23 XXXX.XX (xxxx.xx,xxxx.xx)XX.XXX XX.XX

USER ID: directory/program.sas DDMMMYYYY hh:mm

200mg

24

1

14

24

21

XXXX.XX

XXXX.XX

206817

Example: PK\_T1

Population: xxxxx

Table x.x

XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX

| Parameter | Effect | n Sl | lope Point | SE | 90% CI |
|------------|------------------|------|------------|-----|----------|
| | | Es | stimate | | |
| Parameter1 | Log(dose levels) | XX | XXX | xxx | (xx,xx) |
| Parameter2 | Log(dose levels) | XX | XXX | XXX | (xx, xx) |
| ٠ | • | | • | • | • |
| ٠ | • | | • | • | • |

206817

Example: PK\_T2

Population: xxxxx

#### Table x.x xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx

| Parameter | Treatment | N | n | Geometric LS Mean | Ratio (Fasted/Fed) | 90% CI | CVw(%)[1] |
|---|---|---|---|---|---|---|---|
| Parameter1 (unit) | Trt1 | XX | XX | XXX | Xxx | (xx,xx) | XX |
| | Trt2 | XX | XX | xxx | | | |
| Parameter2 (unit) | Trt1 | XX | XX | xxx | xxx | (xx, xx) | xx |
| | | | | | • | • | |
| • | • | • | • | • | • | • | • |
| • | • | • | • | • | • | • | • |
| ParameterX (unit) | XX | XX | XX | XXX | XXX | (xx, xx) | XX |

Example: PK16b

Population: xxxxx

Figure x.x
xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK24

Population: xxxxx

#### Treatment = tablet original fed



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK18




USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK\_F1

Population: xxxxx



USER ID: directory/program.sas DDMMMYYYY hh:mm

Example: PK28


Population: xxxxx



USER ID: directory/program.sas DDMMMYYYY hh:mm

206817

Example: PK08 (pkcl1x)
Protocol: GSK123456
Population: xxxxx


| {Inv./}<br>Subj. | {Age(y)/<br>Sex/<br>Race} | Period<br>/Tmt. | Date | Study<br>Day /<br>Period<br>Day | Planned<br>Relative<br>Time | Actual<br>time | Time dev.<br>(units) | Actual<br>Relative<br>Time | Concentration (units) |
|---|---|---|---|---|---|---|---|---|---|
| PPD | 36/<br>M/<br>Mixed Race | 1/<br>50mg | PPD | 1/1 | pre-dose | 11:55 | 0 | 0h 0m 0s | 123 |
| | | | | | 5m | 12:05 | 0 | 0h 5m 0s | 1434 |
| | | | | | 1h | 13:00 | 0 | 1h 0m 0s | NQ (<0.23) |
| | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |
| | | 2/<br>100mg | | 17/1 | pre-dose | 11:57 | 0 | 0h 0m 0s | 435 |
| | | 2 | | | 5m | 12:10 | 0.83 | 0h 10m 0s | 34566 |
| | | | | | 1h | 12:56 | -0.67 | 0h 56m 0s | 3452 |
| | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |
| | 33/<br>M/<br>Mixed Race | 1/<br>50mg | | 1/1 | pre-dose | 11:58 | 0 | 0h 0m 0s | 2345 |
| | mana nace | | | | 5m | 12:04 | -0.17 | 0h 4m 0s | 234 |
| | | | | | 1h | 12:35 | 0.83 | 1h 0m 0s | NR |
| | | | | | 1h 30m | 13:30 | 0 | 1h 30m 0s | 30 |

206817

Example: PK14


Population: xxxxx

# Listing x.x Xxxxxxxxxxxxxxxxxxxxx

| {Inv./}<br>Subj. | {Age(y)/<br>Sex/<br>Race} | Period/<br>Tmt. | AUC(0-inf)<br>(units) | AUC(0-t)<br>(units) | Cmax<br>(units) | t1/2<br>(units) | tmax<br>(units) |
|---|---|---|---|---|---|---|---|
| PPD | 36/<br>M/ | 1/<br>50mg | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| | Mixed Race | 2/<br>100mg | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX |
| | 33/<br>M/ | 1/<br>50mg | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Mixed Race | 2/<br>100mg | xx.xx | xx.xx | XX.XX | XX.XX | XX.XX |
| | 24/<br>M/ | 1/<br>50mg | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | Mixed Race | 2/<br>100mg | xx.xx | xx.xx | xx.xx | XX.XX | XX.XX |